# CLINICAL RESEARCH IN INFECTIOUS DISEASES

# STATISTICAL ANALYSIS PLAN

# for

# **DMID Protocol**

17-0077: A Phase II Study in Healthy Adults (19-64 Years of Age) to Assess the Safety, Reactogenicity and Immunogenicity of Sequential or Simultaneous Intramuscular Administration of an AS03-adjuvanted A/H7N9 Inactivated Influenza Vaccine with Seasonal Influenza Vaccine

17-0077: NCT03318315

Version 1.0

DATE: 14 November 2018

THIS COMMUNICATION IS PRIVILEGED AND CONFIDENTIAL

#### **STUDY TITLE**

| <b>Protocol Number Code:</b> | DMID Protocol: 17-0077 |
|---|---|
| <b>Development Phase:</b> | Phase II |
| Products: | Sanofi A/H7N9 Inactivated Influenza Vaccine<br>GSK AS03 Adjuvant<br>Seasonal influenza vaccine (IIV4) |
| Form/Route: | IM |
| Indication Studied: | Influenza A/H7N9 |
| Sponsor: | Division of Microbiology and Infectious Diseases National Institute of Allergy and Infectious Diseases National Institutes of Health |
| Clinical Trial Initiation Date: | 20 February 2018 |
| Clinical Trial Completion Date: | Expected June 2019 |
| Date of the Analysis Plan: | 14 November 2018 |
| Version Number: | 1.0 |

This study was performed in compliance with Good Clinical Practice.

Information contained in this publication is the property of Division of Microbiology and Infectious Diseases and is confidential. This information may not be disclosed to third parties without written authorization from Division of Microbiology and Infectious Diseases. This report may not be reproduced, stored in a retrieval system or transmitted in any form or by any means - electronic, mechanical, recording or otherwise - without the prior authorization from Division of Microbiology and Infectious Diseases. This document must be returned to Division of Microbiology and Infectious Diseases upon request.

# **TABLE OF CONTENTS**

| STUDY TITI | LE | II |
|---|---|---|
| TABLE OF C | CONTENTS | III |
| LIST OF AB | BREVIATIONS | VI |
| 1. PREFAC | CE | 1 |
| 2. INTROI | DUCTION | 2 |
| 2.1. Purp | pose of the Analyses | 2 |
| 3. STUDY | OBJECTIVES AND ENDPOINTS | 3 |
| 3.1. Stud | ly Objectives | 3 |
| 3.1.1. | Primary | 3 |
| 3.1.2. | Secondary | 3 |
| 3.1.3. | Exploratory | 3 |
| 3.2. End | points | 4 |
| 3.2.1. | Primary | 4 |
| 3.2.2. | Secondary | 5 |
| 3.2.3. | Exploratory | 5 |
| 3.3. Stud | ly Definitions and Derived Variables | 6 |
| 4. INVEST | TIGATIONAL PLAN | 7 |
| 4.1. Ove | rall Study Design and Plan | 7 |
| 4.2. Disc | cussion of Study Design, Including the Choice of Control Groups | 8 |
| 4.3. Sele | ction of Study Population | 8 |
| 4.4. Trea | itments | 8 |
| 4.4.1. | Treatments Administered | 8 |
| 4.4.2. | Identity of Investigational Product | 8 |
| 4.4.3. | Method of Assigning Subjects to Treatment Groups (Randomization) | 8 |
| 4.4.4. | Selection of Doses in the Study | 8 |
| 4.4.5. | Selection and Timing of Dose for Each Subject | 9 |
| 4.4.6. | Blinding | 9 |
| 4.4.7. | Prior and Concomitant Therapy | 9 |
| 4.4.8. | Treatment Compliance | 9 |
| 4.5. Imm | nunogenicity and Safety Variables | 10 |
| 4.5.1. | Safety Variables | 10 |
| 4.5.2. | Immunogenicity Variables | 10 |

# TABLE OF CONTENTS (continued)

| 5. | S | SAMPL | E SIZE CONSIDERATIONS | 12 |
|---|---|---|---|---|
| 6. | ( | GENER. | AL STATISTICAL CONSIDERATIONS | 13 |
| | 6.1. | Gen | eral Principles | 13 |
| | 6.2. | Tim | ing of Analyses | 13 |
| | | 6.2.1. | Preliminary Report and CSR | 13 |
| | 6.3. | Ana | lysis Populations | 14 |
| | | 6.3.1. | Safety Population | 14 |
| | | 6.3.2. | Modified Intention-to-Treat (mITT) Population | 14 |
| | | 6.3.3. | Per Protocol Population | 14 |
| | 6.4. | Cov | ariates and Subgroups | 15 |
| | 6.5. | Miss | sing Data | 15 |
| | 6.6. | Inter | rim Analyses and Data Monitoring | 15 |
| | | 6.6.1. | Interim Safety Review | 15 |
| | | 6.6.2. | Interim Immunogenicity Review | 16 |
| | 6.7. | Mul | ticenter Studies | 16 |
| | 6.8. | Mul | tiple Comparisons/Multiplicity | 16 |
| 7. | 5 | STUDY | SUBJECTS | 17 |
| | 7.1. | Subj | ect Disposition | 17 |
| | 7.2. | Prot | ocol Deviations | 17 |
| 8. | I | MMUN | OGENICITY EVALUATION | 18 |
| | 8.1. | Prin | nary Immunogenicity Analysis | 18 |
| | 8.2. | Seco | ondary Immunogenicity Analyses | 19 |
| | 8.3. | Expl | loratory Immunogenicity Analyses | 19 |
| | | 8.3.1. | Covariate Analysis | 19 |
| | | 8.3.2. | Regression Modeling. | 19 |
| | | 8.3.3. | NA Serum Antibody Responses | 20 |
| 9. | 5 | SAFETY | Y EVALUATION | 21 |
| | 9.1. | Dem | nographic and Other Baseline Characteristics | 21 |
| | | 9.1.1. | Prior and Concurrent Illnesses and Medical Conditions | 21 |
| | | 9.1.2. | Prior and Concurrent Medications | 21 |
| | 9.2. | Mea | surements of Treatment Compliance | 22 |
| | 9.3. | Adv | erse Events | 22 |

# TABLE OF CONTENTS (continued)

| | 9.3.1. | Solicited Events and Symptoms | 22 |
|---|---|---|---|
| | 9.3.2. | Unsolicited Adverse Events | 23 |
| 9.4. | Deatl | hs, Serious Adverse Events and other Significant Adverse Events | 24 |
| 9.5. | Pregi | nancies | 24 |
| 9.6. | Clini | cal Laboratory Evaluations | 25 |
| 9.7. | Vital | Signs and Physical Evaluations | 25 |
| 9.8. | Conc | comitant Medications | 25 |
| 10. R | EPORT | TING CONVENTIONS | 26 |
| 11. T | ECHNI | CAL DETAILS | 27 |
| 12. S | UMMA | ARY OF CHANGES IN THE CONDUCT OF THE STUDY OR PLANNED ANAL | YSES28 |
| 13. R | EFERE | NCES | 29 |
| 14. A | PPEND | DICES | 30 |
| APPE | NDIX 1 | . TABLE MOCK-UPS | 31 |
| APPE | NDIX 2 | FIGURE MOCK-UPS | 145 |
| APPE | NDIX 3 | LISTINGS MOCK-UPS | 163 |

# LIST OF ABBREVIATIONS

| AE | Adverse Event |
|--------|--------------------------------------------------|
| ALT | Alanine Aminotransferase |
| BP | Blood Pressure |
| С | Celsius |
| CI | Confidence Interval |
| Cr | Creatinine |
| CRF | Case Report Form |
| CSR | Clinical Study Report |
| DMID | Division of Microbiology and Infectious Diseases |
| DSMB | Data and Safety Monitoring Board |
| eCRF | Electronic Case Report Form |
| F | Fahrenheit |
| FDA | U.S. Food and Drug Administration |
| GMT | Geometric Mean Titer |
| GSK | GlaxoSmithKline |
| HAI | hemagglutination inhibition antibody |
| Hgb | Hemoglobin |
| HHS | U.S. Department of Health and Human Services |
| ICH | International Conference on Harmonisation |
| IIV | Inactivated Influenza Vaccine |
| IM | Intramuscularly |
| IRB | Institutional Review Board |
| L | Liter |
| MAAE | Medically Attended Adverse Event |
| mcg | Microgram |
| MedDRA | Medical Dictionary for Regulatory Activities |
| mg | Milligram |
| mITT | Modified Intention to Treat |
| N, n | Number |
| NA | neuraminidase |
| Neut | Neutralizing Antibody |

# LIST OF ABBREVIATIONS (continued)

| NIH | National Institutes of Health |
|---------|-----------------------------------------------|
| NOCMC | New Onset Chronic Medical Condition |
| PIMMC | Potentially Immune Mediated Medical Condition |
| PP | Per Protocol |
| PLT | Platelets |
| PT | Preferred Term |
| RCD | Reverse Cumulative Distribution |
| SAE | Serious Adverse Event |
| SD | Standard Deviation |
| SDCC | Statistical and Data Coordinating Center |
| SMC | Safety Monitoring Committee |
| SOC | System Organ Class |
| T. Bili | Total Bilirubin |
| WBC | White Blood Cell |
| WHO | World Health Organization |

#### 1. PREFACE

This Statistical Analysis Plan (SAP) for DMID Protocol 17-0077, "A Phase II Study in Healthy Adults (19-64 Years of Age) to Assess the Safety, Reactogenicity and Immunogenicity of Sequential or Simultaneous Intramuscular Administration of an AS03-adjuvanted A/H7N9 Inactivated Influenza Vaccine with Seasonal Influenza Vaccine," describes and expands upon the statistical information presented in the protocol.

This document describes all planned analyses and provides reasons and justifications for these analyses. It also includes sample tables, figures, listings (TFLs) planned for (1) final analyses included in the preliminary report, and (2) analyses included in the Clinical Study Report (CSR). Regarding the final analyses and CSR, this SAP follows the International Conference on Harmonisation of Technical Requirements for Registration of Pharmaceuticals for Human Use (ICH) Guidelines, as indicated in Topic E3 (Structure and Content of Clinical Study Reports), and more generally is consistent with Topic E8 (General Considerations for Clinical Trials) and Topic E9 (Statistical Principles for Clinical Trials). The structure and content of the SAP provides sufficient detail to meet the requirements identified by the FDA and ICH, while all work planned and reported for this SAP will follow internationally accepted guidelines published by the American Statistical Association and the Royal Statistical Society for statistical practice.

This document contains four sections: (1) a review of the study design, (2) general statistical considerations, (3) comprehensive statistical analysis methods for immunogenicity and safety outcomes, and (4) a list of proposed tables, figures and listings (TFLs). Following any protocol amendment, this SAP will be reviewed and revised (if needed) to address any changes in the protocol impacting analysis. Any deviation from the final SAP will be described and justified in the CSR. The reader of this SAP is encouraged to also review the study protocol for details on conduct of the study and the operational aspects of clinical assessments.

#### 2. INTRODUCTION

Since March of 2013 [1], avian influenza A/H7N9 viruses have continued to circulate in China causing discrete outbreaks (or waves) in humans with high mortality over the past 5 years. By late 2016, a fifth wave of outbreaks was identified in China and as of May 18, 2017, a total of 1,463 laboratory-confirmed human infections with avian influenza A/H7N9 virus have been reported by the World Health Organization [2, 3]. Since the onset of the fifth wave of A/H7N9 outbreaks in October 2016, more human cases of A/H7N9 infection have been reported in China than any prior A/H7N9 epidemic wave [3]. The U.S. Department of Health and Human Services (HHS) recently assessed A/H7N9 influenza virus as having a significant potential to cause a pandemic, and the greatest risk of causing severe disease. As a result, HHS has supported the production of fifth wave A/H7N9 inactivated influenza 9 vaccines (IIVs) for the U.S. stockpile and for an assessment of their safety and immunogenicity in clinical trials.

The goal of this clinical trial is to assess in healthy adults the safety, reactogenicity, and immunogenicity of two doses of AS03-adjuvanted 2017 A/H7N9 inactivated influenza vaccine (IIV) administered simultaneously (Group 1) or sequentially (Group 2) with seasonal influenza vaccine (IIV4), and to assess potential interference with the immunogenicity of either vaccine. A comparator group will receive IIV4 only at baseline (Group 3). The two doses of the A/H7N9 vaccine given with AS03 adjuvant will be administered approximately 21 days apart.

# 2.1. Purpose of the Analyses

These analyses will assess the safety and immunogenicity of two doses of AS03-adjuvanted 2017 A/H7N9 IIV administered sequentially or simultaneously with seasonal influenza vaccine and will be included in the clinical study report.

#### 3. STUDY OBJECTIVES AND ENDPOINTS

## 3.1. Study Objectives

#### **3.1.1. Primary**

## Safety:

• To assess the safety and reactogenicity following sequential or simultaneous intramuscular (IM) administration of 2 doses of AS03-adjuvanted 2017 A/H7N9 IIV and one dose of seasonal influenza vaccine (IIV4).

## Immunogenicity:

- To assess the serum hemagglutination inhibition (HAI) and neutralizing (Neut) antibody responses against A/H7N9 at approximately 21 days following receipt of two doses of AS03-adjuvanted 2017 H7N9 IIV administered IM approximately 21 days apart.
- To assess the serum HAI and Neut antibody responses against the seasonal influenza strains at approximately 21 days following receipt of IIV4.

#### 3.1.2. Secondary

#### Safety:

- To assess unsolicited non-serious adverse events following sequential or simultaneous IM administration of AS03-adjuvanted 2017 A/H7N9 IIV and seasonal influenza vaccine (IIV4).
- To assess medically attended adverse events (MAAEs), including new onset chronic medical conditions (NOCMCs) and potentially immune mediated conditions (PIMMCs), following sequential or simultaneous IM administration of AS03-adjuvanted 2017 A/H7N9 IIV and IIV4.

#### Immunogenicity:

• To assess the HAI and Neut antibody responses at 21 days following receipt of 1 dose of AS03-adjuvanted 2017 A/H7N9 IIV.

#### 3.1.3. Exploratory

#### Immunogenicity:

 To assess the effects of age, sex, BMI, and receipt of prior year(s) seasonal influenza vaccine(s) on serum HAI antibody responses following receipt of two doses of AS03adjuvanted 2017 A/H7N9 IIV.

- To assess the durability of the antibody response to the 2017 A/H7N9 study vaccine strain and the IIV4 strains at approximately 180 days following the second dose of AS03-adjuvanted 2017 A/H7N9 IIV vaccine.
- To assess the neuraminidase (NA) content of the 2017 H7N9 IIV and the licensed seasonal IIV4 and determine the serum antibody responses to NA following receipt of 2017 H7N9 IIV. *Note: analysis plans for this objective will be described in an addendum to this SAP once the NA assay has been selected.*

# 3.2. Endpoints

#### **3.2.1. Primary**

#### Safety:

- Occurrence of all serious adverse events (SAEs) following the first study vaccination through approximately 12 months after the last study vaccination.
- Occurrence of study vaccine-related SAEs following the first study vaccination through approximately 12 months after the last study vaccination.
- Occurrence of solicited injection site and systemic adverse events (AEs) following each study vaccination through 7 days after each study vaccination.
- Occurrence of clinical safety laboratory AEs following each study vaccination through approximately 7 days after each study vaccination.

#### Immunogenicity:

- For HAI and Neut antibodies, percentage of subjects achieving seroconversion against the 2017 H7N9 study vaccine strain (defined as either a pre-vaccination titer <1:10 and a post-vaccination titer ≥1:40 or a pre-vaccination titer ≥1:10 and a minimum four-fold rise in post-vaccination antibody titer) at approximately 21 days after 2 doses of AS03-adjuvanted 2017 H7N9 IIV (Group 1− Day 43; Group 2 − Day 64; Group 3 − N/A).
- For HAI and Neut antibodies, percentage of subjects achieving seroconversion against each of the study IIV4 strains at approximately 21 days after receipt of study IIV4 (Groups 1, 2 and 3 Day 22).
- For HAI and Neut antibodies, percentage of subjects with an antibody titer of ≥1:40 against the influenza 2017 H7N9 study vaccine strain at approximately 21 days following receipt of 2 doses of AS03-adjuvanted 2017 H7N9 IIV (Group 1 Day 43; Groups 2 Day 64; Group 3 N/A).
- For HAI and Neut antibodies, percentage of subjects with an antibody titer of ≥1:40 against each of the study IIV4 strains at approximately 21 days after receipt of study IIV4 (Groups 1, 2 and 3 Day 22).

- GMTs of serum HAI and Neut antibodies against the 2017 H7N9 IIV strain at approximately 21 days following receipt of 2 doses of AS03-adjuvanted 2017 H7N9 IIV (Group 1– Day 43; Group 2 Day 64; Group 3 N/A).
- GMTs of serum HAI and Neut antibodies against each of the 2017 IIV4 strains at approximately 21 days after receipt of IIV4 (Group 1, 2 and 3– Day 22).

#### 3.2.2. Secondary

#### Safety:

- Occurrence of study vaccine-related unsolicited non-serious AEs following each study vaccination through approximately 21 days after each study vaccination.
- Occurrence of all unsolicited non-SAEs following each study vaccination through approximately 21 days after each study vaccination.
- Occurrence of MAAEs, including NOCMCs and PIMMCs, following the first study vaccination through approximately 12 months after the last study vaccination.

#### Immunogenicity:

- For HAI and Neut antibodies, percentage of subjects achieving seroconversion against the 2017 H7N9 vaccine strain at approximately 21 days after receipt of 1 dose of AS03-adjuvanted 2017 H7N9 IIV (Group 1– Day 22; Group 2 – Day 43; Group 3 – N/A).
- For HAI and Neut antibodies, percentage of subjects achieving serum HAI and Neut antibody titers ≥1:40 against the influenza 2017 H7N9 vaccine strain at baseline and approximately 21 days after receipt of 1 dose of AS03-adjuvanted 2017 H7N9 IIV (Group 1–Day 1 (baseline) and Day 22; Group 2 –Day 22 (baseline) and Day 43; Group 3 N/A).
- GMTs of serum HAI and Neut antibodies against the influenza 2017 H7N9 vaccine virus at baseline and at approximately 21 days after receipt of 1 dose of AS03-adjuvanted 2017 H7N9 IIV. (Group 1–Day 1 (baseline) and Day 22; Group 2 –Day 22 (baseline) and Day 43; Group 3 N/A).

#### 3.2.3. Exploratory

#### Immunogenicity:

• For HAI and Neut antibodies, percentage of subjects achieving seroconversion, percentage with titer ≥1:40 and the GMTs against the 2017 H7N9 study vaccine strain approximately 21 and 180 days after 2 doses of adjuvanted 2017 H7N9 IIV, stratified by age, sex, BMI, and prior receipt of seasonal influenza vaccine(s) for Groups 1 and 2.

- For HAI and Neut antibodies, percentage of subjects achieving seroconversion, percentage with a titer ≥1:40 and the GMTs against the IIV4 vaccine strains approximately 21 and 180 days after receipt of IIV4, stratified by age, sex, BMI, and prior receipt of seasonal influenza vaccine(s).
- For HAI and Neut antibodies, percentage of subjects achieving seroconversion, percentage with titer ≥1:40, and GMTs against the 2017 H7N9 study vaccine strain at approximately 180 days after 2 doses of adjuvanted 2017 H7N9 IIV for Groups 1 and 2.
- Percentage of subjects with detectable levels of serum N1, N2 and N9 NA-specific antibody elicited by 2017 H7N9 and seasonal IIV4 vaccination, and the correlation of the NA content of 2017 H7N9 IIV and seasonal IIV4 with the elicited NA specific antibody responses at baseline and approximately 21 and 180 days after 2 doses of adjuvanted 2017 H7N9 IIV for Groups 1 and 2; and approximately 21 and 180 days after receipt of the seasonal IIV4 vaccine for all Groups. Note: analysis plans for this endpoint will be described in an addendum to this SAP once the NA assay has been selected

# 3.3. Study Definitions and Derived Variables

For individual subjects, fold rise will be calculated as the ratio of:  $\frac{post-vaccination\ titer}{pre-vaccination\ titer}$ , where pre-vaccination value is always the result obtained at Day 0, prior to the priming dose.

HAI Seroconversion is defined as either a pre-vaccination HAI titer <10 and a post-vaccination HAI titer  $\ge 40$  or a pre-vaccination HAI titer  $\ge 10$  and a minimum four-fold rise in post-vaccination HAI titer [5].

Neut Seroconversion is defined as either a pre-vaccination Neut titer <1:10 and a post-vaccination Neut titer  $\ge 1:40$  or a pre-vaccination Neut titer  $\ge 1:10$  and a minimum four-fold rise in post-vaccination Neut antibody titer.

#### 4. INVESTIGATIONAL PLAN

# 4.1. Overall Study Design and Plan

DMID Protocol 17-0077 follows a Phase II randomized, open-label study design enrolling males and non-pregnant females aged 19-64 years who are in good health as determined by medical history and physical examination, and meet all eligibility criteria, including erythrocyte sedimentation rate (ESR) and negative urine or serum pregnancy test (for females). This clinical trial is designed to assess the safety, reactogenicity, and immunogenicity of a pre-pandemic AS03 (GSK) adjuvanted 2017 monovalent inactivated influenza A/H7N9 vaccine (2017 H7N9 IIV) manufactured by Sanofi Pasteur (3.75 mcg of HA per dose), when two doses are administered 21 days apart either sequentially or simultaneously (within 15 minutes) with licensed seasonal influenza vaccine.

Subjects will be randomly assigned to 1 of 3 study groups with allocation 2:2:1 (see Table 1). All study doses will be administered IM approximately 21 days apart. Subjects assigned to treatment group 1 will receive seasonal IIV4 and AS03 adjuvanted 2017 H7N9 IIV concurrently at the first dose, and will return after approximately 21 days to receive a second dose of AS03 adjuvanted 2017 H7N9 IIV. Subjects assigned to treatment group 2 will receive seasonal IIV4 at the first dose followed by two doses at 21 and 42 days post IIV4 of AS03 adjuvanted 2017 H7N9 IIV. Subjects assigned to treatment group 3 will receive a single dose of IIV4.

Reactogenicity will be measured by the occurrence of solicited injection site and systemic reactions from the time of each study vaccination through 7 days after each study vaccination. Unsolicited non-serious AEs will be collected from the time of each study vaccination through approximately 21 days after each study vaccination. SAEs and MAAEs, including NOCMCs and PIMMCs, will be collected from the time of the first study vaccination through approximately 12 months after the last study vaccination. Clinical laboratory evaluations for safety will be performed on venous blood collected prior to each study vaccination and approximately 7 days after each study vaccination.

Immunogenicity testing will include performing HAI and Neut antibody assays against the 2017 H7N9 vaccine virus on serum samples collected for Group 1 on Days 1 (baseline), 22, and 43, and at approximately 180 days post second adjuvanted 2017 H7N9 IIV dose (Day 202), and for Group 2 on Study Days 22 (baseline), 43, and 64, and at approximately 180 days post second 2017 H7N9 IIV adjuvanted dose (Day 223). Serological antibody assays will be performed against the vaccine viruses in IIV4 from serum samples collected at baseline (Day 1) and approximately 21 and 180 days following receipt of seasonal IIV4 (Groups 1, 2, and 3).

Novel methods for identifying and assessing alternative correlates of protection against influenza infection are needed. To assess the NA-specific antibody response to vaccination, it is first necessary to determine the NA content of inactivated influenza vaccine; this assay is

under development. If successful, the NA content in a dosage-specific manner can be correlated to the N9 NA-specific antibody responses elicited by the 2017 H7N9 IIV.

# **4.2.** Discussion of Study Design, Including the Choice of Control Groups

This study uses a dose comparison concurrent control design. All subjects receive seasonal IIV4 vaccine either alone or administered simultaneously or sequentially with two doses of AS03 adjuvanted 2017 A/H7N9 IIV.

# **4.3.** Selection of Study Population

The study population for this clinical trial is 150 males and non-pregnant females, 19-64 years old, who are in good health and meet all eligibility criteria. The subjects will be recruited from the general population at the participating Vaccine Trial and Evaluation Unit (VTEU) sites that have substantial experience conducting large influenza vaccine studies.

#### 4.4. Treatments

#### 4.4.1. Treatments Administered

Seasonal IIV4 will be administered to all enrolled subjects. The 2017 A/H7N9 Vaccine with AS03 Adjuvant will be administered to subjects in treatment groups 1 and 2.

## 4.4.2. Identity of Investigational Product

See the study protocol for details of study product formulation.

# **4.4.3.** Method of Assigning Subjects to Treatment Groups (Randomization)

Enrollment/randomization will be performed through the enrollment module in the electronic data capture system maintained by the Statistical and Data Coordinating Center (SDCC).

Eligible subjects will be stratified by clinical site and randomly assigned with allocation (2:2:1) to 1 of 3 treatment groups indicated in Table 1. The treatment sequence was generated using permuted block randomization to provide an approximately balanced allocation to the treatment groups during the study.

### 4.4.4. Selection of Doses in the Study

Participants in this study are to receive one dose of seasonal IIV4 (all subjects), as well as two doses of AS03 adjuvanted 2017 A/H7N9 at HA dose of 3.75 mcg (treatment groups 1 and 2). The 3.75 mcg with AS03 dose was selected to evaluate safety and immunogenicity of antigen sparing dose strategies.

#### 4.4.5. Selection and Timing of Dose for Each Subject

Each subject is to be randomly assigned to a study group which will define the number and timing of AS03 adjuvanted 2017 A/H7N9 vaccinations. The first dose takes place on the day of randomization and will include vaccination with IIV4 for all subjects. Subjects in Group 1 will also receive the first A/H7N9 vaccination at the randomization visit. The second dose, a single A/H7N9 vaccination, if applicable, takes place approximately 21 days after the first dose (protocol defined window of 21-28 days post first dose). The third dose, a single A/H7N9 vaccination, if applicable, takes place approximately 21 days after the second dose (protocol defined window of 21-28 days post second dose).

## 4.4.6. Blinding

This trial is open-label. Subjects, investigators, and study personnel performing any study-related assessments following study vaccine administration are not blinded to study treatment. However, laboratory personnel performing HAI and Neut antibody assays will receive serum samples blinded to subject ID number and sample visit number.

The randomization scheme was generated by the SDCC and each subject's treatment assignment is displayed in AdvantageEDC upon enrollment.

The Data and Safety Monitoring Board (DSMB) may receive data in aggregate and presented by treatment group, including expected and observed rates of the expected AEs. The DSMB will review grouped data in the closed session only.

#### 4.4.7. Prior and Concomitant Therapy

Administration of any medications, therapies, or vaccines (including prescription and over-the-counter drugs as well as herbals, vitamins, and supplements) from 60 days prior to study vaccination through 21 days post final dose will be solicited from the participant during screening, enrollment, and follow-up. Any reported prior therapies from up to 30 days prior to vaccination through 21 days post final dose will be recorded in the appropriate data collection form.

Use of concomitant medications is allowed prior to and during the trial with the exception of medications and therapies that might interfere with the evaluation of the investigational product. Medications in this category include the prohibited medication per the Subject Exclusion Criteria (protocol Section 5.1.2). In addition, the site principal investigator or appropriate sub-investigator may identify other medications that should not be used due to a risk to subject safety or assessment of reactogenicity and immunogenicity.

#### 4.4.8. Treatment Compliance

All subjects are to receive one dose of seasonal IIV4 and subjects in treatment groups 1 and 2 are to receive two doses of AS03 adjuvanted 2017 A/H7N9 IIV vaccine administered in the clinic based on study group assignment.

## 4.5. Immunogenicity and Safety Variables

See Table 2, Table 3, Table 4, Table 5, Table 6, and Table 7 for schedules of study procedures by treatment group.

#### 4.5.1. Safety Variables

Safety will be assessed by the frequency and severity of:

- 1. SAEs occurring from the time of the first study vaccination through approximately 12 months after the last study vaccination.
- 2. Solicited AEs reactogenicity events occurring from the time of each study vaccination through 7 days after each study vaccination:
  - a) Injection site reactions including pruritus, ecchymosis, erythema, induration (hardness)/edema (swelling), pain, and tenderness.
  - b) Systemic reactions including fever, feverishness, fatigue, malaise, myalgia, arthralgia, headache, and nausea.
- 3. Clinical safety laboratory AEs occurring from the time of each study vaccination through approximately 7 days after each study vaccination. Parameters to be evaluated include white blood cells (WBC), hemoglobin (Hgb), platelets (PLT), alanine aminotransferase (ALT), total bilirubin (T. Bili), and creatinine (Cr).
- 4. Unsolicited AEs non-serious AEs occurring from the time of each study vaccination through approximately 21 days after each study vaccination.
- 5. MAAEs, including NOCMCs, and PIMMCs occurring from the time of the first study vaccination through approximately 12 months after the last study vaccination.

Grading scales for injection site and systemic solicited reactions, vital signs, and clinical laboratory parameters are provided in Table 13, Table 14, Table 15, and Table 16.

#### 4.5.2. Immunogenicity Variables

Individual HAI and Neut results will be reported by the central immunology laboratory for the homologous 2017 A/H7N9 vaccine strain, A/Hong Kong/125/2017, the homologous strains in the seasonal 2017/2018 IIV4 Fluzone vaccine (A/Michigan/45/2015 X-275 (H1N1), A/Hong Kong/4801/2014 X263B(H3N2), B/Phuket/3073/2013 (B Yamagata lineage), and B/Brisbane/60/2008 (B Victoria lineage)). Assay results are reported as a reciprocal titer with values of 10\*2<sup>k</sup>, where k=0, 1, 2, etc. The lower limit of detection for the HAI and Neut assays is 1:10; values below the limit of detection are reported as '<10', and for analysis are imputed as one-half the limit of detection (10/2 = 5). For analysis, the geometric mean (calculated on natural log scale) of repeated results for each sample will be computed and used as the response for all subsequent calculations. The variation arising from multiple measurements for an individual at a single time point is not used in subsequent calculations. See Section 3.3 for definitions of derived variables for the analysis of HAI and Neut data.

The assay to determine the influenza virus N9 Neuraminidase (NA) antibody response to vaccination is under development. An addendum to the SAP will be generated to outline the planned analyses when assay development is complete.

For subjects in Group 1 (Simultaneous Administration) there is potential for an overlap between the windows for Visit 9 (Day 181 post vaccination  $1 \pm 14$  days) and Visit 10 (Day 181 post vaccination  $2 \pm 14$  days). Should a subject complete both visits on the same date, HAI and Neut results against the seasonal IIV4 vaccine strains on that date will be associated with Visit 9, while HAI and Neut results against the 2017 H7N9 vaccine strain on that date will be associated with Visit 10.

All immunogenicity data will be uploaded into the SDCC's electronic data capture system.

#### 5. SAMPLE SIZE CONSIDERATIONS

This study is planned to enroll a minimum of 60 subjects in Groups 1-2, and 30 subjects in Group 3. This study is not designed to test a formal null hypothesis. Rather, it is intended to obtain sufficient data to obtain meaningful estimates of the immune response and to uncover any safety issues that occur at a sufficiently high rate that they might be observed in a study of this size. As such, the type one error rate, alpha = 0.05, is not adjusted for multiple comparisons. While this study is not designed to test any specific null hypothesis, the following tables illustrate the precision and power that is available for select estimates and comparisons of interest.

Table 8 indicates the probability of observing one or more safety events, such as solicited injection site or systemic reactogenicity events or an unsolicited non-serious AE of a particular type for a single treatment group (N = 30 or 60), and for all subjects receiving AS03-adjuvanted 2017 H7N9 IIV (N = 120).

Binomial confidence intervals (CI) are widest (have the least precision) when the response rate is 50%. Table 9 is presented to indicate the worst case scenario for precision of observed exact (Clopper-Pearson) binomial confidence intervals.

For each of the primary immunogenicity objective, a power analysis is provided below for testing the following hypotheses with the planned sample size, where  $p_c$  = proportion responders in comparator arm;  $p_e$  = proportion responders in experimental arm.

Test for difference in proportion responders:

 $H_0$ :  $p_c - p_e = 0$  – No difference in proportion responders

 $H_1$ :  $p_c - p_e \neq 0$  – difference in response rates

*Primary Immunogenicity Objective 1:* Evaluate antibody responses against A/H7N9 at approximately 21 days following receipt of two doses of AS03-adjuvanted 2017 H7N9 IIV. Comparison between simultaneous and sequential receipt to IIV4, i.e., Group 1 at Day 43 vs. Group 2 at Day 64.

*Primary Immunogenicity Objective 2:* Evaluate antibody responses against the seasonal influenza strains at approximately 21 days following receipt of IIV4.

Comparator Group (N = 75):

• Group 2 (IIV4/H7N9/H7N9) + Group 3 (IIV4) at Day 22

Experimental Groups (N = 50/group):

• Group 1 (IIV4+H7N9 /H7N9) at Day 64

Table 10 and Table 11 illustrate the minimum detectable differences in the proportion of subjects responding (e.g., attaining seroconversion or a titer  $\ge 1:40$ ) between two treatment groups using a two-sided Likelihood Ratio Test and alpha = 0.05.

#### 6. GENERAL STATISTICAL CONSIDERATIONS

# **6.1.** General Principles

All continuous variables will be summarized using the following descriptive statistics: n (non-missing sample size), mean, standard deviation, median, maximum and minimum. The frequency and percentages (based on the non-missing sample size) of observed levels will be reported for all categorical measures. In general, all data will be listed, sorted by site, treatment and subject, and when appropriate by visit number within subject. All summary tables will be structured with a column for each treatment group in the following order:

- Group 1: Simultaneous Administration (D1: IIV4/H7N9; D22: H7N9)
- Group 2: Sequential Administration (D1: IIV4; D22: H7N9; D43: H7N9)
- Group 3: IIV4 Only (D1: IIV4)

All tables will be annotated with the total population size relevant to that table/treatment, including any missing observations.

# **6.2.** Timing of Analyses

### 6.2.1. Preliminary Report and CSR

Clinical, safety, and reactogenicity data through Day 64 will represent the primary clinical database for this trial. Once the last subject completes the Day 64 visit, the primary clinical database will be cleaned, monitored, and locked. Analyses of safety, reactogenicity, and available immunogenicity (HAI and Neut antibody assays through day 64) data by treatment arm are planned. A preliminary report will be prepared by the SDCC after the primary clinical database is locked and all HAI and Neut data through 21 days after the last study vaccination are received. Immunogenicity and safety analyses will be presented in aggregate by treatment group; individual subject data will not be presented in the preliminary report. These analyses may be made available to the sponsor for planning subsequent trials and to the lead principal investigator for publication. These analyses will not be used to make any decisions concerning the conduct of this trial. All analyses of data included in the preliminary report for early release will be considered the final analysis of these data, and also included in the final CSR.

Tables and figures to be included in the Preliminary Report are indicated with the symbol \* in the title.

Analysis of exploratory immunogenicity endpoints may be performed and released as the data are available from the research laboratory. Any such analyses would be considered the final analysis for the endpoint, and included in the CSR.

The final CSR will be completed after the last subject's last visit is completed, and the final clinical database including all long-term safety follow-up data is cleaned, monitored and

locked. Additional exploratory immunogenicity endpoint data not available at the time of CSR preparation may be included in an addendum to the CSR.

# 6.3. Analysis Populations

#### **6.3.1.** Safety Population

The Safety Analysis population includes all subjects who received at least one study vaccination.

#### 6.3.2. Modified Intention-to-Treat (mITT) Population

The modified intent-to-treat (mITT) population includes all subjects who received at least one dose of study vaccine and contributed both pre- and at least one post-study vaccination venous blood samples for immunogenicity testing (HAI or Neut antibody assays) for which valid results were reported. For analyses using the mITT population, subjects in Group 2 who discontinue treatment after receiving the single IIV4 dose (Dose 1) but prior to receiving the first dose of the H7N9 vaccine (Dose 2) will be analyzed with group 3. All other subjects will be grouped based on randomized treatment group.

#### **6.3.3.** Per Protocol Population

The per protocol (PP) population includes all subjects in the mITT subset with the following exclusions:

- Data from all available visits for subjects found to be ineligible at baseline.
- Data from all visits subsequent to major protocol deviations, such as:
  - Second or third dose not received,
  - o Second or third dose received out of window,
  - Receipt of non-study licensed live vaccine within 30 days before or after each study vaccination,
  - o Receipt of non-study licensed inactivated vaccine within 14 days before or after each study vaccination,
  - Receipt of immunosuppressive therapy (e.g., corticosteroids) within 30 days before or after each study vaccination.
- Data from any visit that occurs out of window by more than one day.

For analyses using the PP population, subjects will be grouped based on study vaccinations received - subjects in Group 2 who discontinue treatment after receiving the single IIV4 dose (Dose 1) but prior to receiving the first dose of the H7N9 vaccine (Dose 2) will be analyzed with Group 3.

# 6.4. Covariates and Subgroups

As a protocol defined exploratory analysis, HAI antibody response following the second vaccination will be summarized stratified by the following covariates: age (categorical: 19-34, 35-49, 50-64), sex (male, female), body mass index (<30,  $\ge$ 30), and prior receipt of seasonal influenza vaccine(s) (received 2016-2017, did not receive 2016-2017, unknown), and these covariates will be considered in statistical modeling as described in Section 8.3. As these analyses are exploratory the study was not powered for any subgroup analyses.

## 6.5. Missing Data

All attempts will be made to collect all data per protocol. As missing data are expected to be minimal, no imputation will be performed for missing values. Any data point that appears to be erroneous or inexplicable based on clinical judgment will be investigated as a possible outlier. If data points are identified as outliers, sensitivity analyses will be performed to examine the impact of including or excluding the outliers. Any substantive differences in these analyses will be reported.

## 6.6. Interim Analyses and Data Monitoring

Interim analyses will only be used to terminate this trial in the event that unanticipated safety events deemed to be of sufficient concern require such action by the sponsor. These assessments will not be made on the basis of testing a formal statistical hypothesis; therefore, p-value adjustment will not be made to any analyses. A DSMB will be convened by DMID to review study progress and participant, clinical, safety, and reactogenicity and immunogenicity data.

A preliminary report of safety and immunogenicity data through Day 64 will be prepared as described in section protocol section 11.6; though this report will be released while subjects remain in the trial for long-term safety and immunogenicity follow-up, it will be considered the final analysis of these data.

Emergent public health needs may dictate additional interim safety, reactogenicity, and/or immunogenicity analyses be performed on available information at any time during the trial. If this occurs, immunogenicity data will be analyzed as results are available from the central immunogenicity laboratory.

#### **6.6.1.** Interim Safety Review

An interim safety review may include enrollment and demographic information, medical history, concomitant medications, physical assessments, clinical laboratory values, dosing compliance, and solicited and unsolicited AE/SAEs. Additional data may be requested by the DSMB, and interim statistical reports may be generated as deemed necessary and appropriate by DMID. The DSMB may receive data in aggregate and presented by treatment group. The DSMB may also be provided with expected and observed rates of the expected AEs by

treatment group, and may request the treatment assignment for an individual subject if required for safety assessment. The DSMB will review data grouped by treatment group in the closed session only. The DSMB will meet and review this data at scheduled time points or ad hoc as needed during this trial as defined in the DSMB charter. As an outcome of each review/meeting, the DSMB will make a recommendation as to the advisability of proceeding with study vaccinations (as applicable), and to continue, modify, or terminate this trial. Summaries prepared for the DSMB are defined separately in a report shell reviewed and approved by the DSMB.

Additionally, this trial will be monitored to determine if any of the halting rules described in Protocol Section 9.5 are met.

## 6.6.2. Interim Immunogenicity Review

No interim immunogenicity analysis is planned. Should emergent public health needs dictate immunogenicity review, immune responses will be summarized in terms of strain-specific 2017 A/H7N9 and IIV4 HAI and Neut antibody titers for subjects that receive sequential or simultaneous administration of AS03-adjuvanted 2017 H7N9 IIV and seasonal IIV4. It is anticipated that all analyses will be carried out in parallel for both assays, but reports may be prepared separately for HAI and Neuts if results are available on different timelines. Interim analyses will focus on rates of titers ≥1:40, seroconversion (see definition in Section 3.3) and GMTs, along with corresponding 95% CIs. No formal hypothesis testing will be included in the interim analysis, and interim results will not have impact on conduct of this trial.

Any immunogenicity reports would be provided by the SDCC to the DMID Scientific Lead and Clinical Project manager, and the DSMB. Reports will include data summarized by treatment group.

#### 6.7. Multicenter Studies

Randomization was stratified by site, but data will be pooled across all clinical sites for all analyses. Center effects are not anticipated because the sites use standardized procedures for vaccination and assessment of solicited and unsolicited AEs, and the study relies on a central laboratory for immunogenicity assessments.

# 6.8. Multiple Comparisons/Multiplicity

This study was designed to obtain preliminary estimates of safety and immune response to A/H7N9 and IIV4 vaccination in healthy adults. The study was not designed to test any specific null hypothesis, and as such no adjustment for multiple comparisons will be performed.

#### 7. STUDY SUBJECTS

# 7.1. Subject Disposition

Table 17 will present a summary of the reasons that subjects were screened but not enrolled.

The number and percentage of enrolled subjects excluded from each analysis population by treatment group are presented in Table 18. A listing of subjects excluded from each analysis population will be presented in Listing 5.

The disposition of subjects in the study will be tabulated by treatment group (Table 19). The table will show the total number of subjects screened, randomized, receiving the first dose, receiving the second dose, receiving the third dose, completing the blood draw for the primary immunogenicity endpoints, and completing the last visit.

A flowchart showing the disposition of study subjects, adapted from the CONSORT Statement [4] will be included and will present the number of subjects screened, randomized, lost to follow up, and analyzed, by treatment group (Figure 1).

A listing of subjects who were discontinued from treatment or terminated from study followup and the reason will be included in <u>Listing 2</u>.

#### 7.2. Protocol Deviations

A summary of subject-specific protocol deviations will be presented by the deviation category and deviation type, and treatment group for all enrolled subjects (Table 12). Major deviations that will be reviewed for possible exclusion of immunogenicity results from the PP population include deviations related to eligibility/enrollment, treatment administration schedule, follow-up visit schedule, and receipt of exclusionary vaccines or medications. All subject-specific protocol deviations and non subject-specific protocol deviations will be included in Listing 3 and Listing 4.

#### 8. IMMUNOGENICITY EVALUATION

Immunogenicity data summaries and analysis for primary and secondary endpoints will be presented for the mITT and PP populations. Immune responses in terms of strain-specific A/H7N9 HAI and Neut antibody titers will be summarized by treatment group at each time point. Descriptive summary statistics will be provided for all assays and time points including number of subjects with non-missing results, percentage of subjects with titers ≥1:40, percentage of subjects achieving seroconversion, and GMTs along with corresponding 95% CI. Exact confidence intervals will be presented for proportional endpoints. Summaries of primary and secondary immunogenicity endpoints are presented for the 2017 H7N9 strain in Table 28, Table 29, Table 30, and Table 31 and for the seasonal IIV4 strain in Table 32, Table 33, Table 34, and Table 35.

Reverse cumulative distribution (RCD) curves will be presented for post-vaccination HAI and Neut antibody titers. Plots for each assay will be generated with 5 panels (21 days post dose 1, 21 days post dose 2, 21 days post dose 3, 180 days post dose 1, and 180 days post final dose), and separate curves within each panel for each treatment group, as shown in Figure 2, Figure 3, Figure 4, and Figure 5 for the 2017 A/H7N9 strain. RCD curves for the IIV4 strains will be presented as in Figure 6, Figure 7, Figure 8, Figure 9, Figure 10, Figure 11, Figure 12, Figure 13, Figure 14, Figure 15, Figure 16, Figure 17, Figure 18, Figure 19, Figure 20, and Figure 21.

Figure 22, Figure 23, Figure 24, and Figure 25 for the 2017 A/H7N9 strain, and for the IIV4 strains in Figure 26, Figure 27, Figure 28, Figure 29, Figure 30, Figure 31, Figure 32, Figure 33, Figure 34, Figure 35, Figure 36, Figure 37, Figure 38, Figure 39, Figure 40, and Figure 41.

The spearman correlation between HAI and Neut antibody titers will be calculated at each time point over all groups. The correlation will be depicted in scatter plots as Figure 42 and Figure 43 for the 2017 A/H7N9 strain. Scatterplots depicting correlation for the IIV4 strains will be created as Figure 44, Figure 45, Figure 46, Figure 47, Figure 48, Figure 49, Figure 50, and Figure 51.

Individual HAI and Neut assay results will be provided in Listing 8.

# 8.1. Primary Immunogenicity Analysis

The primary immunogenicity endpoints HAI and Neut seroconversion, percentage of subjects with titer ≥1:40, and GMTs against the seasonal IIV4 strains 21 days after the IIV4 vaccination for all groups and against the homologous A/H7N9 vaccine strain 21 days after the second dose of AS03 adjuvanted 2017 H7N9 IIV will be summarized as described above. The primary analysis population will be mITT, with results from the PP population providing a comparison of the sensitivity of immunogenicity results to subject adherence to protocol-

defined conditions. Regression modelling of seroconversion and log titers is planned as described in Section 8.3.2.

## 8.2. Secondary Immunogenicity Analyses

The secondary immunogenicity endpoints HAI and Neut seroconversion, percentage of subjects with titer >40, and GMTs against the homologous A/H7N9 vaccine strain 21 days after the first AS03-adjuvanted 2017 H7N9 vaccination will be summarized as described above. No formal hypothesis testing is planned.

# 8.3. Exploratory Immunogenicity Analyses

Immunogenicity data summaries and analysis for exploratory endpoints will be presented for the PP populations.

#### 8.3.1. Covariate Analysis

As an exploratory analysis, seroconversion and GMT of serum antibody for both HAI and Neut against the homologous 2017 A/H7N9 strain at 21 and 180 days after the second dose of AS03 adjuvanted 2017 H7N9 IIV (treatment groups 1 and 2 only) will be summarized by treatment group stratified by age (categorized as those subjects ages 19-34, 34-49, and 50-64 years) (Table 36, Table 37, Table 38, and Table 39), by sex (Table 44, Table 45, Table 46, and Table 47), by BMI (Table 52, Table 53, Table 54, and Table 55), and by prior receipt of the 2016-2017 seasonal influenza vaccine (Table 60, Table 61, Table 62, and Table 63). These analyses will be repeated for HAI and Neut titer results against each of the four IIV4 vaccine strains at 21 and 180 days post receipt of seasonal IIV4 vaccine (by age category: Table 40, Table 41, Table 42, and Table 43; by sex: Table 48, Table 49, Table 50, and Table 51; by BMI: Table 56, Table 57, Table 58, and Table 59; by prior receipt of seasonal influenza vaccine: Table 64, Table 65, Table 66, and Table 67).

The stratified summaries will be presented for the PP population. For the 2017 A/H7N9 strain it is anticipated that subjects will have little to no pre-existing antibody at baseline, so seroconversion and titer  $\geq$ 40 endpoints will be similar.

#### **8.3.2.** Regression Modeling

Logistic and multivariate linear regression will be utilized to test for the effects of the treatment schedule on seroconversion and GMT against the homologous 2017 A/H7N9 strain and against each of the seasonal IIV4 strains for the PP population. Similar models will be fit for HAI and Neut Antibodies for each strain and time point. Separate models will be fit for data from Day 21 post dose and Day 180 post dose.

Logistic regression will be fit to examine the relationship of HAI or Neut seroconversion at 21 or 180 days after the dose of interest (second dose of AS03 adjuvanted A/H7N9 IIV for the 2017 A/H7N9 strain; IIV4 vaccination for the seasonal IIV4 strains) with treatment schedule. If the available titer data meets the required assumptions of normality after log

transformation, multiple linear regression will be fit to examine the relationship of log transformed titers at 21 or 180 days after the dose of interest (second dose of AS03 adjuvanted A/H7N9 IIV for the 2017 A/H7N9 strain; IIV4 vaccination for the seasonal IIV4 strains) with treatment schedule. All models will be fit with and without adjustment for the following covariates (Z): age in years, sex (female, male), BMI ( $<30, \ge 30$ ), and prior receipt of seasonal influenza vaccine (did not receive 2016-2017 seasonal vaccine, received 2016-2017 seasonal vaccine). The models as shown below assume a linear relationship between age in years and both probability of seroconversion and GMT. The validity of this assumption will be assessed prior to analysis and, if the relationship between age and response is found to be non-linear, adjustments will be made to model parameters to satisfy regression assumptions. Modeling assumptions will be checked using standard diagnostic methods (e.g., using the INFLUENCE option in PROC LOGISTIC or PROC GLM). Parameter estimates and odds ratio estimates for the logistic models will be presented for the 2017 A/H7N9 strain without covariate adjustment in Table 68, Table 69, Table 70, Table 71, and with covariate adjustment in Table 76, Table 77, Table 78, Table 79; and for the seasonal IIV4 strains without covariate adjustment in Table 72, Table 73, Table 74, Table 75, and with covariate adjustment in Table 80, Table 81, Table 82, Table 83. Parameter estimates for the multiple linear regression models will be presented for the 2017 A/H7N9 strain without covariate adjustment in Table 84, Table 85, Table 86, Table 87, and with covariate adjustment in Table 92, Table 93, Table 94, Table 95; and for the seasonal IIV4 strains without covariate adjustment in Table 88, Table 89, Table 90, Table 91, and with covariate adjustment in Table 96, Table 97, Table 98, Table 99.

Model 1A: Logistic Regression (without covariate adjustment):

 $logit[P(seroconversion)] = \beta_0 + \beta_1 \times Treatment + \varepsilon$ 

Model 1B: Logistic Regression (with covariate adjustment):

 $logit[P(seroconversion)] = \beta_0 + \beta_1 \times Treatment + \beta_2 \times Z + \varepsilon$ 

Model 2A: Multiple Linear Regression (without covariate adjustment):

 $log(titer) = \beta_0 + \beta_1 \times Treatment + \varepsilon$ 

Model 2B: Multiple Linear Regression (with covariate adjustment):

 $log(titer) = \beta_0 + \beta_1 \times Treatment + \beta_2 \times Z + \varepsilon$ 

Subjects missing data for one or more covariates will be excluded from Models 1B and 2B.

#### 8.3.3. NA Serum Antibody Responses

Descriptions of the NA assays and planned analyses will be described in an addendum to this SAP.

#### 9. SAFETY EVALUATION

All summaries and analysis of safety data will be presented for the Safety Analysis Population. Safety summaries will be presented overall and grouped by treatment group.

Continuous variables will be summarized using the following descriptive statistics: n (non-missing sample size), mean, standard deviation, median, maximum and minimum. All categorical measures will be summarized by the frequency and percentages of observed levels will be reported for all categorical measures. The denominator for the percentages may be based on the number of non-missing observations for an assessment or based on the number of subjects in a population. This will be described for each table.

# 9.1. Demographic and Other Baseline Characteristics

Summaries of age, sex, ethnicity, race, BMI, and prior receipt of seasonal influenza vaccine will be presented by site (Table 23, Table 24) and by treatment group (Table 25, Table 26). Age will be summarized as a continuous variable. Ethnicity is categorized as Hispanic or Latino, or not Hispanic and not Latino. In accordance with NIH reporting policy, subjects may self-designate as belonging to more than one race or may refuse to identify a race, the latter reflected in the electronic case report form (eCRF) as "No" to each racial option. BMI will be summarized as a continuous as well as categorical variable, categorized as (<30, ≥30). Self-reported history of prior receipt of seasonal influenza vaccine will be categorized as follows: received 2016-2017 seasonal vaccine, did not receive 2016-2017 seasonal vaccine, or unknown. Demographic information for individual subjects will be provided in Listing 6. Subjects' prior influenza vaccination history (seasonal and non-seasonal) will be provided in Listing 8.

#### 9.1.1. Prior and Concurrent Illnesses and Medical Conditions

All current illnesses and past or pre-existing medical conditions will be coded using Medical Dictionary for Regulatory Activities (MedDRA) version 20.0 or higher.

Summaries of subjects' prior and concurrent medical conditions will be presented by treatment group (Table 27).

Individual subject listings will be presented for all reported medical history including prior and concurrent medical conditions (Listing 7).

#### 9.1.2. Prior and Concurrent Medications

Concomitant medications will be coded to the Anatomical Therapeutic Classification using the WHO Drug Dictionary. The use of concomitant medications during the study will be summarized by ATC1 and ATC2 code and treatment group for the Safety population (Table 149). A listing of concomitant medications will be presented (Listing 17).

## 9.2. Measurements of Treatment Compliance

All subjects are to receive IIV4 vaccine on Study Day 1. Subjects in Group 1 (Simultaneous Administration) will also receive the first dose of 2017 A/H7N9 in the contralateral arm on Study Day 1, with the second dose of 2017 A/H7N9 administered 21 days later (Study Day 22). Subjects in Group 2 will have two doses of 2017 A/H7N9 vaccine administered 21 days apart (Study Days 22 and 43). Subjects in Group 3 will receive no further doses. The number of study vaccinations administered to subjects will be presented by treatment group and by site in Table 20, Table 21, Table 22, and as part of the subject disposition table (Table 19). Listing 1 presents subjects who received investigational product with randomized treatment group and study product received for each vaccination.

#### 9.3. Adverse Events

A summary of all adverse events is provided in Table 100. A summary of those events that occurred in  $\geq$ 5% of subjects in any treatment group is provided in Table 101.

## 9.3.1. Solicited Events and Symptoms

Systemic solicited adverse events were collected pre-vaccination, and systemic and local solicited adverse events were collected at-least 20 minutes post-vaccination and then daily for 7 days after each vaccination and graded on a scale of 0 (absent), 1 (mild), 2 (moderate) and 3 (severe). Systemic events include fever, feverishness, fatigue, malaise, myalgia, arthralgia, headache, and nausea. Local events include pruritus, ecchymosis, erythema, induration/swelling, pain, and tenderness. Ecchymosis, erythema, and induration are measured by both functional and measurement grading scales as defined in Table 13. The grading scale for systemic events, including quantitative grading for fever, is included in Table 14.

When calculating the incidence of solicited events, each subject will be counted once at the highest severity following the applicable vaccination, and any repetitions will be ignored. For summaries presented separately for each vaccination, the denominator for percentages will be the number of subjects who received the respective vaccination with non-missing data for the event summarized. For summaries over all vaccinations the denominator will be the number of subjects who received at least one vaccination with non-missing data for the event summarized.

The number and percentage of subjects reporting at least one solicited adverse event of each severity will be summarized for each solicited symptom, any systemic symptom, any local symptom, and any symptoms. For each event the denominator is the number of subjects who received the applicable vaccination with non-missing data for the specific event. The 95% CI calculated using Clopper-Pearson methodology from a binomial distribution (SAS Proc Freq with a binomial option) will be presented (Table 102, Table 103, Table 104, Table 105). Logistic regression models will be fit to estimate the effect of treatment schedule on the

probability of reporting any local event or reporting any systemic event (Table 106, Table 107). If statistically significant effects are observed in the model for local events or systemic events, then additional models will be fit for each individual event of that type.

$$logit[P(Event)] = \beta_0 + \beta_1 \times Treatment + \varepsilon,$$

For each systemic and local event, any systemic event, any local event, and any solicited event, the maximum severity over 7 days after each vaccination will be summarized for the Safety population. The number and percentage of subjects reporting each event will be summarized by the maximum severity and treatment group, separately for each dose and over all doses. For each event the denominator is the number of subjects who received the applicable vaccination with non-missing data for the specific event. The 95% CI calculated using Clopper-Pearson methodology from a binomial distribution (SAS Proc Freq with a binomial option) will be presented (Table 108, Table 109, Table 110, Table 111).

The number of subjects reporting a solicited adverse event will be summarized for each day post vaccination for each vaccination and for all vaccinations combined both in a summary table (Table 112, Table 113, Table 114, Table 115) and graphically in a bar chart (Figure 52 and Figure 53). A comparison of the event rate for each treatment group between study vaccinations will be presented for those groups receiving multiple vaccinations, including p-values from McNemar's test performed (Table 116, Table 117).

Systemic and Local solicited events reported by subject will be presented in Listing 10 and Listing 11, sorted by subject ID, vaccination number, parameter, and study day.

#### 9.3.2. Unsolicited Adverse Events

When calculating the incidence of unsolicited AEs (i.e., on a per subject basis), each subject will only be counted once at the highest severity and/or relationship, and any repetitions of AEs within a subject will be ignored; the denominator will be the total number of subjects in the safety population. All AEs reported will be included in the summaries and analyses.

The number and percentage of subjects reporting at least one unsolicited AE will be summarized by MedDRA system organ class and preferred term. A 95% CI will be presented for the percentage of subjects reporting any unsolicited AE (serious or non-serious) for each MedDRA system organ class and preferred term over all study vaccinations (Table 118).

The following summaries for unsolicited AEs will be presented by MedDRA system organ class, preferred term, and treatment group:

- Incidence of AEs by severity and relationship to study product (Table 119);
- Incidence of non-serious, related AEs by severity (Table 120);
- Incidence of AEs over time (Days 1-8, Days 9-22 post each study vaccination) (Table 121);

- Incidence of non-serious, related AEs over time (Days 1-8, Days 9-22 post each study vaccination) (Table 122) note this table presents results for secondary safety endpoint, "Occurrence of study vaccine-related unsolicited non-serious AEs from the time of each study vaccination through approximately 21 days after each study vaccination";
- Total frequency of AEs over time (Days 1-8, Days 9-22 post each study vaccination) (Table 123);
- Subject listing of non-serious AEs of moderate or greater severity (Table 128);
- Bar chart displaying total frequency of AEs by severity and MedDRA system organ class and treatment group (Figure 54);
- Bar chart displaying incidence of AEs by severity and MedDRA system organ class, and treatment group (Figure 55);
- Bar chart displaying total frequency and incidence of AEs by relationship to study product, MedDRA system organ class, and treatment group (Figure 56 and Figure 57).

# 9.4. Deaths, Serious Adverse Events and other Significant Adverse Events

The following listings will be presented including Subject ID, Age (years) AE Description, AE Onset Date/End Date, Last Vaccination Received/Days Post Vaccination, Reason Reported as an SAE, Relationship to Treatment, Alternate Etiology if not Related, Outcome, and Duration of Event (days):

- Deaths and Serious Adverse Events (Table 124);
- Medically Attended Adverse Events (Table 125);
- Potentially Immune Mediated Medical Conditions (Table 126);
- New Onset Chronic Medical Conditions (Table 127).

A listing of all reported AEs by subject will be presented in Listing 12, sorted by Treatment group, Subject ID, and AE Number.

# 9.5. Pregnancies

For any subjects in the Safety population who became pregnant during the study, every attempt will be made to follow these subjects to completion of pregnancy to document the outcome, including information regarding any complications with pregnancy and/or delivery.

Listing 18, Listing 19, Listing 20, Listing 21, and Listing 22 will present any study pregnancies and their outcomes.

# 9.6. Clinical Laboratory Evaluations

Clinical safety laboratory parameters (WBC, Hgb, PLT, ALT, T. Bili, Cr) will be collected from each subject prior to each study vaccination and approximately 7 days after each study vaccination. These evaluations will be performed by the central clinical laboratory. The grading scale for clinical laboratory evaluations is presented in Table 16. Clinical laboratory evaluations assessed on Day 1 prior to the first study vaccination will be considered as baseline.

The distribution of laboratory results by severity, study day and treatment group will be presented in Table 129, Table 130, Table 131, Table 132, Table 133, Table 134, and Table 135. Descriptive statistics including mean, standard deviation, median, minimum and maximum values and change from baseline by study day will be summarized for each parameter in Table 136, Table 137, Table 138, Table 139, Table 140, Table 141. Box plots illustrating the change from baseline for each laboratory parameter will be presented in Figure 58, Figure 59, Figure 60, Figure 61, Figure 62, and Figure 63. Subject visits with abnormal laboratory results, Grade 1 severity or higher, will be presented in Table 142 and Table 143 for Chemistry and Hematology parameters, respectively.

A complete listing of individual clinical laboratory results will be presented in Listing 13 and Listing 14 for chemistry and hematology, respectively, sorted by subject ID, parameter, and visit number.

# 9.7. Vital Signs and Physical Evaluations

Vital signs oral temperature, systolic blood pressure, diastolic blood pressure, and pulse will be assessed prior to study vaccination on Day 1 and Day 22. The grading scale for vital sign evaluations is presented in Table 15. Summaries of vital signs by maximum severity will be tabulated by visit, and treatment group (Table 144, Table 145, Table 146, Table 147, Table 148). A listing of vital signs will be presented (Listing 15).

Targeted physical examinations will be performed, if indicated, based a subject's medical history. A listing of physical exam findings will be presented (Listing 16).

#### 9.8. Concomitant Medications

Concomitant medications will be collected for the 30 days prior to the first study vaccination through 21 days after the second study vaccination. Concomitant medications will be coded to the Anatomical Therapeutic Classification using the WHO Drug Dictionary. The use of prior and concomitant medications taken during the study will be recorded on the CRFs. A by-subject listing of concomitant medication use will be presented (Listing 17). The use of concomitant medications during the study will be summarized by ATC1, ATC2 code, treatment group for the Safety population (Table 149).

#### 10. REPORTING CONVENTIONS

P-values ≥0.001 and ≤0.999 will be reported to 3 decimal places; p-values less than 0.001 will be reported as "<0.001"; p-values greater than 0.999 will be reported as "> 0.999". The mean, standard deviation, and any other statistics other than quantiles, will be reported to one decimal place greater than the original data. Quantiles, such as median, or minimum and maximum will use the same number of decimal places as the original data. Proportions will be presented as two decimal places; values <0.01 will be presented as "<0.01". Percentages will be reported to the nearest whole number; non-zero values < 1% will be presented as "<1"; values greater than 99% but less than 100% will be presented as >99. Estimated parameters, not on the same scale as raw observations (e.g. regression coefficients) will be reported to 3 significant figures.

# 11. TECHNICAL DETAILS

SAS version 9.4 or above will be used to generate all tables, figures and listings.

# 12. SUMMARY OF CHANGES IN THE CONDUCT OF THE STUDY OR PLANNED ANALYSES

This SAP does not include any changes from the analyses described in the protocol.

# 13. REFERENCES

- 1. Gao, R., et al., *Human infection with a novel avian-origin influenza A (H7N9) virus.* N Engl J Med, 2013. **368**(20): p. 1888-97.
- 2. Analysis of recent scientific information on avian influenza A(H7N9) virus. WHO Influenza Update, 2017.
- 3. Human infection with avian influenza A(H7N9) virus China: 18 May 2017. WHO Emergencies preparedness, response, 2017.
- 4. Drummond R. CONSORT Revised: Improving the Reporting of Randomized Clinical Trials. JAMA. 2001; 285(15):2006-2007.
- 5. FDA Guidance for Industry: Clinical Data Needed to Support the Licensure of Seasonal Inactivated Influenza Vaccines (US DHHS, FDA, CBER, May 2007).
## 14. APPENDICES

Table, figure, and listing shells are presented in Appendices 1, 2, and 3. Tables and figures included in the Preliminary Report are indicated by \*.

# **Appendix 1. TABLE MOCK-UPS**

## LIST OF TABLES

| Table 1: | Study Design | 39 |
|---|---|---|
| Table 2: | Schedule of Study Procedures – Group 1: Vaccination Period | 40 |
| Table 3: | Schedule of Study Procedures – Group 1: Follow-Up Period (Including early | |
| | termination and unscheduled visits) | 43 |
| Table 4: | Schedule of Study Procedures – Group 2: Vaccination Period | |
| Table 5: | Schedule of Study Procedures – Group 2: Follow-Up Period (Including early | |
| | termination and unscheduled visits) | 48 |
| Table 6: | Schedule of Study Procedures – Group 3: Vaccination and Follow-up Periods | |
| Table 7: | Schedule of Study Procedures – Group 3: Early Termination and Unscheduled Vis | |
| Table 8: | Power (%) to Detect Safety Events | 53 |
| Table 9: | Precisions of Binomial Confidence Intervals | 53 |
| Table 10: | Objective 1 - Minimum Detectable Difference in Proportion Responders with 80% | |
| | Power (N = 50 per group) | 53 |
| Table 11: | Objective 2 - Minimum Detectable Difference in Proportion Responders with 80% | |
| | Power | |
| Table 12: | Distribution of Protocol Deviations by Category, Type and Treatment Group, All | |
| | Enrolled Subjects | |
| Table 13: | Solicited Adverse Event Grading Scale – Local | 57 |
| Table 14: | Solicited Adverse Event Grading Scale - Systemic | 58 |
| Table 15: | Vital Signs Adverse Event Grading Scale | 59 |
| Table 16: | Laboratory Adverse Event Grading Scale | |
| Table 17: | Ineligibility Summary of Screen Failures* | |
| Table 18: | Analysis Populations by Treatment Group – All Enrolled Subjects* | 62 |
| Table 19: | Subject Disposition by Treatment Group, All Enrolled Subjects* | 66 |
| Table 20: | Dates of First Dose by Site and Treatment Group for the Safety Analysis Populatio | n67 |
| Table 21: | Dates of Second Dose by Site and Treatment Group for the Safety Analysis | |
| | Population | |
| Table 22: | Dates of Third Dose by Site and Treatment Group for the Safety Analysis Population | |
| | | 67 |
| Table 23: | Summary of Categorical Demographic and Baseline Characteristics by Site, All | |
| | Enrolled Subjects | 68 |
| Table 24: | Summary of Continuous Demographic and Baseline Characteristics by Site, All | |
| | Enrolled Subjects | 69 |
| Table 25: | Summary of Categorical Demographic and Baseline Characteristics by Treatment | |
| | Group, All Enrolled Subjects* | 70 |
| Table 26: | Summary of Continuous Baseline Characteristics by Treatment Group, All Enrolle | |
| | Subjects* | 71 |
| Table 27: | Summary of Subjects with Prior or Concurrent Medical Conditions by MedDRA® | |
| | System Organ Class and Treatment Group, Safety Analysis Population | |
| Table 28: | Summaries of Hemagglutination Inhibition Antibody Against 2017 A/H7N9 by Stu | |
| | Day and Treatment Group, Modified Intent-to-Treat Population* | |
| Table 29: | Summaries of Hemagglutination Inhibition Antibody Against 2017 A/H7N9 by Stu | |
| | Day and Treatment Group, Per Protocol Population* | 74 |

| Table 30: | Summaries of Neutralizing Antibody Against 2017 A/H7N9 by Study Day and Treatment Group, Modified Intent-to-Treat Population* |
|---|---|
| Table 31: | Summaries of Neutralizing Antibody Against 2017 A/H7N9 by Study Day and Treatment Group, Per Protocol Population*74 |
| Table 32: | Summaries of Hemagglutination Inhibition Antibody Against Seasonal IIV4 Strains |
| 14010 32. | by Study Day and Treatment Group, Modified Intent-to-Treat Population* |
| Table 33: | Summaries of Hemagglutination Inhibition Antibody Against Seasonal IIV4 Strains |
| 14010 33. | by Study Day and Treatment Group, Per Protocol Population* |
| Table 34: | Summaries of Neutralizing Antibody Against Seasonal IIV4 Strains by Study Day and |
| 1 abic 34. | Treatment Group, Modified Intent-to-Treat Population* |
| Table 35: | Summaries of Neutralizing Antibody Against Seasonal IIV4 Strains by Study Day and |
| 1 4010 33. | Treatment Group, Per Protocol Population* |
| Table 36: | Summary of Hemagglutination Inhibition Antibody Against 2017 A/H7N9 by |
| 14010 30. | Treatment Group and Age Group at 21 Days Post Second Dose of AS03 adjuvanted |
| | A/H7N9 Vaccine, Per-Protocol Population*78 |
| Table 37: | Summary of Hemagglutination Inhibition Antibody Against 2017 A/H7N9 by |
| 1 4010 57. | Treatment Group and Age Group at 180 Days Post Second Dose of AS03 adjuvanted |
| | A/H7N9 Vaccine, Per-Protocol Population |
| Table 38: | Summary of Neutralizing Antibody Against 2017 A/H7N9 by Treatment Group and |
| 14010 30. | Age Group at 21 Days Post Second Dose of AS03 adjuvanted A/H7N9 Vaccine, Per- |
| | Protocol Population* |
| Table 39: | Summary of Neutralizing Antibody Against 2017 A/H7N9 by Treatment Group and |
| 1 4010 37. | Age Group at 180 Days Post Second Dose of AS03 adjuvanted A/H7N9 Vaccine, Per- |
| | Protocol Population |
| Table 40: | Summary of Hemagglutination Inhibition Antibody Against Seasonal IIV4 Strains by |
| rable to. | Treatment Group and Age Group at 21 Days Post IIV4, Per-Protocol Population* 79 |
| Table 41: | Summary of Hemagglutination Inhibition Antibody Against Seasonal IIV4 Strains by |
| 14610 .11 | Treatment Group and Age Group at 180 Days Post Second Dose of AS03 adjuvanted |
| | A/H7N9 Vaccine, Per-Protocol Population |
| Table 42: | Summary of Neutralizing Antibody Against Seasonal IIV4 Strains by Treatment |
| | Group and Age Group at 21 Days Post Second Dose of AS03 adjuvanted A/H7N9 |
| | Vaccine, Per-Protocol Population*80 |
| Table 43: | Summary of Neutralizing Antibody Against Seasonal IIV4 Strains by Treatment |
| | Group and Age Group at 180 Days Post Second Dose of AS03 adjuvanted A/H7N9 |
| | Vaccine, Per-Protocol Population80 |
| Table 44: | Summary of Hemagglutination Inhibition Antibody Against 2017 A/H7N9 by |
| | Treatment Group and Sex at 21 Days Post Second Dose of AS03 adjuvanted A/H7N9 |
| | Vaccine, Per-Protocol Population* |
| Table 45: | Summary of Hemagglutination Inhibition Antibody Against 2017 A/H7N9 by |
| | Treatment Group and Sex at 180 Days Post Second Dose of AS03 adjuvanted |
| | A/H7N9 Vaccine, Per-Protocol Population81 |
| Table 46: | Summary of Neutralizing Antibody Against 2017 A/H7N9 by Treatment Group and |
| | Sex at 21 Days Post Second Dose of AS03 adjuvanted A/H7N9 Vaccine, Per-Protocol |
| | Population* |
| Table 47: | Summary of Neutralizing Antibody Against 2017 A/H7N9 by Treatment Group and |
| | Sex at 180 Days Post Second Dose of AS03 adjuvanted A/H7N9 Vaccine, Per- |
| | Protocol Population81 |
| Table 48: | Summary of Hemagglutination Inhibition Antibody Against Seasonal IIV4 Strains by |
| | Treatment Group and Sex at 21 Days Post IIV4 Vaccination, Per-Protocol Population* |
| | 82 |

| Table 49: | Summary of Hemagglutination Inhibition Antibody Against Seasonal IIV4 Strains by Treatment Group and Sex at 180 Days Post IIV4 Vaccination, Per-Protocol Population |
|---|---|
| Table 50: | Summary of Neutralizing Antibody Against Seasonal IIV4 Strains by Treatment Group and Sex at 21 Days Post IIV4 Vaccination, Per-Protocol Population* |
| Table 51: | Summary of Neutralizing Antibody Against Seasonal IIV4 Strains by Treatment Group and Sex at 180 Days Post IIV4 Vaccination, Per-Protocol Population |
| Table 52: | Summary of Hemagglutination Inhibition Antibody Against 2017 A/H7N9 by Treatment Group and BMI at 21 Days Post Second Dose of AS03 adjuvanted A/H7N9 Vaccine, Per-Protocol Population* |
| Table 53: | Summary of Hemagglutination Inhibition Antibody Against 2017 A/H7N9 by Treatment Group and BMI at 180 Days Post Second Dose of AS03 adjuvanted A/H7N9 Vaccine, Per-Protocol Population |
| Table 54: | Summary of Neutralizing Antibody Against 2017 A/H7N9 by Treatment Group and BMI at 21 Days Post Second Dose of AS03 adjuvanted A/H7N9 Vaccine, Per-Protocol Population* |
| Table 55: | Summary of Neutralizing Antibody Against 2017 A/H7N9 by Treatment Group and BMI at 180 Days Post Second Dose of AS03 adjuvanted A/H7N9 Vaccine, Per-Protocol Population |
| Table 56: | Summary of Hemagglutination Inhibition Antibody Against Seasonal IIV4 Strains by Treatment Group and BMI at 21 Days Post IIV4 Vaccination, Per-Protocol Population* |
| Table 57: | Summary of Hemagglutination Inhibition Antibody Against Seasonal IIV4 Strains by Treatment Group and BMI at 180 Days Post IIV4 Vaccination, Per-Protocol Population |
| Table 58: | Summary of Neutralizing Antibody Against Seasonal IIV4 Strains by Treatment Group and BMI at 21 Days Post IIV4 Vaccination, Per-Protocol Population* |
| Table 59: | Summary of Neutralizing Antibody Against Seasonal IIV4 Strains by Treatment Group and BMI at 180 Days Post IIV4 Vaccination, Per-Protocol Population |
| Table 60: | Summary of Hemagglutination Inhibition Antibody Against 2017 A/H7N9 by Treatment Group and Prior Seasonal Influenza Vaccination at 21 Days Post Second Dose of AS03 adjuvanted A/H7N9 Vaccine, Per-Protocol Population* |
| Table 61: | Summary of Hemagglutination Inhibition Antibody Against 2017 A/H7N9 by Treatment Group and Prior Seasonal Influenza Vaccination at 180 Days Post Second Dose of AS03 adjuvanted A/H7N9 Vaccine, Per-Protocol Population |
| Table 62: | Summary of Neutralizing Antibody Against 2017 A/H7N9 by Treatment Group and Prior Seasonal Influenza Vaccination at 21 Days Post Second Dose of AS03 adjuvanted A/H7N9 Vaccine, Per-Protocol Population* |
| Table 63: | Summary of Neutralizing Antibody Against 2017 A/H7N9 by Treatment Group and Prior Seasonal Influenza Vaccination at 180 Days Post Second Dose of AS03 adjuvanted A/H7N9 Vaccine, Per-Protocol Population |
| Table 64: | Summary of Hemagglutination Inhibition Antibody Against Seasonal IIV4 Strains by Treatment Group and Prior Seasonal Influenza Vaccination at 21 Days Post IIV4 Vaccination, Per-Protocol Population* |
| Table 65: | Summary of Hemagglutination Inhibition Antibody Against Seasonal IIV4 Strains by Treatment Group and Prior Seasonal Influenza Vaccination at 180 Days Post IIV4 Vaccination, Per-Protocol Population |
| Table 66: | Summary of Neutralizing Antibody Against Seasonal IIV4 Strains by Treatment Group and Prior Seasonal Influenza Vaccination at 21 Days Post IIV4 Vaccination, Per-Protocol Population* |

| Table 67: | Summary of Neutralizing Antibody Against Seasonal IIV4 Strains by Treatment Group and Prior Seasonal Influenza Vaccination at 180 Days Post IIV4 Vaccination, |
|---|---|
| | Per-Protocol Population 89 |
| Table 68: | Logistic Regression Model to Evaluate the Relationship of Administration Schedule with HAI Seroconversion Against 2017 A/H7N9 at 21 Days post Second Dose of |
| | AS03 adjuvanted A/H7N9 Vaccine, Per Protocol Population*90 |
| Table 69: | Logistic Regression Model to Evaluate the Relationship of Administration Schedule with HAI Seroconversion Against 2017 A/H7N9 at 180 Days Post Second Dose of |
| T 11 70 | AS03 adjuvanted A/H7N9 Vaccine, Per Protocol Population * |
| Table 70: | Logistic Regression Model to Evaluate the Relationship of Administration Schedule with Neut Seroconversion Against 2017 A/H7N9 at 21 Days Post Second Dose of |
| T.1.1. 71. | AS03 adjuvanted A/H7N9 Vaccine, Per Protocol Population |
| Table 71: | Logistic Regression Model to Evaluate the Relationship of Administration Schedule with Neut Seroconversion Against 2017 A/H7N9 at 180 Days Post Second Dose of |
| T 11 70 | AS03 adjuvanted A/H7N9 Vaccine, Per Protocol Population |
| Table 72: | Logistic Regression Model to Evaluate the Relationship of Administration Schedule with HAI Seroconversion Against Seasonal IIV4 Strains at 21 Days post IIV4 |
| T 11 72 | Vaccination, Per Protocol Population* 91 |
| Table 73: | Logistic Regression Model to Evaluate the Relationship of Administration Schedule with HAI Seroconversion Against Seasonal IIV4 Strains at 180 Days Post IIV4 |
| T 11 74 | Vaccination, Per Protocol Population 91 |
| Table 74: | Logistic Regression Model to Evaluate the Relationship of Administration Schedule with Neut Seroconversion Against Seasonal IIV4 Strains at 21 Days Post IIV4 |
| T 11 75 | Vaccination, Per Protocol Population* |
| Table 75: | Logistic Regression Model to Evaluate the Relationship of Administration Schedule with Neut Seroconversion Against Seasonal IIV4 Strains at 180 Days Post IIV4 |
| T 11 76 | Vaccination, Per Protocol Population 91 |
| Table 76: | Logistic Regression Model to Evaluate the Relationship of Administration Schedule |
| | with HAI Seroconversion Against 2017 A/H7N9 at 21 Days Post Second Dose of |
| | AS03 adjuvanted A/H7N9 Vaccine, Adjusted for Baseline Covariates, Per Protocol |
| T-1.1. 77. | Population* 92 |
| Table 77: | Logistic Regression Model to Evaluate the Relationship of Administration Schedule |
| | with HAI Seroconversion Against 2017 A/H7N9 at 180 Days Post Second Dose of |
| | AS03 adjuvanted A/H7N9 Vaccine, Adjusted for Baseline Covariates, Per Protocol |
| Table 78: | Population |
| Table 76. | with Neut Seroconversion Against 2017 A/H7N9 at 21 Days Post Second Dose of |
| | AS03 adjuvanted A/H7N9 Vaccine, Adjusted for Baseline Covariates, Per Protocol |
| | Population* |
| Table 79: | Logistic Regression Model to Evaluate the Relationship of Administration Schedule |
| Table 19. | with Neut Seroconversion Against 2017 A/H7N9 at 180 Days Post Second Dose of |
| | AS03 adjuvanted A/H7N9 Vaccine, Adjusted for Baseline Covariates, Per Protocol |
| | Population |
| Table 80: | Logistic Regression Model to Evaluate the Relationship of Administration Schedule |
| 1 4010 00. | with HAI Seroconversion Against Seasonal IIV4 Strains at 21 Days Post IIV4 |
| | Vaccination, Adjusted for Baseline Covariates, Per Protocol Population* |
| Table 81: | Logistic Regression Model to Evaluate the Relationship of Administration Schedule with HAI Seroconversion Against Seasonal IIV4 Strains at 180 Days Post IIV4 |
| | Vaccination, Adjusted for Baseline Covariates, Per Protocol Population |

| Table 82: | Logistic Regression Model to Evaluate the Relationship of Administration Schedule |
|---|---|
| | with Neut Seroconversion Against Seasonal IIV4 Strains at 21 Days Post IIV4 |
| | Vaccination, Adjusted for Baseline Covariates, Per Protocol Population*95 |
| Table 83: | Logistic Regression Model to Evaluate the Relationship of Administration Schedule |
| | with Neut Seroconversion Against Seasonal IIV4 Strains at 180 Days Post IIV4 |
| | Vaccination, Adjusted for Baseline Covariates, Per Protocol Population95 |
| Table 84: | Multiple Linear Regression Model to Evaluate the Relationship of Administration |
| | Schedule with Log-Adjusted HAI Titer against 2017 A/H7N9 at 21 Days Post Second |
| | Dose of AS03 adjuvanted A/H7N9 Vaccine, Per Protocol Population*96 |
| Table 85: | Multiple Linear Regression Model to Evaluate the Relationship of Administration |
| | Schedule with Log-Adjusted HAI Titer against 2017 A/H7N9 at 180 Days Post |
| | Second Dose of AS03 adjuvanted A/H7N9 Vaccine, Per Protocol Population96 |
| Table 86: | Multiple Linear Regression Model to Evaluate the Relationship of Administration |
| | Schedule with Log-Adjusted Neut Titer against 2017 A/H7N9 at 21 Days Post Second |
| | Dose of AS03 adjuvanted A/H7N9 Vaccine, Per Protocol Population*96 |
| Table 87: | Multiple Linear Regression Model to Evaluate the Relationship of Administration |
| | Schedule with Log-Adjusted Neut Titer against 2017 A/H7N9 at 180 Days Post |
| | Second Dose of AS03 adjuvanted A/H7N9 Vaccine, Per Protocol Population96 |
| Table 88: | Multiple Linear Regression Model to Evaluate the Relationship of Administration |
| | Schedule with Log-Adjusted HAI Titer against Seasonal IIV4 Strains at 21 Days Post |
| | IIV4 Vaccination, Per Protocol Population* |
| Table 89: | Multiple Linear Regression Model to Evaluate the Relationship of Administration |
| | Schedule with Log-Adjusted HAI Titer against Seasonal IIV4 Strains at 180 Days |
| | Post IIV4 Vaccination, Per Protocol Population |
| Table 90: | Multiple Linear Regression Model to Evaluate the Relationship of Administration |
| | Schedule with Log-Adjusted Neut Titer against Seasonal IIV4 Strains at 21 Days Post |
| | IIV4 Vaccination, Per Protocol Population* |
| Table 91: | Multiple Linear Regression Model to Evaluate the Relationship of Administration |
| | Schedule with Log-Adjusted Neut Titer against Seasonal IIV4 Strains at 180 Days |
| | Post IIV4 Vaccination, Per Protocol Population |
| Table 92: | Multiple Linear Regression Model to Evaluate the Relationship of Administration |
| | Schedule with Log-Adjusted HAI Titer against 2017 A/H7N9 at 21 Days Post Second |
| | Dose of AS03 adjuvanted A/H7N9 Vaccine, Adjusted for Baseline Covariates, Per |
| | Protocol Population*98 |
| Table 93: | Multiple Linear Regression Model to Evaluate the Relationship of Administration |
| | Schedule with Log-Adjusted HAI Titer at 180 Days Post Second Dose of AS03 |
| | adjuvanted A/H7N9 Vaccine, Adjusted for Baseline Covariates, Per Protocol |
| | Population 98 |
| Table 94: | Multiple Linear Regression Model to Evaluate the Relationship of Administration |
| - | Schedule with Log-Adjusted Neut Titer at 21 Days Post Second Dose of AS03 |
| | adjuvanted A/H7N9 Vaccine, Adjusted for Baseline Covariates, Per Protocol |
| | Population* |
| Table 95: | Multiple Linear Regression Model to Evaluate the Relationship of Administration |
| 10010 701 | Schedule with Log-Adjusted Neut Titer at 180 Days Post Second Dose of AS03 |
| | adjuvanted A/H7N9 Vaccine, Adjusted for Baseline Covariates, Per Protocol |
| | Population |
| Table 96: | Multiple Linear Regression Model to Evaluate the Relationship of Administration |
| 1.010 / 0. | Schedule with Log-Adjusted HAI Titer against Seasonal IIV4 Strains at 21 Days Post |
| | IIV4 Vaccination, Adjusted for Baseline Covariates, Per Protocol Population*99 |
| | , , = ================================ |

| Table 97: | Multiple Linear Regression Model to Evaluate the Relationship of Administration<br>Schedule with Log-Adjusted HAI Titer against Seasonal IIV4 Strains at 180 Days |
|---|---|
| Table 98: | Post IIV4 Vaccination, Adjusted for Baseline Covariates, Per Protocol Population. 100 Multiple Linear Regression Model to Evaluate the Relationship of Administration Schedule with Log-Adjusted Neut Titer against Seasonal IIV4 Strains at 21 Days Post IIV4 Vaccination, Adjusted for Baseline Covariates, Per Protocol Population 100 |
| Table 99: | Multiple Linear Regression Model to Evaluate the Relationship of Administration<br>Schedule with Log-Adjusted Neut Titer against Seasonal IIV4 Strains at 180 Days<br>Post IIV4 Vaccination, Adjusted for Baseline Covariates, Per Protocol Population. 100 |
| Table 100: | Overall Summary of Adverse Events, Safety Population*101 |
| Table 101: | Number of Adverse Events Occurring in 5% of Subjects in Any Treatment Group by MedDRA® System Organ Class and Preferred Term, and Treatment Group - Safety Population |
| Table 102: | Number and Percentage of Subjects Experiencing Solicited Events with 95% Confidence Intervals by Symptom and Treatment Group (Safety Population) – Post Any Study Dose* |
| Table 103: | Number and Percentage of Subjects Experiencing Solicited Events with 95% Confidence Intervals by Symptom and Treatment Group (Safety Population) – Post |
| m 11 104 | Study Dose 1* |
| Table 104: | Number and Percentage of Subjects Experiencing Solicited Events with 95% |
| | Confidence Intervals by Symptom and Treatment Group (Safety Population) – Post |
| Talala 105. | Study Dose 2* |
| Table 105: | Number and Percentage of Subjects Experiencing Solicited Events with 95% Confidence Intervals by Symptom and Treatment Group (Safety Population) – Post Study Dose 3* |
| Table 106: | Logistic Regression Model to Evaluate the Relationship of Treatment with Reporting |
| 14010 100. | Any Local Event Post Any Study Dose (Safety Population) * |
| Table 107: | Logistic Regression Model to Evaluate the Relationship of Treatment with Reporting Any Systemic Event Post Any Study Dose (Safety Population) * |
| Table 108: | Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Maximum Severity and Treatment Group (Safety Population) – Post Any Study Dose* 107 |
| Table 109: | Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Maximum Severity and Treatment Group (Safety Population) – Post Study Dose 1* |
| Table 110: | Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Maximum Severity and Treatment Group (Safety Population) – Post Study Dose 2* |
| Table 111: | Number and Percentage of Subjects Experiencing Solicited Events by Symptom,<br>Maximum Severity and Treatment Group (Safety Population) – Post Study Dose 3* |
| T 11 112 | 111 N. J. D. J. CO.L. J. E. J. C. C. L. J. C. J. J. C. J. J. C. J. J. C. |
| Table 112: | Number and Percentage of Subjects Experiencing Solicited Events by Symptom, |
| | Severity, Day Post Dose, and Treatment Group (Safety Population) – Post Any Study Dose |
| Table 113: | Number and Percentage of Subjects Experiencing Solicited Events by Symptom, |
| Table 113. | Severity, Day Post Dose, and Treatment Group (Safety Population) – Post Study Dose 1 |
| Table 114: | Number and Percentage of Subjects Experiencing Solicited Events by Symptom, |
| 1 | Severity, Day Post Dose, and Treatment Group (Safety Population) – Post Study Dose |
| | 2 |

| Table 115: | Number and Percentage of Subjects Experiencing Solicited Events by Symptom,<br>Severity, Day Post Dose, and Treatment Group (Safety Population) – Post Study Dos | |
|---|---|---|
| Table 116: | 3 | |
| Table 117: | Comparison of the Number and Percentage of Subjects Experiencing Solicited Local Events by Dose and Treatment Group – Safety Population | |
| Table 118: | Number and Percentage of Subjects Experiencing Unsolicited Adverse Events with 95% Confidence Intervals by MedDRA® System Organ Class and Preferred Term, | |
| Table 119: | and Treatment Group – Safety Population* | |
| Table 120: | Relationship, and Treatment Group – Safety Population* | |
| Table 121: | Number and Percentage of Subjects Experiencing Unsolicited Adverse Events Within 21 Days Post Dose by MedDRA® System Organ Class and Preferred Term, Day Pos | 1<br>t |
| Table 122: | Dose, and Treatment Group – Safety Population | |
| Table 123: | Number of Unsolicited Adverse Events by MedDRA® System Organ Class and Preferred Term, Day Post Dose, and Treatment Group – Safety Population | |
| Table 124: | Listing of Serious Adverse Events * | |
| Table 125: | Listing of Medically Attended Adverse Events* | |
| Table 126: | Listing of Potentially Immune Mediated Medical Conditions* | |
| Table 127: | Listing of New Onset Chronic Medical Conditions* | |
| Table 128: | Listing of Non-Serious, Unsolicited, Moderate or Severe Adverse Events* | |
| Table 129: | Laboratory Results by Parameter, Maximum Severity, Study Day, and Treatment | |
| 14010 12). | Group (Safety Population) – All Laboratory Parameters * | 12 |
| Table 130: | Laboratory Results by Parameter, Maximum Severity, Study Day, and Treatment | _ |
| 14010 150. | Group (Safety Population) – White Blood Cells* | 14 |
| Table 131: | Laboratory Results by Parameter, Maximum Severity, Study Day, and Treatment | - |
| 14010 151. | Group (Safety Population) – Hemoglobin* | 15 |
| Table 132: | Laboratory Results by Parameter, Maximum Severity, Study Day, and Treatment | J |
| 14010 132. | Group (Safety Population) – Platelets* | 15 |
| Table 133: | Laboratory Results by Parameter, Maximum Severity, Study Day, and Treatment | J |
| 14010 133. | Group (Safety Population) – Alanine aminotransferase (ALT) * | 15 |
| Table 134: | Laboratory Results by Parameter, Maximum Severity, Study Day, and Treatment | |
| | Group (Safety Population) – Total Bilirubin * | 5 |
| Table 135: | Laboratory Results by Parameter, Maximum Severity, Study Day, and Treatment Group (Safety Population) – Creatinine* | 2 5 |
| Table 136: | Laboratory Summary Statistics of Value and Change from Baseline by Study Day, an | |
| 1 autc 150. | Treatment Group (Safety Population) – White Blood Cells* | |
| Table 137: | Laboratory Summary Statistics of Value and Change from Baseline by Study Day, an | |
| 1 autc 137. | Treatment Group (Safety Population) – Hemoglobin* | |
| Table 138: | Laboratory Summary Statistics of Value and Change from Baseline by Study Day, an | |
| 1 4010 130. | Treatment Group (Safety Population) – Platelets* | |
| Table 139: | Laboratory Summary Statistics of Value and Change from Baseline by Study Day, an | |
| 1 auit 137. | Treatment Group (Safety Population) – Alanine Aminotransferase* (ALT) | |

| Laboratory Summary Statistics of Value and Change from Baseline by Study Day, | |
|---|---|
| Treatment Group (Safety Population) – Total Bilirubin* | 137 |
| Laboratory Summary Statistics of Value and Change from Baseline by Study Day, | and |
| Treatment Group (Safety Population) – Creatinine* | 137 |
| Listing of Abnormal Laboratory Results - Chemistry | 139 |
| Listing of Abnormal Laboratory Results - Hematology | 140 |
| Vital Signs by Assessment, Maximum Severity, Study Day, Treatment Group (Saf | ety |
| Population) – Any Assessment* | 141 |
| Vital Signs by Assessment, Maximum Severity, Study Day, Treatment Group (Saf | ety |
| Population) – Oral Temperature | 141 |
| Vital Signs by Assessment, Maximum Severity, Study Day, and Treatment Group | |
| (Safety Population) – Systolic Blood Pressure | 142 |
| Vital Signs by Assessment, Maximum Severity, Study Day, and Treatment Group | |
| (Safety Population) – Diastolic Blood Pressure | 143 |
| Vital Signs by Assessment, Maximum Severity, Study Day, and Treatment Group | |
| (Safety Population) – Pulse | 143 |
| Number and Percentage of Subjects with Prior and Concurrent Medications by WI | OF |
| Drug Classification and Treatment Group – Safety Population | 144 |
| | Treatment Group (Safety Population) – Total Bilirubin* Laboratory Summary Statistics of Value and Change from Baseline by Study Day, Treatment Group (Safety Population) – Creatinine* Listing of Abnormal Laboratory Results - Chemistry Listing of Abnormal Laboratory Results - Hematology Vital Signs by Assessment, Maximum Severity, Study Day, Treatment Group (Saf Population) – Any Assessment* Vital Signs by Assessment, Maximum Severity, Study Day, Treatment Group (Saf Population) – Oral Temperature Vital Signs by Assessment, Maximum Severity, Study Day, and Treatment Group (Safety Population) – Systolic Blood Pressure Vital Signs by Assessment, Maximum Severity, Study Day, and Treatment Group (Safety Population) – Diastolic Blood Pressure Vital Signs by Assessment, Maximum Severity, Study Day, and Treatment Group (Safety Population) – Diastolic Blood Pressure Vital Signs by Assessment, Maximum Severity, Study Day, and Treatment Group (Safety Population) – Pulse Number and Percentage of Subjects with Prior and Concurrent Medications by Wi |

## 9.1 Overall Study Design and Plan Description

**Table 1: Study Design** 

| | Day 1 | Approximately Day 22 | Approximately Day 43 |
|---|---|---|---|
| | Dose 1 | Dose 2 | Dose 3 |
| Group 1 (Age 19-64) n=60 | Dose 1 (First and Second Study Vaccinations): Sanofi Pasteur H7N9 vaccine 3.75 mcg/ PBS diluent, plus GSK AS03 adjuvant + IIV4 | Dose 2 (Third Study<br>Vaccination):<br>Sanofi Pasteur H7N9<br>vaccine 3.75 mcg/ PBS<br>diluent, plus GSK AS03<br>adjuvant | N/A |
| Group 2<br>(Age 19-64)<br>n=60 | Dose 1 (First Study<br>Vaccination):<br>IIV4 | Dose 2 (Second Study<br>Vaccination):<br>Sanofi Pasteur H7N9<br>vaccine 3.75 mcg/ PBS<br>diluent, plus GSK AS03<br>adjuvant | Dose 3 (Third Study<br>Vaccination):<br>Sanofi Pasteur H7N9<br>vaccine 3.75 mcg/ PBS<br>diluent, plus GSK AS03<br>adjuvant |
| Group 3<br>(Age 19-64)<br>n=30 | Dose 1 (First Study<br>Vaccination):<br>IIV4 | N/A | N/A |
| Total Enrollment, $n = \sim 150$ | Blood for HAI/Neut assays for 2017 H7N9 IIV will be collected: • for Group 1 on Days 1 (baseline), 22, and 43, and at approximately 180 days post second adjuvanted 2017 H7N9 IIV dose (Day 202) • for Group 2, on Days 22 (baseline), 43, and 64, and at approximately 180 days post second 2017 H7N9 IIV dose (Day 223). Serological antibody assays will also be performed against the vaccine viruses in IIV4 from serum samples collected at baseline (Day 1) and approximately 21 and 180 days following receipt of IIV4 (Groups 1, 2 and 3). Safety Lab Timepoints: Group 1: 4 timepoints per subject (Days 1, 8, 22, and 29) Group 2: 6 timepoints per subject (Days 1, 8, 22, 29, 43, and 50) Group 3: 2 timepoints per subject (Days 1 and 8) and Early Termination and /or Unscheduled Visits | | |

## 9.5.1 Efficacy/Immunogenicity and Safety Measurements Assessed and Flow Chart

 Table 2:
 Schedule of Study Procedures – Group 1: Vaccination Period

| Study Visit<br>Number | 00A | V01 | V02 | V03 | V04 <sup>\(\pi\)</sup> | V05 | 90Λ |
|---|---|---|---|---|---|---|---|
| Study Day post<br>Dose 1 | Screening<br>(Optional)<br>D-28 to -1 | Enrollment<br>Dose 1<br>D1 | D4[±1] | D8[+2] | D22[+7] | D25 | D29 |
| Study Day post<br>Dose 2 | | | | | Dose 2<br>D1 | D4[±1] | D8[+2] |
| Obtain Informed<br>Consent∞ | X | Х¬ | | | | | |
| Collect<br>Demographic<br>Information | X | $X^{\dagger*}$ | | | | | |
| Review Eligibility<br>Criteria | X | $X^{\dagger - 1}$ | | | Χ <sup>†</sup> | | |
| Medical History <sup>@</sup> | X | $X^{\dagger \lnot^*}$ | | X | X | | X |
| Concomitant<br>Medications | Χ <sup>ς</sup> | $X^{\dagger ightarrow arsigma}$ | $\mathbf{X}^{arsigma}$ | $\mathbf{X}^{\varsigma}$ | $\mathbf{X}^{\varsigma}$ | $X^{\varsigma}$ | $X^{\varsigma}$ |
| Vital Signs\$ (Oral Temperature%, Pulse, and BP) | X | Χ <sup>†</sup> | | | $X^{\dagger 2}$ | | |
| Height and Weight | X | $X^{\dagger *}$ | | | | | |
| Physical<br>Examination <sup>3</sup> | X | $\{X\}^{\dagger*}$ | | {X} | {X} | | {X} |
| Urine or Serum<br>Pregnancy Test | Χ^ | $X^{\dagger \wedge}$ | | | X <sup>†</sup> ^ | | |
| Venous Blood<br>Collection for ESR | X | $\mathrm{X}^{\neq^*}$ | | | | | |
| Venous Blood<br>Collection for<br>Clinical Safety<br>Laboratory<br>Evaluations~ | | $X^{\dagger}$ | | X | Χ <sup>†</sup> | | X |
| Venous Blood<br>Collection for<br>Immunogenicity<br>Assays | | Χ <sup>†</sup> | | | $X^{\dagger}$ | | |
| Serum Sample<br>Collected for Future<br>Research <sup>4</sup> | | Χ <sup>†</sup> | | X | $X^{\dagger}$ | | X |
| Safety Follow-up<br>Phone Call | | | X | | | X | |

**Table 2:** Schedule of Study Procedures – Group 1: Vaccination Period (continued)

| Study Visit | | _ | 6) | | <b>&gt;</b> . | 10 | 70 |
|---|---|---|---|---|---|---|---|
| Number | 00A | V01 | V02 | V03 | $V04^{\psi}$ | \$0\! | 90A |
| Study Day post<br>Dose 1 | Screening<br>(Optional)<br>D -28 to -1 | Enrollment<br>Dose 1<br>D1 | D4[±1] | D8[+2] | D22[+7] | D25 | D29 |
| Study Day post<br>Dose 2 | | | | | Dose 2<br>D1 | D4[±1] | D8[+2] |
| Enrollment in AdvantageEDC <sup>SM</sup> and Randomization | | $X^{\dagger}$ | | | | | |
| Pre-Administration<br>Reactogenicity<br>Assessments | | $X^{\dagger}$ | | | X | | |
| Vaccination | | X | | | X | | |
| 20-minute<br>Evaluation After<br>Study Vaccination | | X | | | X | | |
| Examine Study<br>Vaccination Site | | X | | X | X | | X |
| Post-Administration<br>Reactogenicity<br>Assessments | | X | | | X | | |
| Distribute Memory<br>Aid and Study-<br>Related Materials | | X | | | X | | |
| Review Memory<br>Aid | | | X | X | | X | X |
| AE/SAE<br>Assessment | | X& | X& | X& | X& | X& | X& |

- ∞ Prior to study procedures.
- † Prior to study vaccination.
- <sup>1</sup> Review results of clinical screening (ESR) or safety laboratory evaluations.
- ¬ Review/confirm information or activity in subjects previously consented and screened.
- © Complete medical history will be obtained by interview of subjects at screening (optional) or on Day 1 prior to the first study vaccination and interim medical history will be obtained by interview of subjects at follow-up visits after Dose 1
- Graceipt of non-study influenza vaccines will be solicited through approximately 180 days after the last study vaccination, and reported in the eCRF.
- \* Not required if done at the optional screening visit.
- All current medications and medications taken within 60 days prior to signing the ICF.
- <sup>\$</sup> Vital signs assessed on Day 1 prior to the first study vaccination will be considered as baseline.
- <sup>%</sup> Subjects must not eat or drink anything hot or cold, or smoke within 10 minutes prior to taking oral temperature.
- Vital signs are not required for subjects who are discontinued from receipt of the third study vaccination and are being followed for safety.
- At the screening (or baseline if not done at screening) visit, a physical examination will be performed on all subjects to include the following organs and organ systems: skin, head and neck, lungs, heart, liver, spleen, extremities, lymph nodes, and nervous system.
- {} Targeted physical examination if indicated based on review of interim medical history.
- ^ May be performed on all women of childbearing potential at screening (optional) and will be performed within 24 hours prior to each vaccination and results must be negative and known prior to each study vaccination.

Table 2: Schedule of Study Procedures – Group 1: Vaccination Period (continued)

| Study Visit<br>Number | 000 | V01 | V02 | V03 | ∨04 | V05 | 90Λ |
|---|---|---|---|---|---|---|---|
| Study Day post<br>Dose 1 | Screening<br>(Optional)<br>D -28 to -1 | Enrollment<br>Dose 1<br>D1 | D4[±1] | D8[+2] | D22[+7] | D25 | D29 |
| Study Day post<br>Dose 2 | | | | | Dose 2<br>D1 | D4[±1] | D8[+2] |

To be performed locally by the site. The ESR value must be confirmed as <30 mm/hr prior to randomization and first study vaccination.

<sup>~</sup> Includes WBC, Hgb, PLT, ALT, T. Bili, Cr.

<sup>&</sup>lt;sup>Ψ</sup> Subjects who do not receive the third study vaccination will continue with follow-up safety assessments (may be conducted by phone call) rather than in person continuing through approximately 12 months after their first study vaccination. These subjects will also be encouraged to provide a venous blood sample for immunogenicity assays at approximately 21 and 180 days after their first study vaccination.

<sup>&</sup>lt;sup>4</sup> For subjects who have consented to collected of serum for future research.

<sup>&</sup>amp; Inclusive of reactogenicity assessments performed on the day of each vaccination through 7 days after each study vaccination.

Table 3: Schedule of Study Procedures – Group 1: Follow-Up Period (Including early termination and unscheduled visits)

| Study Visit Number | <b>L</b> 00 | 80Λ | ^60A | V10 | ПА | Early<br>Termination<br>(if needed) | Unscheduled<br>(if needed) |
|---|---|---|---|---|---|---|---|
| Study Day post Dose 1 | D43 | D64 | D181<br>[±14] | D202 | D387 | | |
| Study Day post Dose 2 | D22[+7] | D43[+7] | | D181[±14] | D366[±14] | | |
| Medical History@ | X | X | X | X | | X | X (if indicated) |
| Concomitant<br>Medications | Χ <sup>ς</sup> | Χ <sup>ς</sup> | Χ <sup>ς</sup> | Χ <sup>ς</sup> | | X (if within 21 days after last<br>study vaccination and receipt<br>of any non-study influenza<br>vaccine will be recorded if<br>within 180 days after the 2nd<br>study vaccination) | X (if within 21 days after last study vaccination and receipt of any non-study influenza vaccine will be recorded if within 180 days after the 2nd study vaccination) |
| Vital Signs\$ (Oral Temperature%, Pulse, and BP) | | | | | | X (may be obtained if indicated) | X (may be obtained if indicated) |
| Physical Examination <sup>3</sup> | {X} | {X} | {X} | {X} | | {X} | {X} |
| Venous Blood<br>Collection for Clinical<br>Safety Laboratory<br>Evaluations~ | | | | | | X (if within 7 days after the last study vaccination) | X (if indicated) |
| Venous Blood<br>Collection for<br>Immunogenicity Assays | X | | X | X | | X(if within 21 days after last study vaccination | X(if within 21 days after last study vaccination |
| Serum Sample Collected<br>for Future Research <sup>4</sup> | X | X | X | X | | X(if within 21 days after last study vaccination | X(if within 21 days after last study vaccination |

Table 3: Schedule of Study Procedures – Group 1: Follow-Up Period (Including early termination and unscheduled visits) (continued)

| Study Visit Number | 707 | V08 | ۸60۸ | V10 | VII | Early<br>Termination<br>(if needed) | Unscheduled<br>(if needed) |
|---|---|---|---|---|---|---|---|
| Study Day post Dose 1 | D43 | D64 | D181<br>[±14] | D202 | D387 | | |
| Study Day post Dose 2 | D22[+7] | D43[+7] | | D181[±14] | D366[±14] | | |
| Safety Follow-up Phone<br>Call | | | | | X | | |
| Examine Study<br>Vaccination Site | | | | | | X (if within 7 days after last study vaccination) | X (if within 7 days after last study vaccination) |
| Post-Administration<br>Reactogenicity<br>Assessments | | | | | | X (if within 7 days after last study vaccination) | X (if within 7 days after last study vaccination) |
| Review Memory Aid | | | | | | X (if within 7 days after last study vaccination) | X (if within 7 days after last study vaccination) |
| AE/SAE Assessment | X | X | X | X | X | X& | X& |

<sup>©</sup> Complete medical history will be obtained by interview of subjects at screening (optional) or on Day 1 prior to the first study vaccination and interim medical history will be obtained by interview of subjects at follow-up visits after Dose 1

<sup>6</sup> Receipt of non-study influenza vaccines will be solicited through approximately 180 days after the last study vaccination, and reported in the eCRF.

Vital signs assessed on Day 1 prior to the first study vaccination will be considered as baseline.

Subjects must not eat or drink anything hot or cold, or smoke within 10 minutes prior to taking oral temperature.

<sup>{}</sup> Targeted physical examination if indicated based on review of interim medical history

<sup>.~</sup> Includes WBC, Hgb, PLT, ALT, T. Bili, Cr.

Ψ Subjects who do not receive the third study vaccination will continue with follow-up safety assessments (may be conducted by phone call) rather than in person continuing through approximately 12 months after their first study vaccination. These subjects will also be encouraged to provide a venous blood sample for immunogenicity assays at approximately 21 and 180 days after their first study vaccination.

<sup>&</sup>lt;sup>4</sup> For subjects who have consented to collected of serum for future use.

Table 4: Schedule of Study Procedures – Group 2: Vaccination Period

| | r | | | | T | | | • | |
|---|---|---|---|---|---|---|---|---|---|
| Study Visit Number | V00 | V01 | V02 | V03 | ∨04 | V05 | 90A | <b>∿</b> 202 | V08 |
| Study Day post Dose 1 | Screening<br>(Optional)<br>D -28 to -1 | Enrollment<br>Dose 1<br>D1 | D4[±1] | D8[+2] | D22[+7] | D25 | D29 | D43 | D46 |
| Study Day post Dose 2 | | | | | Dose 2<br>D1 | D4[±1] | D8[+2] | D22[+7] | D25 |
| Study Day post Dose 3 | | | | | | | | Dose 3<br>D1 | D4[±1] |
| | | Study Pr | ocedure/ | Evaluatio | n | | | | |
| Obtain Informed<br>Consent∞ | X | Χ¬ | | | | | | | |
| Collect Demographic<br>Information | X | $X^{\dagger *}$ | | | | | | | |
| Review Eligibility<br>Criteria | X | $X^{\dagger \dashv 1}$ | | | $X^{\dagger}$ | | | $X^{\dagger}$ | |
| Medical History@ | X | $X^{\dagger \neg^*}$ | | X | X | | X | X | |
| Concomitant Medications | Xς | $X^{\dagger ightharpoons \varsigma}$ | $X^{\varsigma}$ | Xς | Xς | $X^{\varsigma}$ | $X^{\varsigma}$ | Χ <sup>ς</sup> | $X^{\varsigma}$ |
| Vital Signs\$ (Oral Temperature%, Pulse, and BP) | X | Χ <sup>†</sup> | | | $X^{\dagger 2}$ | | | $X^{\dagger 2}$ | |
| Height and Weight | X | $X^{\dagger^*}$ | | | | | | | |
| Physical Examination <sup>3</sup> | X | $X^{\dagger *}$ | | {X} | {X} | | {X} | {X} | |
| Urine or Serum<br>Pregnancy Test | Χ^ | X <sup>†</sup> ^ | | | X <sup>†</sup> ^ | | | X <sup>†</sup> ^ | |
| Venous Blood Collection<br>for ESR | X | $X^{\neq *}$ | | | | | | | |
| Venous Blood Collection<br>for Clinical Safety<br>Laboratory Evaluations~ | | $X^{\dagger}$ | | X | Χ <sup>†</sup> | | X | Χ <sup>†</sup> | |
| Venous Blood Collection<br>for Immunogenicity<br>Assays | | Χ <sup>†</sup> | | | Χ <sup>†</sup> | | | Χ <sup>†</sup> | |
| Serum Sample Collected<br>for Future Research <sup>4</sup> | | $X^{\dagger}$ | | X | $X^{\dagger}$ | | X | Χ <sup>†</sup> | |
| Safety Follow-up Phone<br>Call | | | X | | | X | | | X |
| Enrollment in<br>AdvantageEDC <sup>SM</sup> and<br>Randomization | | $X^{\dagger}$ | | | | | | | |

**Table 4:** Schedule of Study Procedures – Group 2: Vaccination Period (continued)

| Study Visit Number | 000 | V01 | V02 | V03 | ∨04 | V05 | 90A | <b>√07</b> | 80A |
|---|---|---|---|---|---|---|---|---|---|
| Study Day post Dose 1 | Screening<br>(Optional)<br>D -28 to -1 | Enrollment<br>Dose 1<br>D1 | D4[±1] | D8[+2] | D22[+7] | D25 | D29 | D43 | D46 |
| Study Day post Dose 2 | | | | | Dose 2<br>D1 | D4[±1] | D8[+2] | D22[+7] | <b>57</b> 0 |
| Study Day post Dose 3 | | | | | | | | Dose 3<br>D1 | D4[±1] |
| | | Study Pr | ocedure/ | Evaluatio | n | • | • | | |
| Pre-Administration<br>Reactogenicity<br>Assessments | | Χ <sup>†</sup> | | | X | | | X | |
| Vaccination | | X | | | X | | | X | |
| 20-minute Evaluation After Vaccination | | X | | | X | | | X | |
| Examine Vaccination Site | | X | | X | X | | X | X | |
| Post-Administration<br>Reactogenicity<br>Assessments | | X | | | X | | | X | |
| Distribute Memory Aid<br>and Study-Related<br>Materials | | X | | | X | | | X | |
| Review Memory Aid | _ | | X | X | | X | X | | X |
| AE/SAE Assessment | | X& | X& | X& | X& | X& | X& | X& | X& |

- ∞ Prior to study procedures.
- † Prior to study vaccination.
- <sup>1</sup> Review results of clinical screening (ESR) or safety laboratory evaluations.
- ¬ Review/confirm information or activity in subjects previously consented and screened.
- @ Complete medical history will be obtained by interview of subjects at screening (optional) or on Day 1 prior to the first study vaccination and interim medical history will be obtained by interview of subjects at follow-up visits after the first study vaccination.
- <sup>6</sup> Receipt of non-study influenza vaccines will be solicited through approximately 180 days after the last study vaccination, and reported in the eCRF.
- \* Not required if done at the optional screening visit.
- All current medications and medications taken within 60 days prior to signing the ICF.
- Vital signs assessed on Day 1 prior to the first study vaccination will be considered as baseline.
- Subjects must not eat or drink anything hot or cold, or smoke within 10 minutes prior to taking oral temperature.
- Vital signs are not required for subjects who are discontinued from receipt of the third study vaccination and are being followed for safety.
- At the screening (or baseline if not done at screening) visit, a physical examination will be performed on all subjects to include the following organs and organ systems: skin, head and neck, lungs, heart, liver, spleen, extremities, lymph nodes, and nervous system.
- {} Targeted physical examination if indicated based on review of interim medical history.
- May be performed on all women of childbearing potential at screening (optional) and will be performed within 24 hours prior to each vaccination and results must be negative and known prior to each study vaccination.

Table 4: Schedule of Study Procedures – Group 2: Vaccination Period (continued)

| Study Visit Number | 000 | V01 | V02 | V03 | ∨04 | V05 | 90Λ | <b>√07</b> | V08 |
|---|---|---|---|---|---|---|---|---|---|
| Study Day post Dose 1 | Screening<br>(Optional)<br>D -28 to -1 | Enrollment<br>Dose 1<br>D1 | D4[±1] | D8[+2] | D22[+7] | 97Q | D29 | D43 | D46 |
| Study Day post Dose 2 | | | | | Dose 2<br>D1 | D4[±1] | D8[+2] | D22[+7] | D25 |
| Study Day post Dose 3 | | | | | | | | Dose 3<br>D1 | D4[±1] |
| Study Procedure/Evaluation | | | | | | | | | |

To be performed locally by the site. The ESR value must be confirmed as <30 mm/hr prior to randomization and first study vaccination.

<sup>~</sup> Includes WBC, Hgb, PLT, ALT, T. Bili, Cr.

Ψ Subjects who do not receive the third study vaccination will continue with follow-up safety assessments (may be conducted by phone call) rather than in person continuing through approximately 12 months after their first study vaccination. These subjects will also be encouraged to provide a venous blood sample for immunogenicity assays at approximately 21 and 180 days after their first study vaccination.

<sup>&</sup>lt;sup>4</sup> For subjects who have consented to collected of serum for future use.

<sup>&</sup>amp; Inclusive of reactogenicity assessments performed on the day of each vaccination through 7 days after each study vaccination.

Table 5: Schedule of Study Procedures – Group 2: Follow-Up Period (Including early termination and unscheduled visits)

| | | | | | | , | |
|---|---|---|---|---|---|---|---|
| Study Visit<br>Number | 60A | V10 | ۷11۳ | V12 | V13 | Early<br>Terminati<br>on (if<br>needed) | Unschedu<br>led (if<br>needed) |
| Study Day post<br>Dose 1 | D50 | D64 | D181 [±14] | D223 | D408 | | |
| Study Day post<br>Dose 2 | D29 | D43 | | D202 | D387 | | |
| Study Day post<br>Dose 3 | D8[+2] | D22[+7] | | D181[±14] | D366[±14] | | |
| Medical<br>History <sup>@</sup> | X | X | X | X | | X | X (if indicated) |
| Concomitant<br>Medications | Χ <sup>ς</sup> | Χ <sup>ς</sup> | Χ¢ | Χ¢ | | X (if within 21 days after last<br>study vaccination and receipt<br>of any non-study influenza<br>vaccine will be recorded if<br>within 180 days after the 2nd<br>study vaccination) | X (if within 21 days after last<br>study vaccination and receipt<br>of any non-study influenza<br>vaccine will be recorded if<br>within 180 days after the 2nd<br>study vaccination) |
| Vital Signs\$ (Oral Temperature%, Pulse, and BP) | | | | | | X (may be obtained if indicated) | X (may be obtained if indicated) |
| Physical<br>Examination <sup>3</sup> | {X} | {X} | {X} | {X} | | {X} | {X} |
| Venous Blood<br>Collection for<br>Clinical Safety<br>Laboratory<br>Evaluations~ | X | | | | | X (if within 7 days after the last study vaccination) | X (if indicated) |
| Venous Blood<br>Collection for<br>Immunogenicity<br>Assays | | Х | X | X | | X(if within 21 days after last study vaccination | X(if within 21 days after last study vaccination |
| Serum Sample<br>Collected for<br>Future<br>Research <sup>4</sup> | X | X | X | X | | X(if within 21 days after last study vaccination | X(if within 21 days after last study vaccination |
| Safety Follow-<br>up Phone Call | | | | | X | | |
| Examine<br>Vaccination<br>Site | X | | | | | X (if within 7 days after last study vaccination) | X (if within 7 days after last study vaccination) |
| Post-<br>Administration<br>Reactogenicity<br>Assessments | | | | | | X (if within 7 days after last study vaccination) | X (if within 7 days after last study vaccination) |

Table 5: Schedule of Study Procedures – Group 2: Follow-Up Period (Including early termination and unscheduled visits) (continued)

| Study Visit<br>Number | 60A | V10 | V114 | V12 | V13 | Early<br>Terminati<br>on (if<br>needed) | Unschedu<br>led (if<br>needed) |
|---|---|---|---|---|---|---|---|
| Study Day post<br>Dose 1 | D50 | D64 | D181 [±14] | D223 | D408 | | |
| Study Day post<br>Dose 2 | D29 | D43 | | D202 | D387 | | |
| Study Day post<br>Dose 3 | D8[+2] | D22[+7] | | D181[±14] | D366[±14] | | |
| Review<br>Memory Aid | X | | | | | X (if within 7 days after last study vaccination) | X (if within 7 days after last study vaccination) |
| AE/SAE<br>Assessment | X& | X | X | X | X | X <sup>&amp;</sup> | X <sup>&amp;</sup> |

<sup>©</sup> Complete medical history will be obtained by interview of subjects at screening (optional) or on Day 1 prior to the first study vaccination and interim medical history will be obtained by interview of subjects at follow-up visits after the first study vaccination.

<sup>&</sup>lt;sup>5</sup> Receipt of non-study influenza vaccines will be solicited through approximately 180 days after the last study vaccination, and reported in the eCRF.

<sup>&</sup>lt;sup>\$</sup> Vital signs assessed on Day 1 prior to the first study vaccination will be considered as baseline.

Subjects must not eat or drink anything hot or cold, or smoke within 10 minutes prior to taking oral temperature.

<sup>{}</sup> Targeted physical examination if indicated based on review of interim medical history.

<sup>~</sup> Includes WBC, Hgb, PLT, ALT, T. Bili, Cr.

<sup>&</sup>lt;sup>Ψ</sup> Subjects who do not receive the second or third study vaccination will continue with follow-up safety assessments (may be conducted by phone call) rather than in person continuing through approximately 12 months after their first study vaccination. These subjects will also be encouraged to provide a venous blood sample for immunogenicity assays at approximately 21 and 180 days after their first study vaccination.

<sup>&</sup>lt;sup>4</sup> For subjects who have consented to collected of serum for future use

<sup>&</sup>amp; Inclusive of reactogenicity assessments performed on the day of each study vaccination through 7 days after each study vaccination.

Table 6: Schedule of Study Procedures – Group 3: Vaccination and Follow-up Periods

| | | | | | _ | Ī | 1 | | ī |
|---|---|---|---|---|---|---|---|---|---|
| Study Visit Number | $\Lambda$ | V01 | V02 | V03 | $V04^{\psi}$ | V05 | 90Λ | <b>∿</b> 20∆ | 80Λ |
| Study Day post<br>dose | Screening<br>(Optional)<br>D -28 to -1 | Enrollment<br>Dose 1<br>D1 | D4[±1] | D8[+2] | D22[+7] | D43[+7] | D64[+7] | D181[±14] | D366[±14] |
| Obtain Informed<br>Consent | X | Χ¬ | | | | | | | |
| Collect Demographic<br>Information | X | $X^{\dagger *}$ | | | | | | | |
| Review Eligibility<br>Criteria | X | $X^{\dagger \lnot 1}$ | | | | | | | |
| Medical History <sup>@</sup> | X | $X^{\dagger \lnot^*}$ | | X | X | X | X | X | |
| Concomitant<br>Medications | Χς | $X^{\dagger o \varsigma}$ | $\mathbf{X}^{\varsigma}$ | Χς | Χ <sup>ς</sup> | Χç | Χç | Χ¢ | |
| Vital Signs\$ (Oral Temperature%, Pulse, and BP) | X | $X^{\dagger}$ | | | | | | | |
| Height and Weight | X | $X^{\dagger^*}$ | | | | | | | |
| Physical Examination <sup>3</sup> | X | $\{X\}^{\dagger *}$ | | {X} | {X} | {X} | {X} | {X} | |
| Urine or Serum<br>Pregnancy Test | Χ^ | X <sup>†</sup> ^ | | | | | | | |
| Venous Blood<br>Collection for ESR | X | $X^{\neq *}$ | | | | | | | |
| Venous Blood<br>Collection for Clinical<br>Safety Laboratory<br>Evaluations~ | | Х | | X | | | | | |
| Venous Blood<br>Collection for<br>Immunogenicity<br>Assays | | ${ m X}^{\dagger}$ | | | X | | | X | |
| Serum Sample<br>Collected for Future<br>Research <sup>4</sup> | | $X^{\dagger}$ | | X | X | X | X | X | |
| Safety Follow-up<br>Phone Call | | | X | | | | | | X |
| Enrollment in AdvantageEDC <sup>SM</sup> and Randomization | | $X^{\dagger}$ | | | | | | | |
| Pre-Administration<br>Reactogenicity<br>Assessments | | $X^{\dagger}$ | | | | | | | |
| Vaccination | | X | | | | | | | |

**Table 6:** Schedule of Study Procedures – Group 3: Vaccination and Follow-up Periods *(continued)* 

| Study Visit Number | V00 | V01 | V02 | V03 | V04" | V05 | 901 | v07v | 801 |
|---|---|---|---|---|---|---|---|---|---|
| Study Day post<br>dose | Screening<br>(Optional)<br>D -28 to -1 | Enrollment<br>Dose 1<br>D1 | D4[±1] | D8[+2] | D22[+7] | D43[+7] | D64[+7] | D181[±14] | D366[±14] |
| 20-minute Evaluation<br>After Vaccination | | X | | | | | | | |
| Examine Vaccination<br>Site | | X | | X | | | | | |
| Post-Administration<br>Reactogenicity<br>Assessments | | X | | | | | | | |
| Distribute Memory<br>Aid and Study-Related<br>Materials | | X | | | | | | | |
| Review Memory Aid | | | X | X | | | | | |
| AE/SAE Assessment | | X& | X& | X& | X | X | X | X | X |

- ∞ Prior to study procedures.
- † Prior to study vaccination.
- <sup>1</sup> Review results of clinical screening (ESR) or safety laboratory evaluations.
- ¬ Review/confirm information or activity in subjects previously consented and screened
- @ Complete medical history will be obtained by interview of subjects at screening (optional) or on Day 1 prior to study vaccination and interim medical history will be obtained by interview of subjects at follow-up visits after the study vaccination.
- Graph Receipt of non-study influenza vaccines will be solicited through approximately 180 days after the study vaccination, and reported in the eCRF.
- \* Not required if done at the optional screening visit.
- All current medications and medications taken within 60 days prior to signing the ICF.
- Vital signs assessed on Day 1 prior to the study vaccination will be considered as baseline.
- Subjects must not eat or drink anything hot or cold, or smoke within 10 minutes prior to taking oral temperature.
- At the screening (or baseline if not done at screening) visit, a physical examination will be performed on all subjects to include the following organs and organ systems: skin, head and neck, lungs, heart, liver, spleen, extremities, lymph nodes, and nervous system.
- $\{\}\ Targeted\ physical\ examination\ if\ indicated\ based\ on\ review\ of\ interim\ medical\ history.$
- ^ May be performed on all women of childbearing potential at screening (optional) and will be performed within 24 hours prior to study vaccination and results must be negative.
- To be performed locally by the site. The ESR value must be confirmed as <30 mm/hr prior to randomization and study vaccination.</p>
- ~ Includes WBC, Hgb, PLT, ALT, T. Bili, Cr.
- <sup>4</sup> For subjects who have consented to collected of serum for future use.
- & Inclusive of reactogenicity assessments performed on the day of vaccination through 7 days after study vaccination.

Table 7: Schedule of Study Procedures – Group 3: Early Termination and Unscheduled Visits

| Study Visit Number | Early Termination (if<br>needed) | Unscheduled (if<br>needed) |
|---|---|---|
| Study Day post dose | Early Termina<br>needed) | Unschedulec<br>needed) |
| Medical History@ | X | X (if indicated) |
| Concomitant Medications | X (if within 21 days after last study vaccination and receipt of any non-study influenza vaccine will be recorded if within 180 days after the 2nd study vaccination) | X (if within 21 days after last study vaccination and receipt of any non-study influenza vaccine will be recorded if within 180 days after the 2nd study) |
| Vital Signs<br>(Oral Temperature <sup>%</sup> , Pulse, and BP) | X (may be obtained if indicated) | X (may be obtained if indicated) |
| Physical Examination <sup>3</sup> | {X} | {X} |
| Venous Blood Collection for Clinical<br>Safety Laboratory Evaluations~ | X (if within 7 days after the last study vaccination) | X (if indicated) |
| Venous Blood Collection for<br>Immunogenicity Assays | X (if within 21 days after last study vaccination) | X (if within 21 days after last study vaccination) |
| Serum Sample Collected for Future<br>Research <sup>4</sup> | X(if within 21 days after last study vaccination | X(if within 21 days after last study vaccination |
| Examine Vaccination Site | X (if within 7 days after last study vaccination) | X (if within 7 days after last study vaccination) |
| Post-Administration Reactogenicity Assessments | X (if within 7 days after last study vaccination) | X (if within 7 days after last study vaccination) |
| Review Memory Aid | X (if within 7 days after last study vaccination) | X (if within 7 days after last study vaccination) |
| AE/SAE Assessment | X& | X& |

<sup>©</sup> Complete medical history will be obtained by interview of subjects at screening (optional) or on Day 1 prior to study vaccination and interim medical history will be obtained by interview of subjects at follow-up visits after the study

Vital signs assessed on Day 1 prior to the study vaccination will be considered as baseline.

Subjects must not eat or drink anything hot or cold, or smoke within 10 minutes prior to taking oral temperature.

<sup>{}</sup> Targeted physical examination if indicated based on review of interim medical history. ~ Includes WBC, Hgb, PLT, ALT, T. Bili, Cr.

For subjects who have consented to collected of serum for future use.

Inclusive of reactogenicity assessments performed on the day of vaccination through 7 days after study vaccination.

#### 9.7.1 Sample Size

**Table 8:** Power (%) to Detect Safety Events

| Event<br>Frequency | N = 30 | N = 60 | N = 120 |
|---------------------|--------|--------|---------|
| ≥10%<br>Very Common | 96 | >99 | >99 |
| ≥1%<br>Common | 26 | 45 | 70 |
| ≥0.1%<br>Uncommon | 3 | 6 | 11 |
| ≥0.01%<br>Rare | <1 | <1 | 1 |

**Table 9: Precisions of Binomial Confidence Intervals** 

| N | 95% CI |
|-----|--------|
| 30 | 31-69 |
| 60 | 37-63 |
| 120 | 40-60 |

Table 10: Objective 1 -Minimum Detectable Difference in Proportion Responders with 80% Power (N = 50 per group)

| Assumed Proportion Responders comparator arm (pc) | Minimum detectable difference in response rate (p <sub>c</sub> – p <sub>e</sub> ) |
|---|---|
| 0.50 | 0.27 |
| 0.60 | 0.27 |
| 0.70 | 0.27 |
| 0.80 | 0.26 |
| 0.90 | 0.22 |

Table 11: Objective 2 - Minimum Detectable Difference in Proportion Responders with 80% Power

| Assumed Proportion Responders comparator arm (p <sub>c</sub> ) | Minimum detectable decrease in response rate (p <sub>c</sub> - p <sub>e</sub> ) |
|---|---|
| 0.40 | 0.23 |
| 0.50 | 0.24 |
| 0.60 | 0.25 |
| 0.70 | 0.25 |
| 0.80 | 0.23 |
| 0.90 | 0.20 |

#### 10.2 Protocol Deviations

Table 12: Distribution of Protocol Deviations by Category, Type and Treatment Group, All Enrolled Subjects

| | | Group 1:<br>Simultaneous<br>Administration<br>(N=X) | | Group 2:<br>Sequential<br>Administration<br>(N=X) | | Group 3:<br>IIV4 Only<br>(N=X) | | All Subjects<br>(N=X) | |
|---|---|---|---|---|---|---|---|---|---|
| Category | Deviation Type | # of<br>Subj. | # of<br>Dev. | # of<br>Subj. | # of<br>Dev. | # of<br>Subj. | # of<br>Dev. | # of<br>Subj. | # of<br>Dev. |
| Eligibility/enrollment | Any type | | | | | | | | |
| | Did not meet inclusion criterion | x | x | x | x | x | x | x | x |
| | Met exclusion criterion | | | | | | | | |
| | ICF not signed prior to study procedures | | | | | | | | |
| | Other | | | | | | | | |
| Treatment administration schedule | Any type | | | | | | | | |
| | Out of window visit | | | | | | | | |
| | Missed visit/visit not conducted | | | | | | | | |
| | Missed treatment administration | | | | | | | | |
| | Delayed treatment administration | | | | | | | | |
| | Other | | | | | | | | |
| Follow-up visit schedule | Any type | | | | | | | | |
| | Out of window visit | | | | | | | | |
| | Missed visit/visit not conducted | | | | | | | | |
| | Other | | | | | | | | |
| Protocol procedure/assessment | Any type | | | | | | | | |
| | Incorrect version of ICF signed | | | | | | | | |
| | Blood not collected | | | | | | | | |
| | Too few aliquots obtained | | | | | | | | |
| | Specimen result not obtained | | | | | | | | |
| | Required procedure not conducted | | | | | | | | |
| | Required procedure done incorrectly | | | | | | | | |

Table 12: Distribution of Protocol Deviations by Category, Type and Treatment group, All Enrolled Subjects (continued)

| | | Group 1:<br>Simultaneous<br>Administration<br>(N=X) | | Group 2:<br>Sequential<br>Administration<br>(N=X) | | Group 3:<br>IIV4 Only<br>(N=X) | | All Subjects<br>(N=X) | |
|---|---|---|---|---|---|---|---|---|---|
| Category | Deviation Type | # of<br>Subj. | # of<br>Dev. | # of<br>Subj. | # of<br>Dev. | # of<br>Subj. | # of<br>Dev. | # of<br>Subj. | # of<br>Dev. |
| | Study product temperature excursion | | | | | | | | |
| | Specimen temperature excursion | | | | | | | | |
| | Other | | | | | | | | |
| Treatment administration | Any type | | | | | | | | |
| | Required procedure done incorrectly | | | | | | | | |
| | Study product temperature excursion | | | | | | | | |
| | Other | | | | | | | | |
| N = Number of subjects en | nrolled | ı | ı | ı | ı | | | | |

## 12.2.2 Displays of Adverse Events

**Table 13:** Solicited Adverse Event Grading Scale – Local

| | Local (Injection Site) Reactogenicity Grading | | |
|---|---|---|---|
| Local (Injection<br>Site) Reaction | Mild (Grade 1) | Moderate (Grade 2) | Severe (Grade 3) |
| Pain – experienced<br>without touching the<br>injection site<br>(spontaneous<br>discomfort) | Subject is aware of pain,<br>but it does not interfere<br>with daily activity, and<br>no pain medication is<br>taken | Subject is aware of pain; there is interference with daily activity or it requires repeated use of a non-narcotic pain reliever for >24 hours | Subject is aware of pain,<br>and it prevents daily<br>activity or requires any use<br>of a narcotic pain reliever |
| Tenderness – hurts only<br>when injection site is<br>touched or the arm is<br>moved | The area immediately surrounding the injection site hurts only when touched or with arm motion, and it does not interfere with daily activity | The area immediately surrounding the injection site hurts when touched or with arm motion, and it interferes with daily activity | The area immediately surrounding the injection site hurts when touched or with arm motion, and it prevents daily activity |
| Pruritus (Itching) | Does not interfere with daily activity | Interferes with daily activity | Prevents daily activity |
| Ecchymosis<br>(Bruising)* | Does not interfere with daily activity | Interferes with daily activity | Prevents daily activity |
| Erythema (Redness)* | Does not interfere with daily activity | Interferes with daily activity | Prevents daily activity |
| Induration<br>(Hardness)/Swelling* | Does not interfere with daily activity | Interferes with daily activity | Prevents daily activity |
| <u>]</u> | Local (Injection Site) Re | actogenicity Measuremo | ents |
| Local (Injection Site)<br>Reaction | Small (Grade 1) | Medium (Grade 2) | Large (Grade 3) |
| Ecchymosis<br>(Bruising)* | <20 mm | 20 mm – 50 mm | >50 mm |
| Erythema (Redness)* | <20 mm | 20 mm – 50 mm | >50 mm |
| Induration (Hardness)/Swelling* | <20 mm | 20 mm – 50 mm | >50 mm |

**Table 14:** Solicited Adverse Event Grading Scale - Systemic

| Subjective Systemic Reactogenicity Grading | | | |
|---|---|---|---|
| Systemic (Subjective) | Mild (Grade 1) | Moderate (Grade 2) | Severe (Grade 3) |
| Feverishness (Chills/Shivering/Sweating) | No interference with daily activity | Some interference with daily activity | Significant interference, prevents daily activity |
| Fatigue (Tiredness) | No interference with daily activity | Some interference with daily activity | Significant interference, prevents daily activity |
| Malaise (General Unwell<br>Feeling) | No interference with daily activity | Some interference with daily activity | Significant interference, prevents daily activity |
| Myalgia (Body<br>Aches/Muscular Pain)* | No interference with daily activity | Some interference with daily activity | Significant interference, prevents daily activity |
| Arthralgia (Joint Pain)* | No interference with daily activity | Some interference with daily activity | Significant interference, prevents daily activity |
| Headache | No interference with daily activity | Some interference with daily activity | Significant interference, prevents daily activity |
| Nausea | No interference with daily activity | Some interference with daily activity | Significant interference, prevents daily activity |
| | | D 4 C | |

## **Quantitative Systemic Reactogenicity Grading**

| Systemic (Quantitative) | Mild (Grade 1) | Moderate (Grade 2) | Severe (Grade 3) |
|---|---|---|---|
| Fever# - oral <sup>†</sup> | 38.0°C – 38.4°C | 38.5°C – 38.9°C | >38.9°C |
| | 100.4°F – 101.1°F | 101.2°F – 102.0°F | >102.0°F |

<sup>\*</sup> Not at injection site.

# Oral temperature assessed on Day 1 prior to the first study vaccination will be considered as baseline. A fever can be considered not related to the study product if an alternative etiology can be documented.

**Table 15: Vital Signs Adverse Event Grading Scale** 

| For Individuals 19-64 years of age, pulse and blood pressure# will be graded as follows: | | | |
|---|---|---|---|
| Physiologic Parameter Mild (Grade 1) Moderate (Grade 2) Severe (Grade 3) | | | |
| Bradycardia - beats per minute | 45 – 46 | 40 – 44 | <40 |
| Tachycardia - beats per minute | 101 – 130 | 131 – 155 | >155 |
| Hypotension (systolic) mmHg | 80 - 84 | 75 – 79 | <75 |
| Hypotension (diastolic) mmHg | 50 – 54 | 45 – 49 | <45 |
| Hypertension (systolic) mmHg | 151 – 155 | 156 – 160 | >160 |
| Hypertension (diastolic) mmHg | 96 – 100 | 101 – 105 | >105 |

<sup>\*</sup>Pulse and blood pressure assessed on Day 1 prior to the first study vaccination will be considered as baseline.

## 12.4.1 Individual Laboratory Measurements and Abnormal Laboratory Values

**Table 16: Laboratory Adverse Event Grading Scale** 

| Hematology | Mild<br>(Grade 1) | Moderate<br>(Grade 2) | Severe<br>(Grade 3) |
|---|---|---|---|
| WBC 10 <sup>3</sup> /μL (Decrease) | 2.5 – 3.9 | 1.5 – 2.4 | <1.5 |
| WBC 10 <sup>3</sup> /μL (Increase) | 10.6 - 15.0 | 15.1 - 20.0 | >20.0 |
| Hgb g/dL (Decrease) (Female) | 10.1 - 11.4 | 8.5 – 10 | <8.5 |
| Hgb g/dL (Decrease) (Male) | 11.0 – 12.4 | 9.5 – 10.9 | <9.5 |
| Platelets 10 <sup>3</sup> /µL (Decrease) | 125 – 139 | 100 – 124 | <100 |
| Platelets 10 <sup>3</sup> /μL (Increase) | 416 – 550 | 551-750 | >750 |
| Chemistry | Mild<br>(Grade 1) | Moderate<br>(Grade 2) | Severe<br>(Grade 3) |
| ALT IU/L (Increase) (Female) | 44 – 100 | 101 – 200 | >200 |
| ALT IU/L (Increase) (Male) | 61 – 138 | 139 – 275 | >275 |
| Total Bilirubin mg/dL (Increase) – when accompanied by any increase in ALT | 1.30 – 1.59 | 1.60 – 1.80 | >1.80 |
| Total Bilirubin mg/dL (Increase) – when ALT is normal | 1.30 – 1.89 | 1.90 – 2.40 | >2.40 |
| Creatinine mg/dL (Increase)<br>(Female) | 1.1 – 1.7 | 1.8 – 2.0 | >2.0 |
| Creatinine mg/dL (Increase) (Male) | 1.4 - 1.7 | 1.8 – 2.0 | >2.0 |

## 14.1 Description of Study Subjects

#### 14.1.1 Disposition of Subjects

Table 17: Ineligibility Summary of Screen Failures\*

| Inclusion/Exclusion Category | Inclusion/Exclusion Criterion | nª | % b |
|---|---|---|---|
| Inclusion and Exclusion | Number of subjects failing any eligibility criterion | X | х |
| Inclusion | Any inclusion criterion | X | Х |
| | [inclusion criterion 1] | X | х |
| | [inclusion criterion 2] | X | х |
| | [inclusion criterion 3] | X | х |
| Exclusion | Any exclusion criterion | X | х |
| | [exclusion criterion 1] | X | х |
| | [exclusion criterion 2] | X | х |
| | [exclusion criterion 3] | х | х |

<sup>&</sup>lt;sup>a</sup>More than one criterion may be marked per subject.

<sup>&</sup>lt;sup>b</sup>Denominator for percentages is the total number of screen failures.

Table 18: Analysis Populations by Treatment Group – All Enrolled Subjects\*

| | | Simul<br>Admin | Group 1: Simultaneous Administration (N=X) | | Group 2:<br>Sequential<br>Administration<br>(N=X) | | Group 3:<br>IIV4 Only<br>(N=X) | | All Subjects<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| Analysis Populations | Reason Subjects Excluded | n | % | n | % | n | % | n | % |
| Safety Population | Any Reason | х | XX | х | XX | X | xx | х | xx |
| | Study Dose 1 Not Received | | | | | | | | |
| Modified Intent to Treat | Any Reason | | | | | | | | |
| | Study Dose 1 Not Received | | | | | | | | |
| | No Baseline Results Available | | | | | | | | |
| | No Post-Vaccination Results Available | | | | | | | | |
| Per-Protocol, All Visits | Found to be Ineligible After Baseline | | | | | | | | |
| Per-Protocol, Day 22 | Any Reason | | | | | | | | |
| | Study Dose 1 Not Received | | | | | | | | |
| | No Baseline Results Available | | | | | | | | |
| | No Day 22 Result Reported by Lab | | | | | | | | |
| | Lost to Follow-up Before Day 22 | | | | | | | | |
| | Receipt of Non-Study Vaccination | | | | | | | | |
| | Receipt of Immunosuppressive medication | | | | | | | | |
| | Day 22 Visit Out of Window | | | | | | | | |
| Per-Protocol, Day 29 | Any Reason | | | | | NA | NA | | |
| | Study Dose 1 Not Received | | | | | NA | NA | | |
| | Study Dose 2 Not Received | | | | | NA | NA | | |
| | Study Dose 2 Out of Window | | | | | NA | NA | | |
| | No Baseline Results Available | | | | | NA | NA | | |

**Table 18:** Analysis Populations by Treatment Arm – All Enrolled Subjects \* (continued)

**Table 18:** Analysis Populations by Treatment Arm – All Enrolled Subjects \* (continued)

| | No Baseline Results Available | NA | NA | | | NA | NA |
|---|---|---|---|---|---|---|---|
| | No Day 64 Result Reported by Lab | NA | NA | | | NA | NA |
| | Lost to Follow-up Before Day 64 | NA | NA | | | NA | NA |
| | Receipt of Non-Study Vaccination | NA | NA | | | NA | NA |
| | Receipt of Immunosuppressive medication | NA | NA | | | NA | NA |
| Per-Protocol, Day 181 | Any Reason | | | | | | |
| | Study Dose 1 Not Received | | | | | | |
| | No Baseline Results Available | | | | | | |
| | No Day 181 Result Reported by Lab | | | | | | |
| | Lost to Follow-up Before Day 181 | | | | | | |
| | Receipt of Non-Study Vaccination | | | | | | |
| | Receipt of Immunosuppressive medication | | | | | | |
| Per Protocol, Day 202 | Any Reason | | | NA | NA | NA | NA |
| | Study Dose 2 Not Received | | | NA | NA | NA | NA |
| | Study Dose 2 Out of Window | | | | | | |
| | No Baseline Results Available | | | NA | NA | NA | NA |
| | No Day 202 Result Reported by Lab | | | NA | NA | NA | NA |
| | Lost to Follow-up Before Day 202 | | | NA | NA | NA | NA |
| | Receipt of Non-Study Vaccination | | | NA | NA | NA | NA |
| | Receipt of Immunosuppressive medication | | | NA | NA | NA | NA |
| Per Protocol, Day 223 | Any Reason | NA | NA | | | NA | NA |
| | Study Dose 3 Not Received | NA | NA | | | NA | NA |
| | Study Dose 3 Out of Window | NA | NA | | | NA | NA |

**Table 18:** Analysis Populations by Treatment Arm – All Enrolled Subjects \* (continued)

| | No Baseline Results Available | NA | NA | NA | NA |
|---|---|---|---|---|---|
| | No Day 223 Result Reported by Lab | NA | NA | NA | NA |
| | Lost to Follow-up Before Day 223 | NA | NA | NA | NA |
| | Receipt of Non-Study Vaccination | NA | NA | NA | NA |
| | Receipt of Immunosuppressive medication | NA | NA | NA | NA |
| N=Number of subjects enrolled | d | | | | |
Table 19: Subject Disposition by Treatment Group, All Enrolled Subjects\*

| | Simult<br>Admini | up 1:<br>taneous<br>stration<br>=X) | Sequential A | Group 2:<br>Sequential Administration<br>(N=X) | | up 3:<br>Only<br>=X) | All Subjects<br>(N=X) | |
|---|---|---|---|---|---|---|---|---|
| Subject<br>Disposition | n | % | n | % | n | % | n | % |
| Screened | X | | X | | Х | | X | |
| Enrolled/Randomized | X | 100 | X | 100 | Х | 100 | X | 100 |
| Received Dose 1 | X | XX | X | XX | Х | XX | X | XX |
| Received Dose 2 | Х | XX | X | XX | NA | NA | X | xx |
| Received Dose 3 | NA | NA | X | XX | NA | NA | X | xx |
| Received All Scheduled Doses <sup>a</sup> | х | XX | Х | XX | Х | XX | Х | xx |
| Completed Blood Draw for Primary Immunogenicity<br>Analysis <sup>b</sup> | х | XX | х | xx | х | xx | х | xx |
| Included in Per Protocol Primary Immunogenicity Analysis <sup>b c</sup> | Х | XX | X | XX | Х | XX | X | xx |
| Completed Primary Follow-up <sup>a b c</sup> | Х | XX | Х | XX | Х | XX | X | xx |
| Completed Final Study Visit | X | XX | X | XX | X | XX | Х | xx |

N=Number of subjects enrolled

<sup>&</sup>lt;sup>a</sup>Refer to Listing 2 for reasons subjects discontinued from study vaccinations or terminated early.

<sup>&</sup>lt;sup>b</sup>The final blood draw for Primary Immunogenicity Analysis occurs at 21 days post final dose (Day 43 for Group 1; Day 64 for Group 2; Day 21 for Group 3).

<sup>&</sup>lt;sup>c</sup>Refer to Listing 5 for reasons subjects are excluded from the per protocol population.

Table 20: Dates of First Dose by Site and Treatment Group for the Safety Analysis Population

| Dates of Dosing | Group 1:<br>Simultaneous<br>Administration<br>(N=X) | Group 2:<br>Sequential<br>Administration<br>(N=X) | Group 3:<br>IIV4 Only<br>(N=X) | All Subjects<br>(N=X) |
|---|---|---|---|---|
| | [Site 1] | | | |
| Total (Entire period of enrollment) | х | X | x | х |
| DDMMMYYYY-DDMMMYYYY | х | Х | х | х |
| | [Site 2] | | | |
| Total (Entire period of enrollment) | х | Х | х | х |
| DDMMMYYYY-DDMMMYYYY | х | Х | х | х |
| | [Repeat for all s | ites] | | |
| N= Number of subjects in the Safety population. | | | | |

Table 21: Dates of Second Dose by Site and Treatment Group for the Safety Analysis Population

Table 22: Dates of Third Dose by Site and Treatment Group for the Safety Analysis Population

# 14.1.2 Demographic Data

Table 23: Summary of Categorical Demographic and Baseline Characteristics by Site, All Enrolled Subjects

| | | [Sit | te 1]<br>=X) | [Sit<br>(N: | te 2]<br>=X) | | te 3]<br>=X) | [Sit<br>(N: | te 4]<br>=X) | | Subjects<br>N=X) |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Variable | Characteristic | n | % | n | % | n | % | n | % | n | % |
| Sex | Male | Х | xx | х | XX | х | xx | х | xx | х | xx |
| | Female | | | | | | | | | | |
| вмі | < 30 | | | | | | ĺ | | | | |
| | ≥30 | | | | | | | | | | |
| Ethnicity | Not Hispanic or Latino | x | xx | x | xx | x | xx | X | XX | x | xx |
| | Hispanic or Latino | | | | | | | | | | |
| | Not Reported | | | | | : | : | | | | |
| | Unknown | | | | | | | | | | |
| Race | American Indian or Alaska Native | x | xx | x | xx | x | xx | X | XX | x | xx |
| | Asian | | | | | | | | | | |
| | Native Hawaiian or Other Pacific Islander | | | | | | ĺ | | | | |
| | Black or African American | | | | | | | | | | |
| | White | | | | | : | : | | | | |
| | Multi-Racial | | | | | | | | | | |
| | Unknown | | | | | : | : | | | | |
| Prior Seasonal Influenza Vaccination | Received 2016-2017 | | | | | | | | | | |
| | Did not receive 2016-2017 | | | | | | | | | | |
| | Unknown | | | | | | | | | | |
| N= Number of subjects enrolled | • | • | • | | • | • | • | • | • | • | |

Table 24: Summary of Continuous Demographic and Baseline Characteristics by Site, All Enrolled Subjects

| Variable | Statistic | [Site 1]<br>(N=X) | [Site 2]<br>(N=X) | [Site 3]<br>(N=X) | [Site 4]<br>(N=X) | All Subjects (N=X) |
|---|---|---|---|---|---|---|
| Age | Mean | x.x | x.x | X.X | x.x | x.x |
| | Standard Deviation | x.x | x.x | X.X | x.x | x.x |
| | Median | X.X | x.x | X.X | x.x | X.X |
| | Minimum | x | x | X | X | X |
| | Maximum | x | x | X | X | x |
| BMI | Mean | x.x | x.x | X.X | x.x | x.x |
| | Standard Deviation | x.x | x.x | X.X | x.x | x.x |
| | Median | X.X | x.x | X.X | x.x | X.X |
| | Minimum | х | х | X | X | х |
| | Maximum | х | х | X | X | х |
| N= Number of subjects enrolled | <u>.</u><br>1 | | • | • | | • |

Table 25: Summary of Categorical Demographic and Baseline Characteristics by Treatment Group, All Enrolled Subjects\*

| Variable | Characteristic | Group 1:<br>Simultaneous<br>Administration<br>(N=X) | | Sequ<br>Admin | Group 2:<br>Sequential<br>Administration<br>(N=X) | | Group 3:<br>IIV4 Only<br>(N=X) | | All Subjects<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| | | n | % | n | % | n | % | n | % |
| Sex | Male | | | | | | | | |
| | Female | | | | | | | | |
| BMI | < 30 | | | | | | | | |
| | ≥ 30 | | | | | | | | |
| Ethnicity | Not Hispanic or Latino | | | | | | | | |
| | Hispanic or Latino | | | | | | | | |
| | Not Reported | | | | | | | | |
| | Unknown | | | | | | | | |
| Race | American Indian or Alaska Native | | | | | | | | |
| | Asian | | | | | | | | |
| | Native Hawaiian or Other Pacific Islander | | | | | | | | |
| | Black or African American | | | | | | | | |
| | White | | | | | | | | |
| | Multi-Racial | | | | | | | | |
| | Unknown | | | | | | | | |
| Prior Seasonal Influenza<br>Vaccination | Received 2016-2017 | | | | | | | | |
| | Did not receive 2016-2017 | | | | | | | | |
| | Unknown | | | | | | | | |
| N=Number of subjects enrol | led | | _1 | | | 1 | | 1 | |

Table 26: Summary of Continuous Baseline Characteristics by Treatment Group, All Enrolled Subjects\*

| Variable | Statistic | Group 1 Simultaneous Administration (N=X) | Group 2<br>Sequential Administration<br>(N=X) | Group 3<br>IIV4 Only<br>(N=X) | All Subjects<br>(N=X) |
|---|---|---|---|---|---|
| Age | Mean | x.x | X.X | X.X | X.X |
| | Standard Deviation | x.x | X.X | X.X | X.X |
| | Median | х | X | X | X |
| | Minimum | х | X | X | X |
| | Maximum | х | X | X | X |
| BMI | Mean | x.x | X.X | X.X | X.X |
| | Standard Deviation | x.x | X.X | X.X | X.X |
| | Median | х | X | X | X |
| | Minimum | х | X | X | X |
| | Maximum | X | X | X | X |

## 14.1.3 Summary of Prior or Concurrent Medical Conditions

Table 27: Summary of Subjects with Prior or Concurrent Medical Conditions by MedDRA® System Organ Class and Treatment Group, Safety Analysis Population

| | Simultaneous | up 1:<br>Administration<br>=X) | Sequential A | up 2:<br>dministration<br>=X) | Group 3:<br>IIV4 Only<br>(N=X) | |
|---|---|---|---|---|---|---|
| MedDRA® System Organ Class | n | % | n | % | n | % |
| Any SOC | X | XX | Х | XX | Х | XX |
| [SOC 1] | X | XX | Х | XX | Х | XX |
| [SOC 2] | X | xx | X | xx | X | xx |

Note: N=Number of subjects in the Safety population;

n = Number of subjects reporting medical history within the specified SOC. A subject is only counted once per SOC.

## 14.2 Immunogenicity Tables

## 14.2.1 Immune Response Against Vaccine Strains

Table 28: Summaries of Hemagglutination Inhibition Antibody Against 2017 A/H7N9 by Study Day and Treatment Group, Modified Intent-to-Treat Population\*

| | Group 1: Simultaneous Administration (N=X) | Group 2: Sequential Administration (N=X) | Group 3:<br>IIV4 Only<br>(N=X) |
|---|---|---|---|
| Time Point | (IV A) | (IV A) | (IV A) |
| Baseline (Pre-Dose 1) | | | |
| n | x | x | X |
| GMT (95% CI) | xxx.x (xxx.x,xxx.x) | xxx.x (xxx.x,xxx.x) | xxx.x (xxx.x,xxx.x) |
| Titer ≥ 1:40 - %(95% CI) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| 21 Days Post Dose 1 | | | |
| n | x | x | X |
| GMT (95% CI) | xxx.x (xxx.x,xxx.x) | xxx.x (xxx.x,xxx.x) | xxx.x (xxx.x,xxx.x) |
| Seroconversion - % (95% CI) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| Titer ≥ 1:40 - % (95% CI) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| 21 Days Post Dose 2 | | | |
| n | x | X | NA |
| GMT (95% CI) | xxx.x (xxx.x,xxx.x) | xxx.x (xxx.x,xxx.x) | NA |
| Seroconversion - % (95% CI) | xx (xx, xx) | xx (xx, xx) | NA |
| Titer ≥ 1:40 - % (95% CI) | xx (xx, xx) | xx (xx, xx) | NA |
| 21 Days Post Dose 3 | | | |
| n | NA | X | NA |
| GMT (95% CI) | NA | xxx.x (xxx.x,xxx.x) | NA |
| Seroconversion - % (95% CI) | NA | xx (xx, xx) | NA |
| Titer ≥ 1:40 - % (95% CI) | NA | xx (xx, xx) | NA |
| 180 Days Post Dose 1 | | | |

Table 28: Summaries of Hemagglutination Inhibition Antibody Against 2017 A/H7N9 by Study Day and Treatment Group, Modified Intent-to-Treat Population (continued)

| Time Point | Group 1: Simultaneous Administration (N=X) | Group 2: Sequential Administration (N=X) | Group 3:<br>IIV4 Only<br>(N=X) |
|---|---|---|---|
| n | X | x | X |
| GMT (95% CI) | xxx.x (xxx.x,xxx.x) | xxx.x (xxx.x,xxx.x) | xxx.x (xxx.x,xxx.x) |
| Seroconversion - % (95% CI) | xx(xx, xx) | xx (xx, xx) | xx (xx, xx) |
| Titer ≥ 1:40 - % (95% CI) | xx(xx, xx) | xx (xx, xx) | xx (xx, xx) |
| 180 Days Post Second Dose of AS03-adjuvanted H7N9 Vaccine <sup>a</sup> | | | |
| n | X | X | NA |
| GMT (95% CI) | xxx.x (xxx.x,xxx.x) | xxx.x (xxx.x,xxx.x) | NA |
| Seroconversion - % (95% CI) | xx (xx, xx) | xx (xx, xx) | NA |
| Titer ≥ 1:40 - % (95% CI) | xx (xx, xx) | xx (xx, xx) | NA |
| N=number of subjects in the Modified Intent to Treat popul | ation; n = number of subjects with avail | able results; GMT = Geometric Mean Ti | ter |

N=number of subjects in the Modified Intent to Treat population; n = number of subjects with available results; GMT = Geometric Mean Titer

<sup>a</sup> 180 days post second AS03-adjuvanted H7N9 vaccine administration varies by group (Day 202 for Group 1, Day 223 for Group 2, NA for Group 3).

- Table 29: Summaries of Hemagglutination Inhibition Antibody Against 2017 A/H7N9 by Study Day and Treatment Group, Per Protocol Population\*
- Table 30: Summaries of Neutralizing Antibody Against 2017 A/H7N9 by Study Day and Treatment Group, Modified Intent-to-Treat Population\*
- Table 31: Summaries of Neutralizing Antibody Against 2017 A/H7N9 by Study Day and Treatment Group, Per Protocol Population\*

Table 32: Summaries of Hemagglutination Inhibition Antibody Against Seasonal IIV4 Strains by Study Day and Treatment Group, Modified Intent-to-Treat Population\*

| | A/Micl | higan/45/2015<br>(H1N1) | 5 X-275 | A/Hong I | Kong/4801/20<br>(H3N2) | 014 X263B | | huket/3073/2<br>Yamagata lind | | B/Brisbane/60/2008<br>(B Victoria lineage) | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | Group 1<br>Sim.<br>Admin.<br>(N=X) | Group 2<br>Seq.<br>Admin.<br>(N=X) | Group 3<br>IIV4 Only<br>(N=X) | Group 1<br>Sim.<br>Admin.<br>(N=X) | Group 2<br>Seq.<br>Admin.<br>(N=X) | Group 3<br>IIV4 Only<br>(N=X) | Group 1<br>Sim.<br>Admin.<br>(N=X) | Group 2<br>Seq.<br>Admin.<br>(N=X) | Group 3<br>IIV4 Only<br>(N=X) | Group 1<br>Sim.<br>Admin.<br>(N=X) | Group 2<br>Seq.<br>Admin.<br>(N=X) | Group 3<br>IIV4 Only<br>(N=X) |
| Baseline<br>(Pre-Dose 1) | | | | | | | | | | | | |
| n | Х | Х | X | x | х | х | х | х | х | x | x | х |
| GMT<br>(95% CI) | xxx.x<br>(xxx.x,xxx.<br>x) | xxx.x<br>(xxx.x,xxx.<br>x) | xxx.x<br>(xxx.x,xxx.<br>x) | xxx.x<br>(xxx.x,xxx.<br>x) | xxx.x<br>(xxx.x,xxx.<br>x) | xxx.x<br>(xxx.x,xxx.<br>x) | xxx.x<br>(xxx.x,xxx.<br>x) | xxx.x<br>(xxx.x,xxx.<br>x) | xxx.x<br>(xxx.x,xxx.<br>x) | xxx.x<br>(xxx.x,xxx.<br>x) | xxx.x<br>(xxx.x<br>,xxx.x) | xxx.x<br>(xxx.x,<br>xxx.x) |
| Titer ≥ 1:40 - % (95% CI) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| 21 Days Post<br>Dose 1 | | | | | | | | | | | | |
| n | X | X | X | x | x | X | X | X | X | X | x | х |
| GMT<br>(95% CI) | xxx.x<br>(xxx.x,xxx.<br>x) | xxx.x<br>(xxx.x,xxx.<br>x) | xxx.x<br>(xxx.x,xxx.<br>x) | xxx.x<br>(xxx.x,xxx.<br>x) | xxx.x<br>(xxx.x,xxx.<br>x) | xxx.x<br>(xxx.x,xxx.<br>x) | xxx.x<br>(xxx.x,xxx.<br>x) | xxx.x<br>(xxx.x,xxx.<br>x) | xxx.x<br>(xxx.x,xxx.<br>x) | xxx.x<br>(xxx.x,xxx.<br>x) | xxx.x<br>(xxx.x,xxx.<br>x) | xxx.x<br>(xxx.x,xxx.<br>x) |
| Seroconversion<br>% (95% CI) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| Titer ≥ 1:40 - % (95% CI) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| 21 Days Post<br>Dose 2 | | | | | | | | | | | | |
| n | X | х | NA | Х | х | NA | х | х | NA | X | Х | NA |
| GMT<br>(95% CI) | xxx.x<br>(xxx.x,xxx.<br>x) | xxx.x<br>(xxx.x,xxx.<br>x) | NA | xxx.x<br>(xxx.x,xxx.<br>x) | xxx.x<br>(xxx.x,xxx.<br>x) | NA | xxx.x<br>(xxx.x,xxx.<br>x) | xxx.x<br>(xxx.x,xxx.<br>x) | NA | xxx.x<br>(xxx.x,xxx.<br>x) | xxx.x<br>(xxx.x,xxx.<br>x) | NA |
| Seroconversion<br>% (95% CI) | xx (xx, xx) | xx (xx, xx) | NA | xx (xx, xx) | xx (xx, xx) | NA | xx (xx, xx) | xx (xx, xx) | NA | xx (xx, xx) | xx (xx, xx) | NA |

Table 32: Summaries of Hemagglutination Inhibition Antibody Against Seasonal IIV4 Strains by Study Day and Treatment Group, Modified Intent-to-Treat Population (continued)

| | A/Micl | higan/45/2015<br>(H1N1) | 5 X-275 | A/Hong I | Kong/4801/20<br>(H3N2) | 14 X263B | | huket/3073/2<br>/amagata line | | | Brisbane/60/2<br>Victoria linea | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | Group 1<br>Sim.<br>Admin.<br>(N=X) | Group 2<br>Seq.<br>Admin.<br>(N=X) | Group 3<br>IIV4 Only<br>(N=X) | Group 1<br>Sim.<br>Admin.<br>(N=X) | Group 2<br>Seq.<br>Admin.<br>(N=X) | Group 3<br>IIV4 Only<br>(N=X) | Group 1<br>Sim.<br>Admin.<br>(N=X) | Group 2<br>Seq.<br>Admin.<br>(N=X) | Group 3<br>IIV4 Only<br>(N=X) | Group 1<br>Sim.<br>Admin.<br>(N=X) | Group 2<br>Seq.<br>Admin.<br>(N=X) | Group 3<br>IIV4 Only<br>(N=X) |
| Titer ≥ 1:40 - % (95% CI) | xx (xx, xx) | xx (xx, xx) | NA | xx (xx, xx) | xx (xx, xx) | NA | xx (xx, xx) | xx (xx, xx) | NA | xx (xx, xx) | xx (xx, xx) | NA |
| 21 Days Post<br>Dose 3 | | | | | | | | | | | | |
| n | NA | x | NA | NA | x | NA | NA | х | NA | NA | X | NA |
| GMT<br>(95% CI) | NA | xxx.x<br>(xxx.x,xxx.<br>x) | NA | NA | xxx.x<br>(xxx.x,xxx.<br>x) | NA | NA | xxx.x<br>(xxx.x,xxx.<br>x) | NA | NA | xxx.x<br>(xxx.x,xxx.<br>x) | NA |
| Seroconversion<br>% (95% CI) | NA | xx (xx, xx) | NA | NA | xx (xx, xx) | NA | NA | xx (xx, xx) | NA | NA | xx (xx, xx) | NA |
| Titer ≥ 1:40 - % (95% CI) | NA | xx (xx, xx) | NA | NA | xx (xx, xx) | NA | NA | xx (xx, xx) | NA | NA | xx (xx, xx) | NA |
| 180 Days Post<br>Dose 1 (IIV4) | | | | | | | | | | | | |
| n | Х | X | X | x | х | х | х | х | x | х | х | X |
| GMT<br>(95% CI) | xxx.x<br>(xxx.x,xxx.<br>x) | xxx.x<br>(xxx.x,xxx.<br>x) | xxx.x<br>(xxx.x,xxx.<br>x) | xxx.x<br>(xxx.x,xxx.<br>x) | xxx.x<br>(xxx.x,xxx.<br>x) | xxx.x<br>(xxx.x,xxx.<br>x) | xxx.x<br>(xxx.x,xxx.<br>x) | xxx.x<br>(xxx.x,xxx.<br>x) | xxx.x<br>(xxx.x,xxx.<br>x) | xxx.x<br>(xxx.x,xxx.<br>x) | xxx.x<br>(xxx.x,xxx.<br>x) | xxx.x<br>(xxx.x,xxx.<br>x) |
| Seroconversion<br>% (95% CI) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| Titer ≥ 1:40 - % (95% CI) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |

Table 32: Summaries of Hemagglutination Inhibition Antibody Against Seasonal IIV4 Strains by Study Day and Treatment Group, Modified Intent-to-Treat Population (continued)

| | A/Micl | higan/45/2015<br>(H1N1) | 5 X-275 | A/Hong F | Kong/4801/20<br>(H3N2) | 14 X263B | 3B B/Phuket/3073/2013<br>(B Yamagata lineage) | | | | B/Brisbane/60/2008<br>(B Victoria lineage) | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | Group 1<br>Sim.<br>Admin.<br>(N=X) | Group 2<br>Seq.<br>Admin.<br>(N=X) | Group 3<br>IIV4 Only<br>(N=X) | Group 1<br>Sim.<br>Admin.<br>(N=X) | Group 2<br>Seq.<br>Admin.<br>(N=X) | Group 3<br>IIV4 Only<br>(N=X) | Group 1<br>Sim.<br>Admin.<br>(N=X) | Group 2<br>Seq.<br>Admin.<br>(N=X) | Group 3<br>IIV4 Only<br>(N=X) | Group 1<br>Sim.<br>Admin.<br>(N=X) | Group 2<br>Seq.<br>Admin.<br>(N=X) | Group 3<br>IIV4 Only<br>(N=X) |
| 180 Days Post<br>Second Dose of<br>AS03-<br>adjuvanted<br>H7N9<br>Vaccine <sup>a</sup> | | | | | | | | | | | | |
| n | Х | Х | NA | X | х | NA | X | х | NA | X | х | NA |
| GMT<br>(95% CI) | xxx.x<br>(xxx.x,xxx.<br>x) | xxx.x<br>(xxx.x,xxx.<br>x) | NA | xxx.x<br>(xxx.x,xxx.<br>x) | xxx.x<br>(xxx.x,xxx.<br>x) | NA | xxx.x<br>(xxx.x,xxx.<br>x) | xxx.x<br>(xxx.x,xxx.<br>x) | NA | xxx.x<br>(xxx.x,xxx.<br>x) | xxx.x<br>(xxx.x,xxx.<br>x) | NA |
| Seroconversion<br>% (95% CI) | xx (xx, xx) | xx (xx, xx) | NA | xx (xx, xx) | xx (xx, xx) | NA | xx (xx, xx) | xx (xx, xx) | NA | xx (xx, xx) | xx (xx, xx) | NA |
| Titer ≥ 1:40 - % (95% CI) | xx (xx, xx) | xx (xx, xx) | NA | xx (xx, xx) | xx (xx, xx) | NA | xx (xx, xx) | xx (xx, xx) | NA | xx (xx, xx) | xx (xx, xx) | NA |

N=number of subjects in the Modified Intent to Treat population; n = number of subjects with available results; GMT = Geometric Mean Titer

- Table 33: Summaries of Hemagglutination Inhibition Antibody Against Seasonal IIV4 Strains by Study Day and Treatment Group, Per Protocol Population\*
- Table 34: Summaries of Neutralizing Antibody Against Seasonal IIV4 Strains by Study Day and Treatment Group, Modified Intent-to-Treat Population\*
- Table 35: Summaries of Neutralizing Antibody Against Seasonal IIV4 Strains by Study Day and Treatment Group, Per Protocol Population\*

<sup>&</sup>lt;sup>a</sup> 180 days post second AS03-adjuvanted H7N9 vaccine administration varies by group (Day 202 for Group 1, Day 223 for Group 2, NA for Group 3).

Table 36: Summary of Hemagglutination Inhibition Antibody Against 2017 A/H7N9 by Treatment Group and Age Group at 21 Days Post Second Dose of AS03 adjuvanted A/H7N9 Vaccine, Per-Protocol Population\*

| | Group 1: Simultaneous Administration (N=X) | Group 2:<br>Sequential Administration<br>(N=X) |
|---|---|---|
| Age 19-34 years | | |
| n | x | X |
| GMT (95% CI) | xxx.x(xxx.x,xxx.x) | xxx.x(xxx.x,xxx.x) |
| Seroconversion - %(95% CI) | xx (xx, xx) | xx (xx, xx) |
| Titer ≥ 1:40 - %(95% CI) | xx (xx, xx) | xx (xx, xx) |
| Age 35-49 years | | |
| n | x | X |
| GMT (95% CI) | xxx.x(xxx.x,xxx.x) | xxx.x(xxx.x,xxx.x) |
| Seroconversion - %(95% CI) | xx (xx, xx) | xx (xx, xx) |
| Titer $\ge 1:40 - \%(95\% \text{ CI})$ | xx (xx, xx) | xx (xx, xx) |
| Age 50-64 years | | |
| n | x | X |
| GMT (95% CI) | xxx.x(xxx.x,xxx.x) | xxx.x(xxx.x,xxx.x) |
| Seroconversion - %(95% CI) | xx (xx, xx) | xx (xx, xx) |
| Titer $\ge 1:40 - \%(95\% \text{ CI})$ | xx (xx, xx) | xx (xx, xx) |

- Table 37: Summary of Hemagglutination Inhibition Antibody Against 2017 A/H7N9 by Treatment Group and Age Group at 180 Days Post Second Dose of AS03 adjuvanted A/H7N9 Vaccine, Per-Protocol Population
- Table 38: Summary of Neutralizing Antibody Against 2017 A/H7N9 by Treatment Group and Age Group at 21 Days Post Second Dose of AS03 adjuvanted A/H7N9 Vaccine, Per-Protocol Population\*
- Table 39: Summary of Neutralizing Antibody Against 2017 A/H7N9 by Treatment Group and Age Group at 180 Days Post Second Dose of AS03 adjuvanted A/H7N9 Vaccine, Per-Protocol Population

Table 40: Summary of Hemagglutination Inhibition Antibody Against Seasonal IIV4 Strains by Treatment Group and Age Group at 21 Days Post IIV4, Per-Protocol Population\*

| | A/Mic | higan/45/201<br>(H1N1) | 5 X-275 | A/Hong I | Kong/4801/20<br>(H3N2) | 14 X263B | | huket/3073/2<br>/amagata line | | - | Florida/04/20<br>magata linea | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Group 1<br>Sim.<br>Admin.<br>(N=X) | Group 2<br>Seq.<br>Admin.<br>(N=X) | Group 3<br>IIV4 Only<br>(N=X) | Group 1<br>Sim.<br>Admin.<br>(N=X) | Group 2<br>Seq.<br>Admin.<br>(N=X) | Group 3<br>IIV4<br>Only<br>(N=X) | Group 1<br>Sim.<br>Admin.<br>(N=X) | Group 2<br>Seq.<br>Admin.<br>(N=X) | Group 3<br>IIV4<br>Only<br>(N=X) | Group 1<br>Sim.<br>Admin.<br>(N=X) | Group 2<br>Seq.<br>Admin.<br>(N=X) | Group 3<br>IIV4<br>Only<br>(N=X) |
| Age<br>19-34 years | | | | | | | | | | | | |
| n | x | x | X | X | X | X | X | x | x | x | x | х |
| GMT<br>(95% CI) | xxx.x<br>(xxx.x,<br>xxx.x) | xxx.x<br>(xxx.x,<br>xxx.x) | xxx.x<br>(xxx.x,<br>xxx.x) | xxx.x<br>(xxx.x,<br>xxx.x) | xxx.x<br>(xxx.x,<br>xxx.x) | xxx.x<br>(xxx.x,<br>xxx.x) | xxx.x<br>(xxx.x,<br>xxx.x) | xxx.x<br>(xxx.x,<br>xxx.x) | xxx.x<br>(xxx.x,<br>xxx.x) | xxx.x<br>(xxx.x,<br>xxx.x) | xxx.x<br>(xxx.x,<br>xxx.x) | xxx.x<br>(xxx.x,<br>xxx.x) |
| Seroconversi<br>on - %(95%<br>CI) | xx (xx,<br>xx) | xx (xx,<br>xx) | xx (xx, xx) | xx (xx,<br>xx) | xx (xx,<br>xx) | xx (xx,<br>xx) | xx (xx,<br>xx) | xx (xx,<br>xx) | xx (xx,<br>xx) | xx (xx,<br>xx) | xx (xx,<br>xx) | xx (xx,<br>xx) |
| Titer ≥ 1:40 - %(95% CI) | xx (xx,<br>xx) | xx (xx,<br>xx) | xx (xx, xx) | xx (xx,<br>xx) | xx (xx,<br>xx) | xx (xx,<br>xx) | xx (xx,<br>xx) | xx (xx,<br>xx) | xx (xx,<br>xx) | xx (xx,<br>xx) | xx (xx,<br>xx) | xx (xx,<br>xx) |
| Age<br>35-49 years | | | | | | | | | | | | |
| n | x | x | X | X | X | X | X | x | x | x | x | х |
| GMT (95%<br>CI) | xxx.x<br>(xxx.x,<br>xxx.x) | xxx.x<br>(xxx.x,<br>xxx.x) | xxx.x<br>(xxx.x,<br>xxx.x) | xxx.x<br>(xxx.x,<br>xxx.x) | xxx.x<br>(xxx.x,<br>xxx.x) | xxx.x<br>(xxx.x,<br>xxx.x) | xxx.x<br>(xxx.x,<br>xxx.x) | xxx.x<br>(xxx.x,<br>xxx.x) | xxx.x<br>(xxx.x,<br>xxx.x) | xxx.x<br>(xxx.x,<br>xxx.x) | xxx.x<br>(xxx.x,<br>xxx.x) | xxx.x<br>(xxx.x,<br>xxx.x) |
| Seroconversi<br>on - %(95%<br>CI) | xx (xx,<br>xx) | xx (xx,<br>xx) | xx (xx, xx) | xx (xx,<br>xx) | xx (xx,<br>xx) | xx (xx,<br>xx) | xx (xx,<br>xx) | xx (xx,<br>xx) | xx (xx,<br>xx) | xx (xx,<br>xx) | xx (xx,<br>xx) | xx (xx,<br>xx) |
| Titer ≥ 1:40 - %(95% CI) | xx (xx,<br>xx) | xx (xx,<br>xx) | xx (xx, xx) | xx (xx,<br>xx) | xx (xx,<br>xx) | xx (xx,<br>xx) | xx (xx,<br>xx) | xx (xx,<br>xx) | xx (xx,<br>xx) | xx (xx,<br>xx) | xx (xx,<br>xx) | xx (xx,<br>xx) |
| Age<br>50-64 years | | | | | | | | | | | | |

Table 40: Summary of Hemagglutination Inhibition Antibody Against Seasonal IIV4 Strains by Treatment Group and Age Group at 21 Days Post IIV4, Per-Protocol Population (continued)

| | A/Michigan/45/2015 X-275<br>(H1N1) | | | A/Hong Kong/4801/2014 X263B<br>(H3N2) | | | B/Phuket/3073/2013<br>(B Yamagata lineage) | | | B/Florida/04/2006<br>(Yamagata lineage) | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Group 1<br>Sim.<br>Admin.<br>(N=X) | Group 2<br>Seq.<br>Admin.<br>(N=X) | Group 3<br>IIV4 Only<br>(N=X) | Group 1<br>Sim.<br>Admin.<br>(N=X) | Group 2<br>Seq.<br>Admin.<br>(N=X) | Group 3<br>IIV4<br>Only<br>(N=X) | Group 1<br>Sim.<br>Admin.<br>(N=X) | Group 2<br>Seq.<br>Admin.<br>(N=X) | Group 3 IIV4 Only (N=X) | Group 1<br>Sim.<br>Admin.<br>(N=X) | Group 2<br>Seq.<br>Admin.<br>(N=X) | Group 3<br>IIV4<br>Only<br>(N=X) |
| n | х | X | X | X | Х | х | Х | X | X | X | X | X |
| GMT (95%<br>CI) | xxx.x<br>(xxx.x,<br>xxx.x) | xxx.x<br>(xxx.x,<br>xxx.x) | xxx.x<br>(xxx.x,<br>xxx.x) | xxx.x<br>(xxx.x,<br>xxx.x) | xxx.x<br>(xxx.x,<br>xxx.x) | xxx.x<br>(xxx.x,<br>xxx.x) | xxx.x<br>(xxx.x,<br>xxx.x) | xxx.x<br>(xxx.x,<br>xxx.x) | xxx.x<br>(xxx.x,<br>xxx.x) | xxx.x<br>(xxx.x,<br>xxx.x) | xxx.x<br>(xxx.x,<br>xxx.x) | xxx.x<br>(xxx.x,<br>xxx.x) |
| Seroconversi<br>on - %(95%<br>CI) | xx (xx,<br>xx) | xx (xx,<br>xx) | xx (xx, xx) | xx (xx,<br>xx) | xx (xx,<br>xx) | xx (xx,<br>xx) | xx (xx,<br>xx) | xx (xx,<br>xx) | xx (xx,<br>xx) | xx (xx,<br>xx) | xx (xx,<br>xx) | xx (xx,<br>xx) |
| Titer ≥ 1:40 - %(95% CI) | xx (xx,<br>xx) | xx (xx,<br>xx) | xx (xx, xx) | xx (xx,<br>xx) | xx (xx,<br>xx) | xx (xx,<br>xx) | xx (xx,<br>xx) | xx (xx,<br>xx) | xx (xx,<br>xx) | xx (xx,<br>xx) | xx (xx,<br>xx) | xx (xx,<br>xx) |
| N = Number of | N = Number of subjects in the Per Protocol Population; n = number of subjects with results reported | | | | | | | | | | | |

- Table 41: Summary of Hemagglutination Inhibition Antibody Against Seasonal IIV4 Strains by Treatment Group and Age Group at 180 Days Post Second Dose of AS03 adjuvanted A/H7N9 Vaccine, Per-Protocol Population
- Table 42: Summary of Neutralizing Antibody Against Seasonal IIV4 Strains by Treatment Group and Age Group at 21 Days Post Second Dose of AS03 adjuvanted A/H7N9 Vaccine, Per-Protocol Population\*
- Table 43: Summary of Neutralizing Antibody Against Seasonal IIV4 Strains by Treatment Group and Age Group at 180 Days Post Second Dose of AS03 adjuvanted A/H7N9 Vaccine, Per-Protocol Population

Table 44: Summary of Hemagglutination Inhibition Antibody Against 2017 A/H7N9 by Treatment Group and Sex at 21 Days Post Second Dose of AS03 adjuvanted A/H7N9 Vaccine, Per-Protocol Population\*

| | Group 1: Simultaneous Administration (N=X) | Group 2:<br>Sequential Administration<br>(N=X) |
|---|---|---|
| Female | | |
| n | x | x |
| GMT (95% CI) | xxx.x (xxx.x,xxx.x) | xxx.x (xxx.x,xxx.x) |
| Seroconversion - %(95% CI) | xx (xx, xx) | xx(xx, xx) |
| Titer $\ge 1:40$ - %(95% CI) | xx (xx, xx) | xx (xx, xx) |
| Male | | |
| n | x | x |
| GMT (95% CI) | xxx.x (xxx.x,xxx.x) | xxx.x (xxx.x,xxx.x) |
| Seroconversion - %(95% CI) | xx (xx, xx) | xx (xx, xx) |
| Titer $\geq 1:40 - \%(95\% \text{ CI})$ | xx (xx, xx) | xx (xx, xx) |

- Table 45: Summary of Hemagglutination Inhibition Antibody Against 2017 A/H7N9 by Treatment Group and Sex at 180 Days Post Second Dose of AS03 adjuvanted A/H7N9 Vaccine, Per-Protocol Population
- Table 46: Summary of Neutralizing Antibody Against 2017 A/H7N9 by Treatment Group and Sex at 21 Days Post Second Dose of AS03 adjuvanted A/H7N9 Vaccine, Per-Protocol Population\*
- Table 47: Summary of Neutralizing Antibody Against 2017 A/H7N9 by Treatment Group and Sex at 180 Days Post Second Dose of AS03 adjuvanted A/H7N9 Vaccine, Per-Protocol Population

Table 48: Summary of Hemagglutination Inhibition Antibody Against Seasonal IIV4 Strains by Treatment Group and Sex at 21 Days Post IIV4 Vaccination, Per-Protocol Population\*

| | A/Micl | higan/45/2015<br>(H1N1) | 5 X-275 | A/Hong I | Kong/4801/20<br>(H3N2) | 14 X263B | | huket/3073/2<br>Yamagata line | | | risbane/60/2<br>Victoria linea | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Group 1<br>Sim.<br>Admin.<br>(N=X) | Group 2<br>Seq.<br>Admin.<br>(N=X) | Group 3<br>IIV4 Only<br>(N=X) | Group 1<br>Sim.<br>Admin.<br>(N=X) | Group 2<br>Seq.<br>Admin.<br>(N=X) | Group 3<br>IIV4 Only<br>(N=X) | Group 1<br>Sim.<br>Admin.<br>(N=X) | Group 2<br>Seq.<br>Admin.<br>(N=X) | Group 3<br>IIV4 Only<br>(N=X) | Group 1<br>Sim.<br>Admin.<br>(N=X) | Group 2<br>Seq.<br>Admin.<br>(N=X) | Group 3<br>IIV4 Only<br>(N=X) |
| Female | | | | | | | | | | | | |
| n | Х | Х | X | х | Х | х | х | х | х | X | X | х |
| GMT<br>(95% CI) | xxx.x<br>(xxx.x,<br>xxx.x) | xxx.x<br>(xxx.x,<br>xxx.x) | xxx.x<br>(xxx.x,<br>xxx.x) | xxx.x<br>(xxx.x,<br>xxx.x) | xxx.x<br>(xxx.x,<br>xxx.x) | xxx.x<br>(xxx.x,<br>xxx.x) | xxx.x<br>(xxx.x,<br>xxx.x) | xxx.x<br>(xxx.x,<br>xxx.x) | xxx.x<br>(xxx.x,<br>xxx.x) | xxx.x<br>(xxx.x,<br>xxx.x) | xxx.x<br>(xxx.x,<br>xxx.x) | xxx.x<br>(xxx.x,<br>xxx.x) |
| Seroconversion<br>- %(95% CI) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| Titer ≥ 1:40 - %(95% CI) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| Male | | | | | | | | | | | | |
| n | Х | Х | Х | х | X | Х | х | х | х | Х | X | х |
| GMT (95%<br>CI) | xxx.x<br>(xxx.x,<br>xxx.x) | xxx.x<br>(xxx.x,<br>xxx.x) | xxx.x<br>(xxx.x,<br>xxx.x) | xxx.x<br>(xxx.x,<br>xxx.x) | xxx.x<br>(xxx.x,<br>xxx.x) | xxx.x<br>(xxx.x,<br>xxx.x) | xxx.x<br>(xxx.x,<br>xxx.x) | xxx.x<br>(xxx.x,<br>xxx.x) | xxx.x<br>(xxx.x,<br>xxx.x) | xxx.x<br>(xxx.x,<br>xxx.x) | xxx.x<br>(xxx.x,<br>xxx.x) | xxx.x<br>(xxx.x,<br>xxx.x) |
| Seroconversion<br>- %(95% CI) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| Titer ≥ 1:40 - %(95% CI) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| N = Number of s | subjects in the | Per Protocol | Population; n | = number of | subjects with | results report | ed | • | • | • | • | • |

- Table 49: Summary of Hemagglutination Inhibition Antibody Against Seasonal IIV4 Strains by Treatment Group and Sex at 180 Days Post IIV4 Vaccination, Per-Protocol Population
- Table 50: Summary of Neutralizing Antibody Against Seasonal IIV4 Strains by Treatment Group and Sex at 21 Days Post IIV4 Vaccination, Per-Protocol Population\*
- Table 51: Summary of Neutralizing Antibody Against Seasonal IIV4 Strains by Treatment Group and Sex at 180 Days Post IIV4 Vaccination, Per-Protocol Population

Table 52: Summary of Hemagglutination Inhibition Antibody Against 2017 A/H7N9 by Treatment Group and BMI at 21 Days Post Second Dose of AS03 adjuvanted A/H7N9 Vaccine, Per-Protocol Population\*

| | Group 1: Simultaneous Administration (N=X) | Group 2: Sequential Administration (N=X) |
|---|---|---|
| BMI < 30 | | |
| n | x | x |
| GMT (95% CI) | xxx.x (xxx.x,xxx.x) | xxx.x (xxx.x,xxx.x) |
| Seroconversion - %(95% CI) | xx (xx, xx) | xx (xx, xx) |
| Titer ≥ 1:40 - %(95% CI) | xx (xx, xx) | xx (xx, xx) |
| BMI ≥ 30 | | |
| n | x | x |
| GMT (95% CI) | xxx.x (xxx.x,xxx.x) | xxx.x (xxx.x,xxx.x) |
| Seroconversion - %(95% CI) | xx (xx, xx) | xx (xx, xx) |
| Titer ≥ 1:40 - %(95% CI) | xx (xx, xx) | xx (xx, xx) |
| N = Number of subjects in the Per Protocol Population; n = num | ber of subjects with results reported | |

- Table 53: Summary of Hemagglutination Inhibition Antibody Against 2017 A/H7N9 by Treatment Group and BMI at 180 Days Post Second Dose of AS03 adjuvanted A/H7N9 Vaccine, Per-Protocol Population
- Table 54: Summary of Neutralizing Antibody Against 2017 A/H7N9 by Treatment Group and BMI at 21 Days Post Second Dose of AS03 adjuvanted A/H7N9 Vaccine, Per-Protocol Population\*
- Table 55: Summary of Neutralizing Antibody Against 2017 A/H7N9 by Treatment Group and BMI at 180 Days Post Second Dose of AS03 adjuvanted A/H7N9 Vaccine, Per-Protocol Population

Table 56: Summary of Hemagglutination Inhibition Antibody Against Seasonal IIV4 Strains by Treatment Group and BMI at 21 Days Post IIV4 Vaccination, Per-Protocol Population\*

| | A/Micl | higan/45/2015<br>(H1N1) | 5 X-275 | A/Hong I | Kong/4801/20<br>(H3N2) | 14 X263B | | huket/3073/2<br>'amagata line | | B/Brisbane/60/2008<br>(B Victoria lineage) | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Group 1<br>Sim.<br>Admin.<br>(N=X) | Group 2<br>Seq.<br>Admin.<br>(N=X) | Group 3<br>IIV4 Only<br>(N=X) | Group 1<br>Sim.<br>Admin.<br>(N=X) | Group 2<br>Seq.<br>Admin.<br>(N=X) | Group 3<br>IIV4 Only<br>(N=X) | Group 1<br>Sim.<br>Admin.<br>(N=X) | Group 2<br>Seq.<br>Admin.<br>(N=X) | Group 3<br>IIV4 Only<br>(N=X) | Group 1<br>Sim.<br>Admin.<br>(N=X) | Group 2<br>Seq.<br>Admin.<br>(N=X) | Group 3<br>IIV4 Only<br>(N=X) |
| BMI < 30 | | | | | | | | | | | | |
| n | Х | Х | X | х | х | х | х | х | х | X | X | х |
| GMT<br>(95% CI) | xxx.x<br>(xxx.x,<br>xxx.x) | xxx.x<br>(xxx.x,<br>xxx.x) | xxx.x<br>(xxx.x,<br>xxx.x) | xxx.x<br>(xxx.x,<br>xxx.x) | xxx.x<br>(xxx.x,<br>xxx.x) | xxx.x<br>(xxx.x,<br>xxx.x) | xxx.x<br>(xxx.x,<br>xxx.x) | xxx.x<br>(xxx.x,<br>xxx.x) | xxx.x<br>(xxx.x,<br>xxx.x) | xxx.x<br>(xxx.x,<br>xxx.x) | xxx.x<br>(xxx.x,<br>xxx.x) | xxx.x<br>(xxx.x,<br>xxx.x) |
| Seroconversion<br>- %(95% CI) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| Titer ≥ 1:40 - %(95% CI) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| BMI ≥ 30 | | | | | | | | | | | | |
| n | Х | Х | Х | х | X | х | х | х | х | Х | X | х |
| GMT (95%<br>CI) | xxx.x<br>(xxx.x,<br>xxx.x) | xxx.x<br>(xxx.x,<br>xxx.x) | xxx.x<br>(xxx.x,<br>xxx.x) | xxx.x<br>(xxx.x,<br>xxx.x) | xxx.x<br>(xxx.x,<br>xxx.x) | xxx.x<br>(xxx.x,<br>xxx.x) | xxx.x<br>(xxx.x,<br>xxx.x) | xxx.x<br>(xxx.x,<br>xxx.x) | xxx.x<br>(xxx.x,<br>xxx.x) | xxx.x<br>(xxx.x,<br>xxx.x) | xxx.x<br>(xxx.x,<br>xxx.x) | xxx.x<br>(xxx.x,<br>xxx.x) |
| Seroconversion<br>- %(95% CI) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| Titer ≥ 1:40 - %(95% CI) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| N = Number of s | subjects in the | Per Protocol | Population; n | = number of | subjects with | results report | ed | • | • | • | • | • |

- Table 57: Summary of Hemagglutination Inhibition Antibody Against Seasonal IIV4 Strains by Treatment Group and BMI at 180 Days Post IIV4 Vaccination, Per-Protocol Population
- Table 58: Summary of Neutralizing Antibody Against Seasonal IIV4 Strains by Treatment Group and BMI at 21 Days Post IIV4 Vaccination, Per-Protocol Population\*
- Table 59: Summary of Neutralizing Antibody Against Seasonal IIV4 Strains by Treatment Group and BMI at 180 Days Post IIV4 Vaccination, Per-Protocol Population

Table 60: Summary of Hemagglutination Inhibition Antibody Against 2017 A/H7N9 by Treatment Group and Prior Seasonal Influenza Vaccination at 21 Days Post Second Dose of AS03 adjuvanted A/H7N9 Vaccine, Per-Protocol Population\*

| | Group 1:<br>Simultaneous Administration<br>(N=X) | Group 2:<br>Sequential<br>Administration<br>(N=X) |
|---|---|---|
| Did Not Receive 2016-2017 Seasonal Influenza Vaccination | | |
| n | X | x |
| GMT (95% CI) | xxx.x (xxx.x,xxx.x) | xxx.x (xxx.x,xxx.x) |
| Seroconversion - %(95% CI) | xx (xx, xx) | xx (xx, xx) |
| Titer ≥ 1:40 - %(95% CI) | xx (xx, xx) | xx (xx, xx) |
| Received 2016-2017 Seasonal Influenza Vaccination | | |
| n | x | x |
| GMT (95% CI) | xxx.x (xxx.x,xxx.x) | xxx.x (xxx.x,xxx.x) |
| Seroconversion - %(95% CI) | xx (xx, xx) | xx (xx, xx) |
| Titer ≥ 1:40 - %(95% CI) | xx (xx, xx) | xx (xx, xx) |
| N = Number of subjects in the Per Protocol Population; n = number of subjects in the Per Protocol Population; n = numbe | f subjects with results reported | |

- Table 61: Summary of Hemagglutination Inhibition Antibody Against 2017 A/H7N9 by Treatment Group and Prior Seasonal Influenza Vaccination at 180 Days Post Second Dose of AS03 adjuvanted A/H7N9 Vaccine, Per-Protocol Population
- Table 62: Summary of Neutralizing Antibody Against 2017 A/H7N9 by Treatment Group and Prior Seasonal Influenza Vaccination at 21 Days Post Second Dose of AS03 adjuvanted A/H7N9 Vaccine, Per-Protocol Population\*
- Table 63: Summary of Neutralizing Antibody Against 2017 A/H7N9 by Treatment Group and Prior Seasonal Influenza Vaccination at 180 Days Post Second Dose of AS03 adjuvanted A/H7N9 Vaccine, Per-Protocol Population

Table 64: Summary of Hemagglutination Inhibition Antibody Against Seasonal IIV4 Strains by Treatment Group and Prior Seasonal Influenza Vaccination at 21 Days Post IIV4 Vaccination, Per-Protocol Population\*

| | A/Mic | higan/45/201:<br>(H1N1) | 5 X-275 | A/Hong k | Kong/4801/20<br>(H3N2) | 14 X263B | - | huket/3073/2<br>Yamagata line | | - | risbane/60/2<br>Victoria linea | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Group 1<br>Sim.<br>Admin.<br>(N=X) | Group 2<br>Seq.<br>Admin.<br>(N=X) | Group 3<br>IIV4 Only<br>(N=X) | Group 1<br>Sim.<br>Admin.<br>(N=X) | Group 2<br>Seq.<br>Admin.<br>(N=X) | Group 3<br>IIV4 Only<br>(N=X) | Group 1<br>Sim.<br>Admin.<br>(N=X) | Group 2<br>Seq.<br>Admin.<br>(N=X) | Group 3<br>IIV4 Only<br>(N=X) | Group 1<br>Sim.<br>Admin.<br>(N=X) | Group 2<br>Seq.<br>Admin.<br>(N=X) | Group 3<br>IIV4 Only<br>(N=X) |
| Did Not Receive | e 2016-2017 S | Seasonal Infl | uenza Vaccin | ation | | | • | | • | | | |
| n | Х | Х | X | х | x | х | x | x | x | X | х | х |
| GMT<br>(95% CI) | xxx.x<br>(xxx.x,<br>xxx.x) | xxx.x<br>(xxx.x,<br>xxx.x) | xxx.x<br>(xxx.x,<br>xxx.x) | xxx.x<br>(xxx.x,<br>xxx.x) | xxx.x<br>(xxx.x,<br>xxx.x) | xxx.x<br>(xxx.x,<br>xxx.x) | xxx.x<br>(xxx.x,<br>xxx.x) | xxx.x<br>(xxx.x,<br>xxx.x) | xxx.x<br>(xxx.x,<br>xxx.x) | xxx.x<br>(xxx.x,<br>xxx.x) | xxx.x<br>(xxx.x,<br>xxx.x) | xxx.x<br>(xxx.x,<br>xxx.x) |
| Seroconversion<br>- %(95% CI) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| Titer ≥ 1:40 - %(95% CI) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| Received 2016-2 | 2017 Seasona | l Influenza V | accination | • | | | • | | • | | • | |
| n | Х | х | X | X | X | X | x | x | x | X | x | x |
| GMT (95%<br>CI) | xxx.x<br>(xxx.x,<br>xxx.x) | xxx.x<br>(xxx.x,<br>xxx.x) | xxx.x<br>(xxx.x,<br>xxx.x) | xxx.x<br>(xxx.x,<br>xxx.x) | xxx.x<br>(xxx.x,<br>xxx.x) | xxx.x<br>(xxx.x,<br>xxx.x) | xxx.x<br>(xxx.x,<br>xxx.x) | xxx.x<br>(xxx.x,<br>xxx.x) | xxx.x<br>(xxx.x,<br>xxx.x) | xxx.x<br>(xxx.x,<br>xxx.x) | xxx.x<br>(xxx.x,<br>xxx.x) | xxx.x<br>(xxx.x,<br>xxx.x) |
| Seroconversion<br>- %(95% CI) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| Titer ≥ 1:40 - %(95% CI) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| N = Number of s | subjects in the | Per Protocol | Population; n | = number of | subjects with | results report | ed | • | | | | |

- Table 65: Summary of Hemagglutination Inhibition Antibody Against Seasonal IIV4 Strains by Treatment Group and Prior Seasonal Influenza Vaccination at 180 Days Post IIV4 Vaccination, Per-Protocol Population
- Table 66: Summary of Neutralizing Antibody Against Seasonal IIV4 Strains by Treatment Group and Prior Seasonal Influenza Vaccination at 21 Days Post IIV4 Vaccination, Per-Protocol Population\*
- Table 67: Summary of Neutralizing Antibody Against Seasonal IIV4 Strains by Treatment Group and Prior Seasonal Influenza Vaccination at 180 Days Post IIV4 Vaccination, Per-Protocol Population

Table 68: Logistic Regression Model to Evaluate the Relationship of Administration Schedule with HAI Seroconversion Against 2017 A/H7N9 at 21 Days post Second Dose of AS03 adjuvanted A/H7N9 Vaccine, Per Protocol Population\*

| Model Parameter | Parameter Category | Parameter Estimate | SE | p-value | Odds Ratio | 95%CI |
|---|---|---|---|---|---|---|
| Intercept | N/A | XXX.X | XXX.X | X.XXX | 1 | • |
| Treatment | Simultaneous<br>Administration<br>(reference) | - | - | - | - | - |
| | Sequential<br>Administration | XXX.X | XXX.X | X.XXX | XX.X | XX.X-XX.X |

N = XX (Number of subjects in the Per Protocol Population)

- Table 69: Logistic Regression Model to Evaluate the Relationship of Administration Schedule with HAI Seroconversion Against 2017 A/H7N9 at 180 Days Post Second Dose of AS03 adjuvanted A/H7N9 Vaccine, Per Protocol Population \*
- Table 70: Logistic Regression Model to Evaluate the Relationship of Administration Schedule with Neut Seroconversion Against 2017 A/H7N9 at 21 Days Post Second Dose of AS03 adjuvanted A/H7N9 Vaccine, Per Protocol Population
- Table 71: Logistic Regression Model to Evaluate the Relationship of Administration Schedule with Neut Seroconversion Against 2017 A/H7N9 at 180 Days Post Second Dose of AS03 adjuvanted A/H7N9 Vaccine, Per Protocol Population

n = XX (number of subjects with results available at 21 days post second dose of AS03 adjuvanted A/H7N9 IIV in the per protocol population).

XX subjects missing covariate data were excluded from this analysis.

Table 72: Logistic Regression Model to Evaluate the Relationship of Administration Schedule with HAI Seroconversion Against Seasonal IIV4 Strains at 21 Days post IIV4 Vaccination, Per Protocol Population\*

| Model Parameter | Parameter Category | Parameter Estimate | SE | p-value | Odds Ratio | 95%CI |
|---|---|---|---|---|---|---|
| A/Michigan/45/2015 X-275 (H1N1) | | | | | | |
| Intercept | N/A | xxx.x | XXX.X | x.xxx | - | - |
| Treatment | Simultaneous<br>Administration<br>(reference) | - | - | - | - | - |
| | Sequential<br>Administration | XXX.X | XXX.X | X.XXX | XX.X | XX.X-XX.X |
| | IIV4 Only | xxx.x | xxx.x | x.xxx | XX.X | xx.x-xx.x |

#### [Repeat for all IIV4 Strains]

- Table 73: Logistic Regression Model to Evaluate the Relationship of Administration Schedule with HAI Seroconversion Against Seasonal IIV4 Strains at 180 Days Post IIV4 Vaccination, Per Protocol Population
- Table 74: Logistic Regression Model to Evaluate the Relationship of Administration Schedule with Neut Scroconversion Against Seasonal IIV4 Strains at 21 Days Post IIV4 Vaccination, Per Protocol Population\*
- Table 75: Logistic Regression Model to Evaluate the Relationship of Administration Schedule with Neut Seroconversion Against Seasonal IIV4 Strains at 180 Days Post IIV4 Vaccination, Per Protocol Population

N = XX (Number of subjects in the Per Protocol Population)

n = XX (number of subjects with results available at 21 days post IIV4 vaccination in the per protocol population).

XX subjects missing covariate data were excluded from this analysis.

Table 76: Logistic Regression Model to Evaluate the Relationship of Administration Schedule with HAI Seroconversion Against 2017 A/H7N9 at 21 Days Post Second Dose of AS03 adjuvanted A/H7N9 Vaccine, Adjusted for Baseline Covariates, Per Protocol Population\*

| Model Parameter | Parameter Category | Parameter Estimate | SE | p-value | Odds Ratio | 95%CI |
|---|---|---|---|---|---|---|
| Intercept | N/A | xxx.x | xxx.x | x.xxx | - | - |
| Treatment | Simultaneous Administration (reference) | - | - | - | - | - |
| | Sequential Administration | xxx.x | xxx.x | x.xxx | XX.X | xx.x-xx.x |
| Age (years) | N/A | xxx.x | XXX.X | x.xxx | xx.x | xx.x-xx.x |
| Sex | Female (reference) | - | - | - | - | - |
| | Male | xxx.x | XXX.X | x.xxx | XX.X | XX.X-XX.X |
| BMI | <30 (reference) | - | - | - | - | - |
| | ≥30 | xxx.x | xxx.x | x.xxx | XX.X | XX.X-XX.X |
| | Did Not Receive 2016-2017<br>Seasonal Influenza Vaccine<br>(reference) | - | - | - | - | - |
| | Received 2016-2017 Seasonal<br>Influenza Vaccine | XXX.X | XXX.X | x.xxx | XX.X | xx.x-xx.x |

N = XX (number of subjects in the Per Protocol Population)

n= XX (number of subjects with results available at 21 days post second dose of AS03 adjuvanted A/H7N9 IIV in the per protocol population.)

XX subjects missing covariate data were excluded from this analysis.

- Table 77: Logistic Regression Model to Evaluate the Relationship of Administration Schedule with HAI Seroconversion Against 2017 A/H7N9 at 180 Days Post Second Dose of AS03 adjuvanted A/H7N9 Vaccine, Adjusted for Baseline Covariates, Per Protocol Population
- Table 78: Logistic Regression Model to Evaluate the Relationship of Administration Schedule with Neut Seroconversion Against 2017 A/H7N9 at 21 Days Post Second Dose of AS03 adjuvanted A/H7N9 Vaccine, Adjusted for Baseline Covariates, Per Protocol Population\*
- Table 79: Logistic Regression Model to Evaluate the Relationship of Administration Schedule with Neut Seroconversion Against 2017 A/H7N9 at 180 Days Post Second Dose of AS03 adjuvanted A/H7N9 Vaccine, Adjusted for Baseline Covariates, Per Protocol Population

Table 80: Logistic Regression Model to Evaluate the Relationship of Administration Schedule with HAI Seroconversion Against Seasonal IIV4 Strains at 21 Days Post IIV4 Vaccination, Adjusted for Baseline Covariates, Per Protocol Population\*

| Model Parameter | Parameter Category | Parameter Estimate | SE | p-value | Odds Ratio | 95%CI |
|---|---|---|---|---|---|---|
| A/Michigan/45/2015 X-275 | 5 (H1N1) | | | | | |
| Intercept | N/A | xxx.x | XXX.X | x.xxx | - | - |
| Treatment | Simultaneous<br>Administration<br>(reference) | - | - | - | - | - |
| | Sequential<br>Administration | XXX.X | XXX.X | X.XXX | XX.X | XX.X-XX.X |
| | IIV4 Only | XXX.X | xxx.x | x.xxx | xx.x | XX.X-XX.X |
| Age (years) | N/A | xxx.x | xxx.x | x.xxx | xx.x | xx.x-xx.x |
| Sex | Female (reference) | - | - | - | - | - |
| | Male | xxx.x | XXX.X | x.xxx | xx.x | xx.x-xx.x |
| BMI | <30 (reference) | - | - | - | - | - |
| | ≥30 | xxx.x | XXX.X | x.xxx | xx.x | xx.x-xx.x |
| Prior Receipt of Influenza<br>Vaccine | Did Not Receive 2016-<br>2017 Seasonal Influenza<br>Vaccine (reference) | - | - | - | - | - |
| | Received 2016-2017<br>Seasonal Influenza<br>Vaccine | xxx.x | xxx.x | x.xxx | xx.x | XX.X-XX.X |

#### [Repeat for all IIV4 Strains]

N = XX (Number of subjects in the Per Protocol Population)

n = XX (number of subjects with results available at 21 days post IIV4 vaccination in the per protocol population).

XX subjects missing covariate data were excluded from this analysis.

- Table 81: Logistic Regression Model to Evaluate the Relationship of Administration Schedule with HAI Seroconversion Against Seasonal IIV4 Strains at 180 Days Post IIV4 Vaccination, Adjusted for Baseline Covariates, Per Protocol Population
- Table 82: Logistic Regression Model to Evaluate the Relationship of Administration Schedule with Neut Seroconversion Against Seasonal IIV4 Strains at 21 Days Post IIV4 Vaccination, Adjusted for Baseline Covariates, Per Protocol Population\*
- Table 83: Logistic Regression Model to Evaluate the Relationship of Administration Schedule with Neut Seroconversion Against Seasonal IIV4 Strains at 180 Days Post IIV4 Vaccination, Adjusted for Baseline Covariates, Per Protocol Population

Table 84: Multiple Linear Regression Model to Evaluate the Relationship of Administration Schedule with Log-Adjusted HAI Titer against 2017 A/H7N9 at 21 Days Post Second Dose of AS03 adjuvanted A/H7N9 Vaccine, Per Protocol Population\*

| Model Parameter | Parameter Category | Parameter Estimate | SE | 95%CI | p-value |
|---|---|---|---|---|---|
| Intercept | N/A | XXX.X | XXX.X | - | X.XXX |
| Treatment | Simultaneous<br>Administration (reference) | • | - | - | - |
| | Sequential Administration | xxx.x | xxx.x | XX.X-XX.X | x.xxx |

N = XX (Number of subjects in the Per Protocol Population)

- Table 85: Multiple Linear Regression Model to Evaluate the Relationship of Administration Schedule with Log-Adjusted HAI Titer against 2017 A/H7N9 at 180 Days Post Second Dose of AS03 adjuvanted A/H7N9 Vaccine, Per Protocol Population
- Table 86: Multiple Linear Regression Model to Evaluate the Relationship of Administration Schedule with Log-Adjusted Neut Titer against 2017 A/H7N9 at 21 Days Post Second Dose of AS03 adjuvanted A/H7N9 Vaccine, Per Protocol Population\*
- Table 87: Multiple Linear Regression Model to Evaluate the Relationship of Administration Schedule with Log-Adjusted Neut Titer against 2017 A/H7N9 at 180 Days Post Second Dose of AS03 adjuvanted A/H7N9 Vaccine, Per Protocol Population

n = XX (number of subjects with results available at 21 days post second dose of AS03 adjuvanted A/H7N9 IIV in the per protocol population.)

XX subjects missing covariate data were excluded from this analysis.

Table 88: Multiple Linear Regression Model to Evaluate the Relationship of Administration Schedule with Log-Adjusted HAI Titer against Seasonal IIV4 Strains at 21 Days Post IIV4 Vaccination, Per Protocol Population\*

| Model Parameter | Parameter Category | Parameter Estimate | SE | 95%CI | p-value |
|---|---|---|---|---|---|
| A/Michigan/45/2015 X-275 (H1N1) | | | | | |
| Intercept | N/A | XXX.X | xxx.x | - | x.xxx |
| Treatment | Simultaneous<br>Administration (reference) | • | - | - | - |
| | Sequential Administration | XXX.X | XXX.X | XX.X-XX.X | x.xxx |
| | IIV4 Only | XXX.X | xxx.x | XX.X-XX.X | x.xxx |

#### [Repeat for all IIV4 Strains]

- Table 89: Multiple Linear Regression Model to Evaluate the Relationship of Administration Schedule with Log-Adjusted HAI Titer against Seasonal IIV4 Strains at 180 Days Post IIV4 Vaccination, Per Protocol Population
- Table 90: Multiple Linear Regression Model to Evaluate the Relationship of Administration Schedule with Log-Adjusted Neut Titer against Seasonal IIV4 Strains at 21 Days Post IIV4 Vaccination, Per Protocol Population\*
- Table 91: Multiple Linear Regression Model to Evaluate the Relationship of Administration Schedule with Log-Adjusted Neut Titer against Seasonal IIV4 Strains at 180 Days Post IIV4 Vaccination, Per Protocol Population

N = XX (Number of subjects in the Per Protocol Population)

n = XX (number of subjects with results available at 21 days post IIV4 vaccination in the per protocol population).

XX subjects missing covariate data were excluded from this analysis.

Table 92: Multiple Linear Regression Model to Evaluate the Relationship of Administration Schedule with Log-Adjusted HAI Titer against 2017 A/H7N9 at 21 Days Post Second Dose of AS03 adjuvanted A/H7N9 Vaccine, Adjusted for Baseline Covariates, Per Protocol Population\*

| Model Parameter | Parameter Category | Parameter Estimate | SE | 95%CI | p-value |
|---|---|---|---|---|---|
| Intercept | N/A | XXX.X | xxx.x | - | X.XXX |
| Treatment | Simultaneous<br>Administration (reference) | - | - | - | - |
| | Sequential Administration | xxx.x | XXX.X | XX.X-XX.X | x.xxx |
| Age (years) | N/A | xxx.x | XXX.X | XX.X-XX.X | x.xxx |
| Sex | Female (reference) | - | - | - | - |
| | Male | xxx.x | XXX.X | XX.X-XX.X | x.xxx |
| BMI | <30 (reference) | - | - | - | - |
| | ≥30 | XXX.X | XXX.X | XX.X-XX.X | x.xxx |
| Prior Receipt of Influenza<br>Vaccine | Did Not Receive 2016-2017<br>Seasonal Influenza Vaccine<br>(reference) | - | - | - | - |
| | Received 2016-2017<br>Seasonal Influenza Vaccine | XXX.X | XXX.X | XX.X-XX.X | X.XXX |

N = XX (Number of subjects in the Per Protocol Population)

- Table 93: Multiple Linear Regression Model to Evaluate the Relationship of Administration Schedule with Log-Adjusted HAI Titer at 180 Days Post Second Dose of AS03 adjuvanted A/H7N9 Vaccine, Adjusted for Baseline Covariates, Per Protocol Population
- Table 94: Multiple Linear Regression Model to Evaluate the Relationship of Administration Schedule with Log-Adjusted Neut Titer at 21 Days Post Second Dose of AS03 adjuvanted A/H7N9 Vaccine, Adjusted for Baseline Covariates, Per Protocol Population\*
- Table 95: Multiple Linear Regression Model to Evaluate the Relationship of Administration Schedule with Log-Adjusted Neut Titer at 180 Days Post Second Dose of AS03 adjuvanted A/H7N9 Vaccine, Adjusted for Baseline Covariates, Per Protocol Population

n = XX (number of subjects with results available at 21 days post IIV4 vaccination in the per protocol population).

XX subjects missing covariate data were excluded from this analysis.

Table 96: Multiple Linear Regression Model to Evaluate the Relationship of Administration Schedule with Log-Adjusted HAI Titer against Seasonal IIV4 Strains at 21 Days Post IIV4 Vaccination, Adjusted for Baseline Covariates, Per Protocol Population\*

| <b>Model Parameter</b> | | Parameter Estimate | SE | 95%CI | p-value |
|---|---|---|---|---|---|
| A/Michigan/45/2015 X-275 | (H1N1) | | | | |
| Intercept | N/A | XXX.X | XXX.X | - | X.XXX |
| Treatment | Simultaneous<br>Administration (reference) | - | - | - | - |
| | Sequential Administration | xxx.x | xxx.x | XX.X-XX.X | x.xxx |
| | IIV4 Only | xxx.x | XXX.X | XX.X-XX.X | X.XXX |
| Age (years) | N/A | xxx.x | xxx.x | XX.X-XX.X | x.xxx |
| Sex | Female (reference) | - | - | - | - |
| | Male | xxx.x | xxx.x | XX.X-XX.X | x.xxx |
| ВМІ | <30 (reference) | - | - | - | - |
| | ≥30 | XXX.X | XXX.X | XX.X-XX.X | x.xxx |
| Prior Receipt of Influenza<br>Vaccine | a Did Not Receive 2016-2017<br>Seasonal Influenza Vaccine<br>(reference) | - | - | - | - |
| | Received 2016-2017<br>Seasonal Influenza Vaccine | XXX.X | XXX.X | XX.X-XX.X | X.XXX |

### [Repeat for all IIV4 Strains]

N = XX (Number of subjects in the Per Protocol Population)

n = XX (number of subjects with results available at 21 days post IIV4 vaccination in the per protocol population).

XX subjects missing covariate data were excluded from this analysis.

- Table 97: Multiple Linear Regression Model to Evaluate the Relationship of Administration Schedule with Log-Adjusted HAI Titer against Seasonal IIV4 Strains at 180 Days Post IIV4 Vaccination, Adjusted for Baseline Covariates, Per Protocol Population
- Table 98: Multiple Linear Regression Model to Evaluate the Relationship of Administration Schedule with Log-Adjusted Neut Titer against Seasonal IIV4 Strains at 21 Days Post IIV4 Vaccination, Adjusted for Baseline Covariates, Per Protocol Population
- Table 99: Multiple Linear Regression Model to Evaluate the Relationship of Administration Schedule with Log-Adjusted Neut Titer against Seasonal IIV4 Strains at 180 Days Post IIV4 Vaccination, Adjusted for Baseline Covariates, Per Protocol Population

# 14.3 Safety Data

# 14.3.1 Displays of Adverse Events

Table 100: Overall Summary of Adverse Events, Safety Population\*

| | Sin<br>Adn | Group 1:<br>Simultaneous<br>Administration<br>(N=X) | | Group 2:<br>Sequential<br>Administration<br>(N=X) | | Group 3:<br>IIV4 Only<br>(N=X) |
|---|---|---|---|---|---|---|
| Subjects <sup>a</sup> with | n | % | n | % | n | % |
| At least one local solicited adverse event | X | X | X | X | X | X |
| At least one systemic solicited adverse event | X | X | X | X | x | X |
| At least one unsolicited adverse event | X | X | X | X | X | X |
| At least one related unsolicited adverse event | X | X | x | X | x | X |
| Mild (Grade 1) | x | X | X | x | X | X |
| Moderate (Grade 2) | x | X | X | x | X | X |
| Severe (Grade 3) | X | X | X | x | X | X |
| Not yet assessed | | | | | | |
| At least one severe (Grade 3) unsolicited adverse event | X | X | X | X | X | X |
| Related | X | X | X | X | X | X |
| Unrelated | x | X | X | x | X | X |
| Not yet assessed | | | | | | |
| At least one serious adverse event <sup>b</sup> | X | X | X | X | x | X |
| At least one related, serious adverse event | X | X | X | x | X | X |
Table 100: Overall Summary of Adverse Events, Safety Population (continued)

| | Si | Group 1:<br>multaneous<br>ministration<br>(N=X) | Seq<br>Admir | oup 2:<br>uential<br>nistration<br>N=X) | IIV | oup 3:<br>4 Only<br>V=X) |
|---|---|---|---|---|---|---|
| Subjects <sup>a</sup> with | n | % | n | % | n | % |
| At least one adverse event leading to early termination <sup>c</sup> | Х | X | X | Х | Х | X |
| At least one medically attended adverse event | X | X | X | X | x | X |
| At least one new onset chronic medical condition | X | Х | X | X | X | X |
| At least one potentially immune mediated medical condition | X | Х | X | X | X | X |

N = Number of subjects in the safety population.

a Subjects are counted once for each category regardless of the number of events.

b A listing of Serious Adverse Events is included in Table 126

c As reported on the Adverse Event eCRF

Table 101: Number of Adverse Events Occurring in 5% of Subjects in Any Treatment Group by MedDRA® System Organ Class and Preferred Term, and Treatment Group - Safety Population

| | | Si | Group 1:<br>multaneo<br>ministrat<br>(N=X) | us | | Group 2:<br>ial Admin<br>(N=X) | | | y | |
|---|---|---|---|---|---|---|---|---|---|---|
| MedDRA System Organ Class | Preferred Term | n | % | Events | n | % | Events | n | % | Events |
| | Serious | Adverse E | vents | | | | | | | |
| All | All | X | X | X | X | X | x | X | X | X |
| SOC1 | PT1 | x x | | X | X | X | X | X | X | X |
| Etc. | Etc. | X | X | X | X | X | x | X | X | X |
| | Other (Non-ser | rious) Adv | erse Event | ts | | | | | | |
| All | All | X | X | X | X | X | X | X | X | X |
| SOC1 | PT1 | X | X | X | X | х | X | X | х | х |
| Etc | Etc | X | X | X | X | X | X | X | X | х |

N = number of subjects in the safety population. n= number of subjects reporting event. Events = total frequency of events reported. MedDRA Version X.X.

#### 14.3.1.1 Solicited Adverse Events

Table 102: Number and Percentage of Subjects Experiencing Solicited Events with 95% Confidence Intervals by Symptom and Treatment Group (Safety Population) – Post Any Study Dose\*

| | Grou<br>Simultaneous A<br>(N= | up 1:<br>Administration<br>=X) | Grou<br>Sequential Ac<br>(N= | dministration | Group 3:<br>IIV4 Only<br>(N=X) | |
|---|---|---|---|---|---|---|
| Symptom | n | %<br>(95% CI) | n | %<br>(95% CI) | n | %<br>(95% CI) |
| Any Symptom | X | xx<br>(xx-xx) | X | xx<br>(xx-xx) | X | xx<br>(xx-xx) |
| Any Systemic Symptom | | | | | | |
| Fever | | | | | | |
| Feverishness | | | | | | |
| Fatigue | | | | | | |
| Malaise | | | | | | |
| Myalgia | | | | | | |
| Arthralgia | | | | | | |
| Headache | | | | | | |
| Nausea | | | | | | |
| Any Local Symptom | | | | | | |
| Pain | | | | | | |
| Tenderness | | | | | | |
| Pruritus | | | | | | |
| Ecchymosis | | | | | | |
| Ecchymosis (measurement) | | | | | | |
| Erythema | | | | | | |
| Erythema (measurement) | | | | | | |
| Induration/Swelling | | | | | | |

Table 102: Number and Percentage of Subjects Experiencing Solicited Events with 95% Confidence Intervals by Symptom and Treatment Group (Safety Population) – Post Any Study Dose (continued)

| | Grou<br>Simultaneous A<br>(N= | 1 | | up 2:<br>dministration<br>=X) | IIV4 | up 3:<br>Only<br>=X) |
|---|---|---|---|---|---|---|
| Symptom | n | %<br>(95% CI) | n | %<br>(95% CI) | n | %<br>(95% CI) |
| Induration/Swelling (measurement) | | | | | | |
| N = Number of subjects in the Safety F | Onulation who recei | ved any dose | | | | |

N = Number of subjects in the Safety Population who received any dose.

95% CI estimated using Clopper-Pearson exact method

Tables with similar format:

Table 103: Number and Percentage of Subjects Experiencing Solicited Events with 95% Confidence Intervals by Symptom and Treatment Group (Safety Population) – Post Study Dose 1\*

[Footnote update] N = Number of subjects in the Safety Population who received the first dose.

Table 104: Number and Percentage of Subjects Experiencing Solicited Events with 95% Confidence Intervals by Symptom and Treatment Group (Safety Population) – Post Study Dose 2\*

[Footnote update] N = Number of subjects in the Safety Population who received the second dose.

Table 105: Number and Percentage of Subjects Experiencing Solicited Events with 95% Confidence Intervals by Symptom and Treatment Group (Safety Population) – Post Study Dose 3\*

[Footnote update] N = Number of subjects in the Safety Population who received the third dose.

Table 106: Logistic Regression Model to Evaluate the Relationship of Treatment with Reporting Any Local Event Post Any Study Dose (Safety Population) \*

| Model Parameter | Parameter Category | Parameter Estimate | SE | p-value | Odds Ratio | 95%CI |
|---|---|---|---|---|---|---|
| Intercept | N/A | xxx.x | XXX.X | x.xxx | - | - |
| Treatment | Simultaneous<br>Administration<br>(reference) | - | - | - | - | - |
| | Sequential<br>Administration | XXX.X | XXX.X | X.XXX | XX.X | XX.X-XX.X |
| | IIV4 Only | xxx.x | XXX.X | x.xxx | XX.X | XX.X-XX.X |

Table with similar format:

Table 107: Logistic Regression Model to Evaluate the Relationship of Treatment with Reporting Any Systemic Event Post Any Study Dose (Safety Population) \*

Table 108: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Maximum Severity and Treatment Group (Safety Population) – Post Any Study Dose\*

| | | Simulta | Group 1:<br>neous Administration<br>(N=X) | Sequential | roup 2:<br>Administration<br>N=X) | Group 3:<br>IIV4 Only<br>(N=X) | |
|---|---|---|---|---|---|---|---|
| Symptom | Severity | n | %<br>(95% CI) | n | %<br>(95% CI) | n | %<br>(95% CI) |
| Any Symptom | None | х | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) |
| | Mild | | | | | | |
| | Moderate | | | | | | |
| | Severe | | | | | | |
| Any Systemic Symptom | None | Х | xx (xx-xx) | X | xx (xx-xx) | X | xx (xx-xx) |
| | Mild | | | | | | |
| | Moderate | | | | | | |
| | Severe | | | | | | |
| Fever | None | | | | | | |
| | Mild | | | | | | |
| | Moderate | | | | | | |
| | Severe | | | | | | |
| Feverishness | None | | | | | | |
| | Mild | | | | | | |
| | Moderate | | | | | | |
| | Severe | | | | | | |
| Fatigue | None | | | | | | |
| | Mild | | | | | | |
| | Moderate | | | | | | |
| | Severe | | | | | | |
| Malaise | None | | | | | | |
| | Mild | | | | | | |

Table 108: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Maximum Severity and Treatment Arm (Safety Population) – Post Any Study Dose (continued)

| | | Simulta | Group 1:<br>neous Administration<br>(N=X) | Sequential A | oup 2:<br>Administration<br>V=X) | Group 3:<br>IIV4 Only<br>(N=X) | |
|---|---|---|---|---|---|---|---|
| Symptom | Severity | n | %<br>(95% CI) | n | %<br>(95% CI) | n | %<br>(95% CI) |
| | Moderate | | | | | | |
| | Severe | | | | | | |
| Myalgia | None | | | | | | |
| | Mild | | | | | | |
| | Moderate | | | | | | |
| | Severe | | | | | | |
| Arthralgia | None | | | | | | |
| | Mild | | | | | | |
| | Moderate | | | | | | |
| | Severe | | | | | | |
| Headache | None | | | | | | |
| | Mild | | | | | | |
| | Moderate | | | | | | |
| | Severe | | | | | | |
| Nausea | None | | | | | | |
| | Mild | | | | | | |
| | Moderate | | | | | | |
| | Severe | | | | | | |
| Any Local Symptom | None | | | | | | |
| | Mild | | | | | | |
| | Moderate | | | | | | |
| | Severe | | | | | | |

Table 108: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Maximum Severity and Treatment Arm (Safety Population) – Post Any Study Dose (continued)

| | | Simultar | Group 1:<br>neous Administration<br>(N=X) | Gro<br>Sequential A<br>(N | oup 2:<br>Administration<br>N=X) | Group 3:<br>IIV4 Only<br>(N=X) | |
|---|---|---|---|---|---|---|---|
| Symptom | Severity | n | %<br>(95% CI) | n | %<br>(95% CI) | n | %<br>(95% CI) |
| Pain | None | | | | | | |
| | Mild | | | | | | |
| | Moderate | | | | | | |
| | Severe | | | | | | |
| Tenderness | None | | | | | | |
| | Mild | | | | | | |
| | Moderate | | | | | | |
| | Severe | | | | | | |
| Pruritus | None | | | | | | |
| | Mild | | | | | | |
| | Moderate | | | | | | |
| | Severe | | | | | | |
| Ecchymosis | None | | | | | | |
| | Mild | | | | | | |
| | Moderate | | | | | | |
| | Severe | | | | | | |
| Ecchymosis (measurement) | None | | | | | | |
| | Mild | | | | | | |
| | Moderate | | | | | | |
| | Severe | | | | | | |
| Erythema | None | | | | | | |
| | Mild | | | | | | |

Table 108: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Maximum Severity and Treatment Arm (Safety Population) – Post Any Study Dose (continued)

| | | Simultai | Group 1:<br>neous Administration<br>(N=X) | Sequential | oup 2:<br>Administration<br>N=X) | Group 3:<br>IIV4 Only<br>(N=X) | |
|---|---|---|---|---|---|---|---|
| Symptom | Moderate Severe Pasurement) None Mild Moderate Severe Velling None Mild Moderate Severe Velling Moderate Severe | n | %<br>(95% CI) | n | %<br>(95% CI) | n | %<br>(95% CI) |
| | Moderate | | | | | | |
| | Severe | | | | | | |
| Erythema (measurement) | None | | | | | | |
| | Mild | | | | | | |
| | Moderate | | | | | | |
| | Severe | | | | | | |
| Induration/Swelling | None | | | | | | |
| | Mild | | | | | | |
| | Moderate | | | | | | |
| | Severe | | | | | | |
| Induration/Swelling (measurement) | None | | | | | | |
| | Mild | | | | | | |
| | Moderate | | | | | | |
| NI NI 1 C 1' 4 ' 41 | Severe | | | | | | |

N = Number of subjects in the Safety Population who received any study dose.

Severity is the maximum severity reported over all solicited symptoms post dosing for each subject.

<sup>95%</sup> CI estimated using Clopper-Pearson exact method

Tables with similar format:

Table 109: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Maximum Severity and Treatment Group (Safety Population) – Post Study Dose 1\*

[Footnote Update] N = Number of subjects in the Safety Analysis Population who received the first study dose.

Table 110: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Maximum Severity and Treatment Group (Safety Population) – Post Study Dose 2\*

[Footnote Update] N = Number of subjects in the Safety Analysis Population who received the second study dose.

Table 111: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Maximum Severity and Treatment Group (Safety Population) – Post Study Dose 3\*

[Footnote Update] N = Number of subjects in the Safety Analysis Population who received the third study dose.

Table 112: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Severity, Day Post Dose, and Treatment Group (Safety Population) – Post Any Study Dose

| | G | | <u> </u> | | ost- | _ | | | | _ | | _ | | _ | | | | | | | • |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Symptom | Severity | | -Dose | | ose | | ay 1 | | y 2 | | y 3 | | y 4 | | y 5 | | ay 6 | | ay 7 | | y 8+ |
| | | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| | | 1 | Gro | up 1: | Simu | ıltane | ous A | dminis | tration | ı (N= | (X) | 1 | 1 | | ı | 1 | 1 | | ı | | |
| Any Symptom | None | | | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | |
| Any Systemic Symptom | None | | | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | |
| Fever | None | | | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | |
| Feverishness | None | | | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | |
| Fatigue | None | | | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | |
| Malaise | None | | | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | | | |

Table 112: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Severity, Day Post Study Vaccination, and Treatment Arm (Safety Population) – Post Any Study Dose (continued)

| Symptom | Severity | Pre- | -Dose | Po<br>Do | ost-<br>ose | Da | ay 1 | Da | ny 2 | Da | ıy 3 | Da | ıy 4 | Da | ny 5 | Da | ny 6 | Da | ıy 7 | Da | y 8+ |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| | Moderate | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | |
| Myalgia | None | | | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | |
| Arthralgia | None | | | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | |
| Headache | None | | | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | |
| Nausea | None | | | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | |
| Any Local Symptom | None | | | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | |
| Pain | None | | | | | | | | | | | | | | | | | | | | |

Table 112: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Severity, Day Post Study Vaccination, and Treatment Arm (Safety Population) – Post Any Study Dose (continued)

| Symptom | Severity | Pre- | Dose | | ost-<br>ose | Da | ay 1 | Da | ny 2 | Da | ıy 3 | Da | ıy 4 | Da | ıy 5 | Da | ıy 6 | Da | ıy 7 | Day | y 8+ |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| | Mild | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | |
| Tenderness | None | | | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | |
| Pruritus | None | | | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | |
| Ecchymosis | None | | | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | |
| Ecchymosis (measurement) | None | | | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | |
| Erythema | None | | | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | |

Table 112: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Severity, Day Post Study Vaccination, and Treatment Arm (Safety Population) – Post Any Study Dose (continued)

| Symptom | Severity | Pre- | -Dose | | ost-<br>ose | Da | ay 1 | Da | y 2 | Da | ıy 3 | Da | ıy 4 | Da | ıy 5 | Da | ıy 6 | Da | ıy 7 | Da | y 8+ |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| Erythema (measurement) | None | | | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | |
| duration/Swelling | None | | | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | |
| Induration/Swelling (measurement) | None | | | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | |
| N = Number of subjects in the Safety A | | | | | | | | tmen | | | | | | | | | 2 1 | | | | |

N = Number of subjects in the Safety Analysis Population who received the specified dose. Severity is the maximum severity reported post dosing for each subject for each day.

Tables with similar format:

- Table 113: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Severity, Day Post Dose, and Treatment Group (Safety Population) Post Study Dose 1
- Table 114: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Severity, Day Post Dose, and Treatment Group (Safety Population) Post Study Dose 2
- Table 115: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Severity, Day Post Dose, and Treatment Group (Safety Population) Post Study Dose 3

Table 116: Comparison of the Number and Percentage of Subjects Experiencing Solicited Systemic Events by Dose and Treatment Group – Safety Population

| | | Subjects with No<br>Symptoms | Subjects with Mild or Greater<br>Symptoms | Total Number of Subjects<br>n (Percent)<br>[p-value*] |
|---|---|---|---|---|
| | | Study Dose 1 vs Stu | dy Dose 2 | |
| Group 1: | Subjects with No Symptoms | x (%) | x (%) | x (%) |
| Simultaneous<br>Administration<br>(N=X) | Subjects with Mild or Greater<br>Symptoms | x (%) | x (%) | x (%) |
| ` , | Total Number of Subjects | x (%) | x (%) | x (100%)<br>[0.xxx] |
| Group 2: | Subjects with No Symptoms | x (%) | x (%) | x (%) |
| Sequential<br>Administration<br>(N=X) | Subjects with Mild or Greater<br>Symptoms | x (%) | x (%) | x (%) |
| (*) | Total Number of Subjects | x (%) | x (%) | x (100%)<br>[0.xxx] |
| | | Study Dose 1 vs Stu | dy Dose 3 | |
| Group 2: | Subjects with No Symptoms | x (%) | x (%) | x (%) |
| Sequential<br>Administration<br>(N=X) | Subjects with Mild or Greater<br>Symptoms | x (%) | x (%) | x (%) |
| | Total Number of Subjects | x (%) | x (%) | x (100%)<br>[0.xxx] |
| | | Study Dose 2 vs Stu | dy Dose 3 | |
| Group 2: | Subjects with No Symptoms | x (%) | x (%) | x (%) |
| Sequential<br>Administration<br>(N=X) | Subjects with Mild or Greater<br>Symptoms | x (%) | x (%) | x (%) |
| , | Total Number of Subjects | x (%) | x (%) | x (100%)<br>[0.xxx] |

Note: Denominators for percentages are the number of subjects in the safety population who received both the first and second study dose. Subjects who did not receive both indicated doses are not included in this table. [x] subjects did not receive the second dose and [x] subjects did not receive the third dose.

\* P-value is calculated from McNemar's test for each treatment group.

Table with similar format:

Table 117: Comparison of the Number and Percentage of Subjects Experiencing Solicited Local Events by Dose and Treatment Group – Safety Population

#### 14.3.1.2 Unsolicited Adverse Events

Table 118: Number and Percentage of Subjects Experiencing Unsolicited Adverse Events with 95% Confidence Intervals by MedDRA® System Organ Class and Preferred Term, and Treatment Group – Safety Population\*

| MedDRA® System Organ<br>Class | MedDRA® Preferred<br>Term | Simultaneo | Group 1:<br>ous Administration<br>(N=X) | | Group 2:<br>al Administration<br>(N=X) | | Group 3:<br>IV4 Only<br>(N=X) |
|---|---|---|---|---|---|---|---|
| | | n | %<br>(95% CI) | n | %<br>(95% CI) | n | %<br>(95% CI) |
| Any SOC | Any PT | х | xx<br>(xx-xx) | х | xx<br>(xx-xx) | Х | xx<br>(xx-xx) |
| [SOC 1] | Any PT | | | | | | |
| | [PT 1] | | | | | | |
| | [PT 2] | | | | | | |
| [SOC 2] | Any PT | | | | | | |
| | [PT 1] | | | | | | |
| N. A. M. A. C. H. C. H. C. | [PT 2] | . 1 1 | mi' . 11 | 1 1 | | | 1 1 |

Note: N = number of subjects in the Safety Analysis Population who received any dose. This table presents number and percentage of subjects. A subject is only counted once per PT.

Table 119: Number and Percentage of Subjects Experiencing Unsolicited Adverse Events by MedDRA® System Organ Class and Preferred Term, Maximum Severity, Relationship, and Treatment Group – Safety Population\*

| Treatment Group | MedDRA® System | MedDRA® Preferred | | Incide | | | Seve | rity [1] | | | Relat | ionship to | Treatm | ent [2] |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Organ Class | Term | ] | nce | M | ild | Mod | lerate | Se | vere | Not F | Related | Rel | ated |
| | | | n | % | n | % | n | % | n | % | n | % | n | % |
| Group 1:<br>Simultaneous<br>Administration<br>(N=X) | Any SOC | Any PT | х | XX | х | XX | х | xx | Х | xx | х | xx | х | XX |
| | [SOC 1] | Any PT | | | | | | | | | | | | |
| | | [PT 1] | | | | | | | | | | | | |
| | | [PT 2] | | | | | | | | | | | | |
| | [SOC 2] | Any PT | | | | | | | | | | | | |
| | | [PT 1] | | | | | | | | | | | | |
| | | [PT 2] | | | | | | | | | | | | |
| Group 2: Sequential<br>Administration<br>(N=X) | Any SOC | Any PT | X | XX | х | XX | Х | xx | х | xx | х | XX | х | XX |
| | [SOC 1] | Any PT | | | | | | | | | | | | |
| | | [PT 1] | | | | | | | | | | | | |
| | | [PT 2] | | | | | | | | | | | | |
| | [SOC 2] | Any PT | | | | | | | | | | | | |
| | | [PT 1] | | | | | | | | | | | | |
| | | [PT 2] | | | | | | | | | | | | |
| Group 3: IIV4 Only (N=X) | Any SOC | Any PT | х | XX | х | XX | Х | XX | х | XX | Х | XX | Х | XX |
| ` | [SOC 1] | Any PT | | | | | | | | | | | | |
| | | [PT 1] | | | | | | | | | | | | |
| | | [PT 2] | | | | | | | | | | | | |

Table 119: Number and Percentage of Subjects Experiencing Unsolicited Adverse Events by MedDRA® System Organ Class and Preferred Term, Maximum Severity, Relationship, and Treatment Group – Safety Population (continued)

| Ī | Treatment Group | MedDRA® System | MedDRA® Preferred | | Incide | | | Sever | ity [1] | | | Relati | onship to | Treatmo | ent [2] |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Organ Class | Term | ] | ıce | M | ild | Mod | erate | Sev | ere | Not R | elated | Rela | ated |
| | | | | n | % | n | % | n | % | n | % | n | % | n | % |
| | | [SOC 2] | Any PT | | | | | | | | | | | | |
| | | | [PT 1] | | | | | | | | | | | | |
| | | | [PT 2] | | | | | | | | | | | | |

Note: N = Number of subjects in the Safety Analysis Population.

<sup>[1]</sup> For severity, a subject is counted once per preferred term and is summarized according to their highest severity.

<sup>[2]</sup> For relationship, a subject is only counted once per preferred term and is summarized according to their closest relationship.

Table 120: Number and Percentage of Subjects Experiencing Non-Serious Related Unsolicited Adverse Events by MedDRA® System Organ Class and Preferred Term, Maximum Severity, and Treatment Group – Safety Population

| Treatment Group | MedDRA® System Organ | MedDRA® Preferred | Any Iı | ıcidence | | | Sever | ity [1] | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | Class | Term | | | M | ild | Mod | lerate | Sev | vere |
| | | | n | % | n | % | n | % | n | % |
| Group 1: Simultaneous<br>Administration<br>(N=X) | Any SOC | Any PT | X | xx | х | xx | х | xx | х | xx |
| | [SOC 1] | Any PT | x | xx | х | XX | х | XX | х | xx |
| | | [PT 1] | | | | | | | | |
| | | [PT 2] | | | | | | | | |
| | [SOC 2] | Any PT | | | | | | | | |
| | | [PT 1] | | | | | | | | |
| | | [PT 2] | | | | | | | | |
| Group 2: Sequential<br>Administration<br>N=X) | Any SOC | Any PT | X | xx | х | xx | х | XX | Х | xx |
| | [SOC 1] | Any PT | X | xx | х | XX | х | xx | х | xx |
| | | [PT 1] | | | | | | | | |
| | | [PT 2] | | | | | | | | |
| | [SOC 2] | Any PT | | | | | | | | |
| | | [PT 1] | | | | | | | | |
| | | [PT 2] | | | | | | | | |
| Group 3: IIV4 Only (N=X) | Any SOC | Any PT | X | xx | Х | xx | х | xx | х | XX |
| | [SOC 1] | Any PT | X | xx | х | xx | х | XX | х | xx |
| | | [PT 1] | | | | | | | | |
| | | [PT 2] | | | | | | | | |
| | [SOC 2] | Any PT | | | | | | | | |

Table 120: Number and Percentage of Subjects Experiencing Non-Serious Related Unsolicited Adverse Events by MedDRA® System Organ Class and Preferred Term, Maximum Severity, and Treatment Group – Safety Population (continued)

| Treatment Group | MedDRA® System Organ | MedDRA® Preferred | Any In | cidence | | | Sever | ity [1] | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | Class | Term | | | Mild | | Mod | erate | Sev | ere |
| | | | n | % | n | % | n | % | n | % |
| | | [PT 1] | | | | | | | | |
| | | [PT 2] | | | | | | | | |

Note: N = Number of subjects in the Safety Analysis Population. This table presents number and percentage of subjects.

<sup>[1]</sup> For severity, a subject is counted once per preferred term and is summarized according to their highest severity.

Table 121: Number and Percentage of Subjects Experiencing Unsolicited Adverse Events Within 21 Days Post Dose by MedDRA® System Organ Class and Preferred Term, Day Post Dose, and Treatment Group – Safety Population

| MedDRA®<br>System Organ | MedDRA® | F | y 1-8<br>Post<br>ose 1 | 1 | ay 9-<br>22<br>Post<br>ose 1 | P | ny 1-<br>22<br>ost<br>ose 1 | Post | y 1-8<br>Dose<br>2 | Post | 9-22<br>Dose<br>2 | Post | 7 1-22<br>t Dose<br>2 | Po | 1-8<br>ost<br>se 3 | Po | 7 1-8<br>ost<br>se 3 | P | 7 1-8<br>ost<br>se 3 | Post | 1-22<br>t Any<br>ose |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Class | Preferred Term | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| | | | | | Grou | ıp 1: | Simult | aneou | s Adm | inistra | tion ( | N=X) | | | | | | | | | |
| Any SOC | Any PT | x | XX | x | XX | X | XX | X | xx | X | xx | x | XX | NA | NA | NA | NA | NA | NA | X | XX |
| [SOC 1] | Any PT | Х | XX | X | XX | X | XX | Х | XX | X | XX | х | XX | NA | NA | NA | NA | NA | NA | X | XX |
| | [PT 1] | X | XX | X | XX | X | XX | X | XX | X | XX | X | XX | NA | NA | NA | NA | NA | NA | X | XX |
| | [PT 2] | Х | XX | X | XX | X | XX | Х | XX | X | XX | х | XX | NA | NA | NA | NA | NA | NA | X | XX |
| [SOC 2] | Any PT | X | XX | X | XX | X | XX | X | XX | X | XX | X | XX | NA | NA | NA | NA | NA | NA | X | XX |
| | [PT 1] | X | XX | X | XX | X | XX | X | XX | X | XX | X | XX | NA | NA | NA | NA | NA | NA | X | XX |
| | [PT 2] | Х | XX | X | XX | X | XX | Х | XX | X | XX | х | XX | NA | NA | NA | NA | NA | NA | X | XX |
| | | | | | Gr | oup 2 | : Sequ | ential | Admir | nistrat | ion (N | =X) | | | | | | | | | |
| Any SOC | Any PT | X | XX | x | XX | X | XX | х | XX | X | XX | x | XX | X | XX | X | XX | Х | xx | X | XX |
| [SOC 1] | Any PT | X | XX | x | XX | x | XX | х | XX | X | XX | x | XX | x | XX | X | XX | х | xx | X | XX |
| | [PT 1] | X | XX | x | XX | X | XX | х | XX | X | XX | x | XX | X | XX | X | XX | х | xx | X | XX |
| | [PT 2] | х | XX | х | XX | х | XX | х | XX | X | XX | x | XX | x | XX | X | XX | х | xx | X | XX |
| [SOC 2] | Any PT | х | XX | х | XX | х | XX | х | XX | X | XX | x | XX | x | XX | X | XX | х | xx | X | XX |
| | [PT 1] | X | XX | x | XX | X | XX | х | XX | X | XX | x | XX | X | XX | X | XX | х | xx | X | XX |
| | [PT 2] | X | XX | X | XX | X | XX | Х | XX | X | XX | X | XX | X | XX | X | XX | х | XX | X | XX |
| | | | | | | | Group | 3: IIV | V4 Onl | y (N= | <b>X</b> ) | | | | | | | | | | |
| Any SOC | Any PT | X | XX | X | XX | X | XX | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | X | XX |
| [SOC 1] | Any PT | X | XX | X | XX | X | XX | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | X | XX |
| | [PT 1] | Х | XX | X | XX | х | XX | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | X | XX |
| | [PT 2] | X | XX | х | XX | X | xx | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | X | XX |

Table 121: Number and Percentage of Subjects Experiencing Unsolicited Adverse Events Within 21 Days Post Dose by MedDRA® System Organ Class and Preferred Term, Day Post Dose, and Treatment Group – Safety Population (continued)

| MedDRA®<br>System Organ | MedDRA® | P | y 1-8<br>Post<br>ose 1 | P | ay 9-<br>22<br>Post<br>ose 1 | P | y 1-<br>22<br>ost<br>ose 1 | Post | 7 1-8<br>Dose<br>2 | | 9-22<br>Dose<br>2 | | 7 1-22<br>t Dose<br>2 | | 7 1-8<br>Ost<br>Se 3 | Po | 7 1-8<br>Ost<br>Se 3 | | 1-8<br>ost<br>se 3 | Post | 1-22<br>Any<br>ose |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Class | Preferred Term | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| [SOC 2] | Any PT | X | XX | X | XX | X | XX | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | X | XX |
| | [PT 1] | X | xx | x | xx | Х | XX | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | X | XX |
| | [PT 2] | X | XX | х | XX | Х | XX | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | х | XX |

Note: N = Number of subjects in the Safety Analysis Population. This table presents number and percentage of subjects. For each time period, a subject is only counted once per PT.

Table 122: Number and Percentage of Subjects Experiencing Non-Serious, Related Unsolicited Adverse Events Within 21 Days Post Dose by MedDRA® System Organ Class and Preferred Term, Dose and Treatment Group – Safety Population

| | | P | y 1-8<br>Post<br>ose 1 | I | ay 9-<br>22<br>Post<br>ose 1 | P | ny 1-<br>22<br>Post<br>ose 1 | Post | v 1-8<br>Dose<br>2 | Post | 9-22<br>Dose<br>2 | Post | 7 1-22<br>t Dose<br>2 | Pe | 7 1-8<br>Ost<br>se 3 | Pe | 7 1-8<br>ost<br>se 3 | Day<br>Po<br>Dos | 7 1-8<br>Ost<br>se 3 | Post | 1-22<br>Any<br>ose |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| MedDRA®<br>System Organ<br>Class | MedDRA®<br>Preferred Term | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| | • | | | | Grou | ıp 1: S | Simult | aneou | s Admi | inistra | tion ( | (N=X) | | | | | | | | | |
| Any SOC | Any PT | х | xx | x | xx | x | xx | x | XX | х | xx | х | XX | NA | NA | NA | NA | NA | NA | х | xx |
| [SOC 1] | Any PT | | | | | | | | | | | | | | | | | | | | |
| | [PT 1] | | | | | | | | | | | | | | | | | | | | |
| | [PT 2] | | | | | | | | | | | | | | | | | | | | |
| [SOC 2] | Any PT | | | | | | | | | | | | | | | | | | | | |
| | [PT 1] | | | | | | | | | | | | | | | | | | | | |
| | [PT 2] | | | | | | | | | | | | | | | | | | | | |
| | | | | | Gr | oup 2 | 2: Sequ | ıential | Admii | nistrat | ion (N | =X) | | | | | | | | | |
| Any SOC | Any PT | х | XX | х | xx | х | xx | х | XX | х | xx | х | XX | х | XX | х | XX | х | XX | X | xx |
| [SOC 1] | Any PT | | | | | | | | | | | | | | | | | | | | |
| | [PT 1] | | | | | | | | | | | | | | | | | | | | |
| | [PT 2] | | | | | | | | | | | | | | | | | | | | |
| [SOC 2] | Any PT | | | | | | | | | | | | | | | | | | | | |
| | [PT 1] | | | | | | | | | | | | | | | | | | | | |
| | [PT 2] | | | | | | | | | | | | | | | | | | | | |
| | | | | | | | Group | 3: IIV | /4 Onl | y (N=) | <b>X</b> ) | | | | | | | | | | |
| Any SOC | Any PT | х | xx | x | xx | x | XX | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | X | xx |
| [SOC 1] | Any PT | | | | | | | | | | | | | | | | | | | | |
| | [PT 1] | | | | | | | | | | | | | | | | | | | | |

| | | P | y 1-8<br>Post<br>ose 1 | P | ny 9-<br>22<br>Post<br>ose 1 | P | ny 1-<br>22<br>Post<br>ose 1 | 7 1-8<br>Dose<br>2 | 9-22<br>Dose<br>2 | 7 1-22<br>t Dose<br>2 | 1-8<br>ost<br>se 3 | Po | 1-8<br>ost<br>se 3 | Pe | 1-8<br>ost<br>se 3 | Day<br>Post<br>Do | Any |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | [PT 2] | | | | | | | | | | | | | | | | |
| [SOC 2] | Any PT | | | | | | | | | | | | | | | | |
| | [PT 1] | | | | | | | | | | | | | | | | |
| | [PT 2] | | | | | | | | | | | | | | | | |

Note: N = Number of subjects in the Safety Analysis Population. This table presents number and percentage of subjects. For each time period, a subject is only counted once per PT.

Table 123: Number of Unsolicited Adverse Events by MedDRA® System Organ Class and Preferred Term, Day Post Dose, and Treatment Group – Safety Population

| | | | Day 1-<br>8<br>Post<br>Dose 1 | Day 9-<br>22<br>Post<br>Dose 1 | Day 1-<br>22<br>Post<br>Dose 1 | Day 1-<br>8<br>Post<br>Dose 2 | Day 9-<br>22<br>Post<br>Dose 2 | Day 1-<br>22<br>Post<br>Dose 2 | Day 1-<br>8<br>Post<br>Dose 3 | Day 9-<br>22<br>Post<br>Dose 3 | Day 1-<br>22<br>Post<br>Dose 3 | Day 1-<br>22<br>Post<br>Any<br>Dose |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Treatment<br>Group | MedDRA® System<br>Organ Class | MedDRA®<br>Preferred Term | # of<br>Events | # of<br>Events | # of<br>Events | # of<br>Events | # of<br>Events | # of<br>Events | # of<br>Events | # of<br>Events | # of<br>Events | # of<br>Events |
| Group 1:<br>Simultaneous<br>Administration<br>(N=X) | Any SOC | Any PT | х | X | X | X | X | х | NA | NA | NA | х |
| | [SOC 1] | Any PT | | | | | | | | | | |
| | | [PT 1] | | | | | | | | | | |
| | | [PT 2] | | | | | | | | | | |
| | [SOC 2] | Any PT | | | | | | | | | | |
| | | [PT 1] | | | | | | | | | | |
| | | [PT 2] | | | | | | | | | | |
| Group 2:<br>Sequential<br>Administration<br>(N=X) | Any SOC | Any PT | х | X | X | X | X | х | х | X | X | X |
| | [SOC 1] | Any PT | | | | | | | | | | |
| | | [PT 1] | | | | | | | | | | |
| | | [PT 2] | | | | | | | | | | |
| | [SOC 2] | Any PT | | | | | | | | | | |
| | | [PT 1] | | | | | | | | | | |
| | | [PT 2] | | | | | | | | | | |
| Group 3:<br>IIV4 Only<br>(N=X) | Any SOC | Any PT | x | X | х | NA | NA | NA | NA | NA | NA | X |

Table 123: Number of Unsolicited Adverse Events by MedDRA® System Organ Class and Preferred Term, Day Post Dose, and Treatment Group – Safety Population (continued)

| | | Day 1-<br>8<br>Post<br>Dose 1 | Day 9-<br>22<br>Post<br>Dose 1 | Day 1-<br>22<br>Post<br>Dose 1 | Day 1-<br>8<br>Post<br>Dose 2 | Day 9-<br>22<br>Post<br>Dose 2 | Day 1-<br>22<br>Post<br>Dose 2 | Day 1-<br>8<br>Post<br>Dose 3 | Day 9-<br>22<br>Post<br>Dose 3 | Day 1-<br>22<br>Post<br>Dose 3 | Day 1-<br>22<br>Post<br>Any<br>Dose |
|---|---|---|---|---|---|---|---|---|---|---|---|
| [SOC 1] | Any PT | | | | | | | | | | |
| | [PT 1] | | | | | | | | | | |
| | [PT 2] | | | | | | | | | | |
| [SOC 2] | Any PT | | | | | | | | | | |
| | [PT 1] | | | | | | | | | | |
| | [PT 2] | | | | | | | | | | |

# 14.3.2 Listings of Serious and Significant Adverse Events

### **Table 124: Listing of Serious Adverse Events \***

[Implementation Note: If the event is ongoing (no stop date), indicate "ongoing" in the "Duration" column. If more than one reason is selected for the reason reported as an SAE, list all reasons in the column, separated by a comma. In the "If Not Related, Alternate Etiology" column, merge the 2 data fields for collecting alternate etiology, separate by a colon. In the CSR, Subject ID should be USUBJID (not PATID) for purposes of deidentification.]

| Adverse<br>Event | Associated with Dose # | # of Days<br>Post<br>Associated<br>Dose<br>(Duration) | # of<br>Days<br>Post<br>Dose the<br>Event<br>Became<br>Serious | Reason<br>Reported<br>as an SAE | Severity | Relationship<br>to Study<br>Treatment | In Not<br>Related,<br>Alternative<br>Etiology | Action<br>Taken with<br>Study<br>Treatment | Subject<br>Discontinued<br>Due to AE | Outcome | MedDRA®<br>Sytem<br>Organ<br>Class | MedDRA®<br>Preferred<br>Term |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject II | D: , Treatmo | ent Group: , | AE Num | ber: | | | | | | | | |
| Comments | s: | | | | | | | | | | | |
| Subject II | ): , Treatmo | ent Group: , | AE Num | ber: | | | | | | | | |
| Comments | : | | | | | | | | | | | |

## **Table 125: Listing of Medically Attended Adverse Events\***

[Implementation Note: If the event is ongoing (no stop date), indicate "ongoing" in the "Duration" column. In the "If Not Related, Alternate Etiology" column, merge the 2 data fields for collecting alternate etiology, separate by a colon.]

| Adverse<br>Event | Associated with Dose # | # of Days Post Associated Dose (Duration) | SAE?<br>Severity | Relationship<br>to Study<br>Treatment | In Not<br>Related,<br>Alternative<br>Etiology | Action<br>Taken<br>with<br>Study<br>Treatment | Subject<br>Discontinued<br>Due to AE | Outcome | MAAE | MedDRA®<br>System<br>Organ<br>Class | MedDRA®<br>Preferred<br>Term |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject II | D: , Treatm | ent Group: | , AE Numb | er: | | | | | | | |
| | | | SAE: No<br>Mild | | | | | | | | |
| Comments | 3: | | | | | | | | | | |
| Subject II | D: , Treatm | ent Group: | , AE Numb | er: | | | | | | | |
| Comments | s: | | | | | | | | | | |

## Tables with similar format:

Table 126: Listing of Potentially Immune Mediated Medical Conditions\*

Table 127: Listing of New Onset Chronic Medical Conditions\*

Table 128: Listing of Non-Serious, Unsolicited, Moderate or Severe Adverse Events\*

14.3.3 Narratives of Deaths, Other Serious and Significant Adverse Events

(not included in SAP, placeholder for the CSR)

# 14.3.4 Displays of Laboratory Results

Table 129: Laboratory Results by Parameter, Maximum Severity, Study Day, and Treatment Group (Safety Population) – All Laboratory Parameters \*

| Treatment Group | Study Day | N | | None | | ild/<br>de 1 | | lerate/<br>ade 2 | | Severe/<br>Grade 3 | Missing | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | n | % | n | % | n | % | n | % | n | % |
| Group 1: | Baseline | х | х | xx | х | XX | Х | xx | х | XX | X | XX |
| Simultaneous<br>Administration | Day 8 | X | х | XX | х | XX | X | xx | X | xx | X | XX |
| (N=X) | Day 22 | X | X | XX | X | XX | X | xx | X | XX | X | XX |
| | Day 29 | X | X | XX | X | XX | X | XX | X | XX | X | XX |
| | Day 43 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA |
| | Day 50 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA |
| | Max Severity Post<br>Baseline | X | X | XX | Х | xx | X | XX | х | xx | X | XX |
| Group 2: Sequential | Baseline | X | x | XX | x | XX | X | xx | X | XX | X | XX |
| Administration (N=X) | Day 8 | X | X | XX | X | XX | X | XX | X | XX | X | XX |
| | Day 22 | X | X | XX | X | XX | X | XX | X | XX | X | XX |
| | Day 29 | X | X | XX | X | XX | X | XX | X | xx | X | XX |
| | Day 43 | X | X | XX | X | XX | X | xx | X | xx | X | XX |
| | Day 50 | X | x | XX | x | XX | X | xx | X | XX | X | XX |
| | Max Severity Post<br>Baseline | X | X | XX | Х | xx | X | XX | х | xx | X | XX |
| Group 3: IIV4 Only | Baseline | X | X | XX | х | XX | X | xx | X | xx | X | XX |
| (N=X) | Day 8 | X | х | XX | х | XX | X | xx | X | XX | X | XX |
| | Day 22 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA |
| | Day 29 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA |
| | Day 43 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA |
| | Day 50 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA |

Table 129: Laboratory Results by Parameter, Maximum Severity, Study Day, and Treatment Group (Safety Population) – All Laboratory Parameters (continued)

| Max Severity Pos<br>Baseline | Х | xx | X | XX | х | XX | X | xx | X | XX |
|------------------------------|---|----|---|----|---|----|---|----|---|----|
|------------------------------|---|----|---|----|---|----|---|----|---|----|

Note: The "Max Post Baseline" rows indicate the maximum severity experienced by each subject at any time point post baseline, including unscheduled assessments.

N=Number of subjects in the Safety population.

Table 130: Laboratory Results by Parameter, Maximum Severity, Study Day, and Treatment Group (Safety Population) – White Blood Cells\*

| Treatment Group | Study Day | N | No | one | Gra | ild/<br>de 1<br>ow) | Gra | ild/<br>de 1<br>igh) | Gra | erate/<br>ide 2<br>ow) | Gra | erate/<br>de 2<br>igh) | Gra | rere/<br>ade 3<br>ow) | Gra | ere/<br>de 3<br>igh) | Mis | sing |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| Group 1: Simultaneous<br>Administration (N=X) | Baseline | Х | х | XX | х | XX | х | xx | х | xx | х | xx | х | xx | х | xx | х | XX |
| | Day 8 | Х | х | XX | X | XX | х | XX | х | XX | х | XX | X | XX | х | XX | х | XX |
| | Day 22 | х | х | XX | х | XX | х | XX | х | XX | х | XX | х | XX | х | XX | х | x xx<br>NA NA |
| | Day 29 | х | х | XX | Х | XX | х | XX | х | XX | х | XX | х | XX | х | XX | х | |
| | Day 43 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | |
| | Day 50 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | |
| | Max Severity<br>Post Baseline | Х | х | xx | х | xx | х | xx | х | xx | х | xx | х | xx | х | xx | х | XX |
| Group 2: Sequential | Baseline | x x xx x xx x xx x | х | XX | Х | XX | х | XX | х | XX | Х | XX | | | | | | |
| Administration (N=X) | Day 8 | х | X | XX | X | XX | X | XX | X | XX | х | XX | X | XX | X | XX | | |
| | Day 22 | X | X | XX | X | XX | X | XX | X | XX | х | XX | X | XX | X | XX | Х | XX |
| | Day 29 | х | х | XX | X | XX | X | XX | х | XX | х | XX | x | XX | х | XX | х | |
| | Day 43 | х | х | XX | х | XX | х | XX | х | XX | х | XX | х | XX | х | XX | х | |
| | Day 50 | х | х | XX | х | XX | х | XX | х | XX | х | XX | х | XX | х | XX | х | xx |
| | Max Severity<br>Post Baseline | Х | х | XX | х | XX | х | xx | х | xx | х | XX | х | xx | х | xx | х | XX |
| Group 3: IIV4 Only | Baseline | х | X | XX | X | XX | X | XX | х | XX | х | XX | X | XX | х | XX | х | XX |
| (N=X) | Day 8 | х | х | XX | X | XX | X | XX | х | XX | х | XX | х | XX | х | XX | x xx<br>NA NA | xx |
| | Day 22 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | | NA |
| | Day 29 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA |
| | Day 43 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA |

Table 130: Laboratory Results by Parameter, Maximum Severity, Study Day, and Treatment Group (Safety Population) – White Blood Cells (continued)

Note: The "Max Post Baseline" rows indicate the maximum severity experienced by each subject at any time point post baseline, including unscheduled assessments.

N=Number of subjects in the Safety population.

#### Tables with similar format:

- Table 131: Laboratory Results by Parameter, Maximum Severity, Study Day, and Treatment Group (Safety Population) Hemoglobin\*
- Table 132: Laboratory Results by Parameter, Maximum Severity, Study Day, and Treatment Group (Safety Population) Platelets\*
- Table 133: Laboratory Results by Parameter, Maximum Severity, Study Day, and Treatment Group (Safety Population) Alanine aminotransferase (ALT) \*
- Table 134: Laboratory Results by Parameter, Maximum Severity, Study Day, and Treatment Group (Safety Population) Total Bilirubin \*
- Table 135: Laboratory Results by Parameter, Maximum Severity, Study Day, and Treatment Group (Safety Population) Creatinine\*

Table 136: Laboratory Summary Statistics of Value and Change from Baseline by Study Day, and Treatment Group (Safety Population)
– White Blood Cells\*

| | | | | Value | | | Change from Baseline | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Treatment<br>Group | Study<br>Day | N | Mean | Standard<br>Deviation | Median | Min, Max | N | Mean | Standard<br>Deviation | Median | Min, Max |
| Group 1: | Baseline | X | xx.x | XX.X | xx | xx, xx | NA | NA | NA | NA | NA |
| Simultaneous<br>Administration<br>(N=X) | Day 8 | х | xx.x | XX.X | xx | xx, xx | х | XX.X | XX.X | XX | xx, xx |
| | Day 22 | х | xx.x | XX.X | xx | xx, xx | х | XX.X | XX.X | XX | xx, xx |
| | Day 29 | х | XX.X | XX.X | xx | xx, xx | х | XX.X | XX.X | XX | xx, xx |
| | Day 43 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA |
| | Day 50 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA |
| Group 2: | Baseline | X | xx.x | XX.X | xx | xx, xx | NA | NA | NA | NA | NA |
| Sequential<br>Administration | Day 8 | х | XX.X | XX.X | xx | xx, xx | х | XX.X | XX.X | XX | xx, xx |
| (N=X) | Day 22 | X | xx.x | XX.X | xx | xx, xx | X | XX.X | XX.X | XX | xx, xx |
| | Day 29 | X | xx.x | XX.X | xx | xx, xx | Х | XX.X | XX.X | XX | xx, xx |
| | Day 43 | X | xx.x | XX.X | xx | xx, xx | Х | XX.X | XX.X | XX | xx, xx |
| | Day 50 | X | xx.x | XX.X | xx | xx, xx | Х | XX.X | XX.X | XX | xx, xx |
| Group 3: IIV4 | Baseline | х | xx.x | XX.X | xx | xx, xx | NA | NA | NA | NA | NA |
| Only (N=X) | Day 8 | х | xx.x | XX.X | xx | xx, xx | Х | XX.X | XX.X | XX | xx, xx |
| | Day 22 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA |
| | Day 29 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA |
| | Day 43 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA |
| | Day 50 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA |

#### Tables with similar format:

- Table 137: Laboratory Summary Statistics of Value and Change from Baseline by Study Day, and Treatment Group (Safety Population)

   Hemoglobin\*
- Table 138: Laboratory Summary Statistics of Value and Change from Baseline by Study Day, and Treatment Group (Safety Population)

   Platelets\*
- Table 139: Laboratory Summary Statistics of Value and Change from Baseline by Study Day, and Treatment Group (Safety Population)

   Alanine Aminotransferase\* (ALT)
- Table 140: Laboratory Summary Statistics of Value and Change from Baseline by Study Day, and Treatment Group (Safety Population)

   Total Bilirubin\*
- Table 141: Laboratory Summary Statistics of Value and Change from Baseline by Study Day, and Treatment Group (Safety Population)

   Creatinine\*
## 14.3.4.5 Clinical Laboratory Reference Ranges

(Placeholder for the CSR)

## 14.3.5 Abnormal Laboratory Value Listings (by Subject)

**Table 142: Listing of Abnormal Laboratory Results - Chemistry** 

| Subject<br>ID | Treatment<br>Group | Sex | Age<br>(years) | Planned<br>Time<br>Point | Actual<br>Study<br>Day | Laboratory<br>Parameter<br>(Units) | Result<br>(Severity) | Relationship<br>to Treatment | If Not<br>Related,<br>Alternate<br>Etiology | Action<br>Taken with<br>Study<br>Treatment | Subject Discontinued Due to Result? |
|---|---|---|---|---|---|---|---|---|---|---|---|

**Table 143: Listing of Abnormal Laboratory Results - Hematology** 

| Subject<br>ID | Treatment<br>Group | Sex | Age<br>(years) | Planned<br>Time<br>Point | Actual<br>Study<br>Day | Laboratory<br>Parameter<br>(Units) | Result<br>(Severity) | Relationship<br>to Treatment | If Not<br>Related,<br>Alternate<br>Etiology | Action<br>Taken with<br>Study<br>Treatment | Subject Discontinued Due to Result? |
|---|---|---|---|---|---|---|---|---|---|---|---|

#### 14.3.6 Displays of Vital Signs

Table 144: Vital Signs by Assessment, Maximum Severity, Study Day, Treatment Group (Safety Population) - Any Assessment\*

| <b>Treatment Group</b> | Study Day | N | No | one | Mild | | Moderate | | Severe | | Missing | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | n | % | n | % | n | % | n | % | n | % |
| Group 1: Simultaneous | Baseline | x | х | XX | Х | xx | х | xx | Х | XX | х | XX |
| Administration (N=X) | Day 22 | | | | | | | | | | | |
| | Day 43 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA |
| | Max Severity Post Baseline | | | | | | | | | | | |
| Group 2: Sequential | Baseline | | | | | | | | | | | |
| Administration (N=X) | Day 22 | | | | | | | | | | | |
| | Day 43 | | | | | | | | | | | |
| | Max Severity Post Baseline | | | | | | | | | | | |
| Group 3: IIV4 Only | Baseline | | | | | | | | | | | |
| (N=X) | Day 22 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA |
| | Day 43 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA |
| | Max Severity Post Baseline | | | | | | | | | | | |

Note: The "Max Post Baseline" rows indicate the maximum severity experienced by each subject at any time point post baseline, including unscheduled assessments. N= Number of subjects in the Safety population.

#### Table with similar format:

Table 145: Vital Signs by Assessment, Maximum Severity, Study Day, Treatment Group (Safety Population) - Oral Temperature

Table 146: Vital Signs by Assessment, Maximum Severity, Study Day, and Treatment Group (Safety Population) – Systolic Blood Pressure

| Treatment<br>Group | Study Day | N | No | one | | ild<br>ow) | | ild<br>igh) | 1 | erate<br>ow) | | erate<br>gh) | | vere<br>ow) | | vere<br>igh) | Mis | sing |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| Group 1:<br>Simultaneous<br>Administration<br>(N=X) | Baseline | х | х | xx | х | xx | х | xx | х | xx | х | XX | х | xx | х | xx | х | XX |
| | Day 22 | x | х | xx | х | XX | х | xx | х | XX | х | XX | Х | xx | х | XX | х | XX |
| | Day 43 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA |
| | Max Severity<br>Post Baseline | Х | х | xx | х | xx | х | xx | х | xx | х | XX | X | xx | х | xx | х | XX |
| Group 2:<br>Sequential<br>Administration<br>(N=X) | Baseline | х | х | xx | х | xx | х | xx | х | xx | х | XX | х | xx | х | xx | х | XX |
| | Day 22 | х | х | xx | х | XX | х | xx | х | XX | Х | XX | х | XX | х | XX | х | xx |
| | Day 43 | х | х | xx | х | XX | х | xx | х | XX | х | XX | х | xx | х | XX | х | xx |
| | Max Severity<br>Post Baseline | Х | х | xx | х | xx | х | xx | х | xx | х | XX | X | xx | х | xx | х | XX |
| Group 3: IIV4<br>Only (N=X) | Baseline | X | х | xx | х | XX | х | xx | х | xx | х | XX | X | xx | х | XX | х | XX |
| | Day 22 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA |
| | Day 43 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA |
| | Max Severity<br>Post Baseline | х | х | XX | Х | XX | Х | XX | Х | XX | х | XX | X | XX | х | XX | Х | XX |

Note: The "Max Post Baseline" rows indicate the maximum severity experienced by each subject at any time point post baseline, including unscheduled assessments. N=Number of subjects in the Safety population.

#### Tables with similar format:

- Table 147: Vital Signs by Assessment, Maximum Severity, Study Day, and Treatment Group (Safety Population) Diastolic Blood Pressure
- Table 148: Vital Signs by Assessment, Maximum Severity, Study Day, and Treatment Group (Safety Population) Pulse

## 14.4 Summary of Concomitant Medications

Table 149: Number and Percentage of Subjects with Prior and Concurrent Medications by WHO Drug Classification and Treatment Group – Safety Population

| WHO Drug Code<br>Level 1, Anatomic Group | WHO Drug Code<br>Level 2, Therapeutic<br>Subgroup | Simult<br>Admini | up 1:<br>aneous<br>stration<br>=X) | Sequ<br>Admini | up 2:<br>ential<br>stration<br>=X) | Group 3:<br>IIV4 Only (N=X) | |
|---|---|---|---|---|---|---|---|
| | | n | % | n | % | n | % |
| Any Level 1 Codes | Any Level 2 Codes | x | xx | x | xx | X | XX |
| [ATC Level 1 - 1] | Any [ATC 1 – 1] | | | | | | |
| | [ATC 2 - 1] | | | | | | |
| | [ATC 2 - 2] | | | | | | |
| | [ATC 2 - 3] | | | | | | |
| [ATC Level 1 – 2] | [ATC 2 - 1] | | | | | | |
| | [ATC 2 - 2] | | | | | | |
| | [ATC 2 - 3] | | | | | | |

N= Number of subjects in the Safety population. n=Number of subjects reporting taking at least one medication in the specific WHO Drug Class.

## **Appendix 2. FIGURE MOCK-UPS**

## **LIST OF FIGURES**

| Figure 1: | CONSORT Flow Diagram*149 |
|---|---|
| Figure 2: | Reverse Cumulative Distribution of Hemagglutination Inhibition Antibody against 2017 A/H7N9 by Study Day and Treatment Group, Modified Intent to Treat Population* |
| Figure 3: | Reverse Cumulative Distribution of Hemagglutination Inhibition Antibody against 2017 A/H7N9 by Study Day and Treatment Group, Per Protocol Population* 150 |
| Figure 4: | Reverse Cumulative Distribution of Neutralizing Antibody Against 2017 A/H7N9 by Study Day and Treatment Group, Modified Intent to Treat Population* |
| Figure 5: | Reverse Cumulative Distribution of Neutralizing Antibody against 2017 A/H7N9 by Study Day and Treatment Group, Per Protocol Population* |
| Figure 6: | Reverse Cumulative Distribution of Hemagglutination Inhibition Antibody against A/Michigan/45/2015 X-275(H1N1) by Study Day and Treatment Group, Modified Intent to Treat Population* |
| Figure 7: | Reverse Cumulative Distribution of Hemagglutination Inhibition Antibody against A/Michigan/45/2015 X-275(H1N1) by Study Day and Treatment Group, Per Protocol Population* |
| Figure 8: | Reverse Cumulative Distribution of Neutralizing Antibody Against A/Michigan/45/2015 X-275(H1N1) by Study Day and Treatment Group, Modified Intent to Treat Population* |
| Figure 9: | Reverse Cumulative Distribution of Neutralizing Antibody against A/Michigan/45/2015 X-275(H1N1) by Study Day and Treatment Group, Per Protocol Population* |
| Figure 10: | Reverse Cumulative Distribution of Hemagglutination Inhibition Antibody against A/Hong Kong/4801/2014 X263B (H3N2) by Study Day and Treatment Group, Modified Intent to Treat Population* |
| Figure 11: | Reverse Cumulative Distribution of Hemagglutination Inhibition Antibody against A/Hong Kong/4801/2014 X263B (H3N2) by Study Day and Treatment Group, Per Protocol Population* |
| Figure 12: | Reverse Cumulative Distribution of Neutralizing Antibody Against A/ Hong Kong/4801/2014 X263B (H3N2) by Study Day and Treatment Group, Modified Intent to Treat Population* |
| Figure 13: | Reverse Cumulative Distribution of Neutralizing Antibody against A/ Hong Kong/4801/2014 X263B (H3N2) by Study Day and Treatment Group, Per Protocol Population* |
| Figure 14: | Reverse Cumulative Distribution of Hemagglutination Inhibition Antibody against B/Phuket/3073/2013 (B Yamagata lineage) by Study Day and Treatment Group, Modified Intent to Treat Population* |
| Figure 15: | Reverse Cumulative Distribution of Hemagglutination Inhibition Antibody against B/Phuket/3073/2013 (B Yamagata lineage) by Study Day and Treatment Group, Per Protocol Population* |
| Figure 16: | Reverse Cumulative Distribution of Neutralizing Antibody Against B/Phuket/3073/2013 (B Yamagata lineage)by Study Day and Treatment Group, Modified Intent to Treat Population* |

| Figure 17: | Reverse Cumulative Distribution of Neutralizing Antibody against |
|---|---|
| | B/Phuket/3073/2013 (B Yamagata lineage) by Study Day and Treatment Group, Per |
| | Protocol Population* |
| Figure 18: | Reverse Cumulative Distribution of Hemagglutination Inhibition Antibody |
| | against B/Brisbane/60/2008 (B Victoria lineage) by Study Day and Treatment Group, |
| | Modified Intent to Treat Population* |
| Figure 19: | Reverse Cumulative Distribution of Hemagglutination Inhibition Antibody against |
| | B/Brisbane/60/2008 (B Victoria lineage) by Study Day and Treatment Group, Per |
| | Protocol Population* |
| Figure 20: | Reverse Cumulative Distribution of Neutralizing Antibody Against |
| | B/Brisbane/60/2008 (B Victoria lineage) by Study Day and Treatment Group, |
| | Modified Intent to Treat Population* |
| Figure 21: | Reverse Cumulative Distribution of Neutralizing Antibody against B/Brisbane/60/2008 |
| | (B Victoria lineage) by Study Day and Treatment Group, Per Protocol Population*. 151 |
| Figure 22: | Geometric Mean Titers of Hemagglutination Inhibition Antibody Against 2017 |
| | A/H7N9 by Study Day and Treatment Group, Modified Intent to Treat Population* 152 |
| Figure 23: | Geometric Mean Titers of Hemagglutination Inhibition Antibody against 2017 |
| | A/H7N9 by Study Day and Treatment Group, Per Protocol Population* |
| Figure 24: | Geometric Mean Titers of Neutralizing Antibody against 2017 A/H7N9 by Study Day |
| | and Treatment Group, Modified Intent to Treat Population* |
| Figure 25: | Geometric Mean Titers of Neutralizing Antibody against 2017 A/H7N9 by Study Day |
| F: 06 | and Treatment Group, Per Protocol Population* |
| Figure 26: | Geometric Mean Titers of Hemagglutination Inhibition Antibody Against |
| | A/Michigan/45/2015 X-275(H1N1) by Study Day and Treatment Group, Modified |
| E: 07 | Intent to Treat Population* |
| Figure 27: | Geometric Mean Titers of Hemagglutination Inhibition Antibody against |
| | A/Michigan/45/2015 X-275(H1N1) by Study Day and Treatment Group, Per Protocol |
| Ei 20. | Population* |
| Figure 28: | Geometric Mean Titers of Neutralizing Antibody against A/Michigan/45/2015 X-275(H1N1) by Study Day and Treatment Group, Modified Intent to Treat Repulation* |
| | 275(H1N1) by Study Day and Treatment Group, Modified Intent to Treat Population* 152 |
| Figure 29: | Geometric Mean Titers of Neutralizing Antibody against A/Michigan/45/2015 X- |
| rigure 29. | 275(H1N1) by Study Day and Treatment Group, Per Protocol Population* |
| Figure 30: | Geometric Mean Titers of Hemagglutination Inhibition Antibody Against A/Hong |
| rigure 50. | Kong/4801/2014 X263B (H3N2) by Study Day and Treatment Group, Modified Intent |
| | to Treat Population* |
| Figure 31: | Geometric Mean Titers of Hemagglutination Inhibition Antibody against A/Hong |
| 116410 51. | Kong/4801/2014 X263B (H3N2) by Study Day and Treatment Group, Per Protocol |
| | Population* |
| Figure 32: | Geometric Mean Titers of Neutralizing Antibody against A/Hong Kong/4801/2014 |
| 8 | X263B (H3N2) by Study Day and Treatment Group, Modified Intent to Treat |
| | Population* |
| Figure 33: | Geometric Mean Titers of Neutralizing Antibody against A/Hong Kong/4801/2014 |
| 8 | X263B (H3N2) by Study Day and Treatment Group, Per Protocol Population* 153 |
| Figure 34: | Geometric Mean Titers of Hemagglutination Inhibition Antibody Against |
| C | B/Phuket/3073/2013 (B Yamagata lineage) by Study Day and Treatment Group, |
| | Modified Intent to Treat Population* |
| Figure 35: | Geometric Mean Titers of Hemagglutination Inhibition Antibody against |
| - | B/Phuket/3073/2013 (B Yamagata lineage) by Study Day and Treatment Group, Per |
| | Protocol Population* 153 |

| Figure 36: | Geometric Mean Titers of Neutralizing Antibody against B/Phuket/3073/2013 (B |
|---|---|
| | Yamagata lineage) by Study Day and Treatment Group, Modified Intent to Treat |
| Figure 37: | Population* |
| riguic 37. | Yamagata lineage) by Study Day and Treatment Group, Per Protocol Population* 153 |
| Figure 38: | Geometric Mean Titers of Hemagglutination Inhibition Antibody Against |
| 8 | B/Brisbane/60/2008 (B Victoria lineage) by Study Day and Treatment Group, |
| | Modified Intent to Treat Population* |
| Figure 39: | Geometric Mean Titers of Hemagglutination Inhibition Antibody against |
| | B/Brisbane/60/2008 (B Victoria lineage) by Study Day and Treatment Group, Per |
| | Protocol Population* |
| Figure 40: | Geometric Mean Titers of Neutralizing Antibody against B/Brisbane/60/2008 (B |
| | Victoria lineage) by Study Day and Treatment Group, Modified Intent to Treat |
| Figure 41: | Population* |
| rigule 41. | Victoria lineage) by Study Day and Treatment Group, Per Protocol Population* 153 |
| Figure 42: | Correlation of Hemagglutination Inhibition Antibody and Neutralizing Antibody |
| 118010 12. | Against 2017 A/H7N9 by Study Day and Treatment Group, Modified Intent-to-Treat |
| | Population* |
| Figure 43: | Correlation of Hemagglutination Inhibition Antibody and Neutralizing Antibody |
| | Against 2017 A/H7N9 by Study Day and Treatment Group, Per Protocol Population* |
| Figure 44: | Correlation of Hemagglutination Inhibition Antibody and Neutralizing Antibody |
| | Against A/Michigan/45/2015 X-275(H1N1) by Study Day and Treatment Group, |
| Figure 45: | Modified Intent-to-Treat Population* |
| rigule 45. | Against A/Michigan/45/2015 X-275(H1N1) by Study Day and Treatment Group, Per |
| | Protocol Population* |
| Figure 46: | Correlation of Hemagglutination Inhibition Antibody and Neutralizing Antibody |
| C | Against A/Hong Kong/4801/2014 X263B (H3N2) by Study Day and Treatment Group, |
| | Modified Intent-to-Treat Population* |
| Figure 47: | Correlation of Hemagglutination Inhibition Antibody and Neutralizing Antibody |
| | Against A/Hong Kong/4801/2014 X263B (H3N2) by Study Day and Treatment Group, |
| E: 40 | Per Protocol Population* |
| Figure 48: | Correlation of Hemagglutination Inhibition Antibody and Neutralizing Antibody<br>Against B/Phuket/3073/2013 (B Yamagata lineage) by Study Day and Treatment |
| | Group, Modified Intent-to-Treat Population*155 |
| Figure 49: | Correlation of Hemagglutination Inhibition Antibody and Neutralizing Antibody |
| 118010 .51 | Against B/Phuket/3073/2013 (B Yamagata lineage) by Study Day and Treatment |
| | Group, Per Protocol Population* |
| Figure 50: | Correlation of Hemagglutination Inhibition Antibody and Neutralizing Antibody |
| | Against B/Brisbane/60/2008 (B Victoria lineage) by Study Day and Treatment Group, |
| T | Modified Intent-to-Treat Population* |
| Figure 51: | Correlation of Hemagglutination Inhibition Antibody and Neutralizing Antibody |
| | Against B/Brisbane/60/2008 (B Victoria lineage) by Study Day and Treatment Group, |
| Figure 52: | Per Protocol Population* |
| Figure 53: | Maximum Severity of Solicited Local Symptoms per Subject by Day Post Dose 156 |
| Figure 54: | Frequency of Unsolicited Adverse Events by MedDRA® System Organ Class and |
| <i>U</i> - | Severity |

| Figure 55: | Incidence of Unsolicited Adverse Events by MedDRA® System Organ Class and Severity |
|---|---|
| Figure 56: | Frequency of Adverse Events by MedDRA® System Organ Class and Relationship to Treatment |
| Figure 57: | Incidence of Adverse Events by MedDRA® System Organ Class and Relationship to Treatment |
| Figure 58: | Laboratory Results by Scheduled Visits: Mean Changes from Baseline by Laboratory Parameter and Treatment Group – White Blood Cells |
| Figure 59: | Laboratory Summary Statistics of Change from Baseline by Parameter, Maximum Severity, Study Day, and Treatment Group – Hemoglobin |
| Figure 60: | Laboratory Summary Statistics of Change from Baseline Results by Parameter, Maximum Severity, Study Day, and Treatment Group – Platelets |
| Figure 61: | Laboratory Summary Statistics of Change from Baseline by Parameter, Maximum Severity, Study Day, and Treatment Group – Alanine Aminotransferase (ALT) 161 |
| Figure 62: | Laboratory Summary Statistics of Change from Baseline Results by Parameter, Maximum Severity, Study Day, and Treatment Group – Total Bilirubin |
| Figure 63: | Laboratory Summary Statistics of Change from Baseline Results by Parameter, Maximum Severity, Study Day, and Treatment Group – Creatinine |

#### 10.1 Disposition of Subjects Figures

Figure 1: CONSORT Flow Diagram\*



#### 14.2.2 Immunogenicity Figures

Reverse Cumulative Distribution of Hemagglutination Inhibition Antibody Figure 2: against 2017 A/H7N9 by Study Day and Treatment Group, Modified Intent to Treat Population\*

[Implementation Note: A generic sample figure is shown below. The RCD curves should be presented in a single figure with separate panels for each outcome day (21, 42, 63, and 180 days post dose 1 and 180 days post final dose). Figures generated for the preliminary report will include data from all visits through study Day 64. Visit labels should be included in the panel headers. Within each panel individual curves should be used for each Treatment Group (three curves). Each treatment group should have a separate color and marker shape.]





Reverse Cumulative Distribution Curves Hemagglutination Titer

Figures with similar format:

- Figure 3: Reverse Cumulative Distribution of Hemagglutination Inhibition Antibody against 2017 A/H7N9 by Study Day and Treatment Group, Per Protocol Population\*
- Reverse Cumulative Distribution of Neutralizing Antibody Against 2017 A/H7N9 by Figure 4: Study Day and Treatment Group, Modified Intent to Treat Population\*
- Reverse Cumulative Distribution of Neutralizing Antibody against 2017 A/H7N9 by Figure 5: Study Day and Treatment Group, Per Protocol Population\*
- Figure 6: Reverse Cumulative Distribution of Hemagglutination Inhibition Antibody against A/Michigan/45/2015 X-275(H1N1) by Study Day and Treatment Group, **Modified Intent to Treat Population\***
- Figure 7: Reverse Cumulative Distribution of Hemagglutination Inhibition Antibody against A/Michigan/45/2015 X-275(H1N1) by Study Day and Treatment Group, Per **Protocol Population\***

- Figure 8: Reverse Cumulative Distribution of Neutralizing Antibody Against A/Michigan/45/2015 X-275(H1N1) by Study Day and Treatment Group, Modified Intent to Treat Population\*
- Figure 9: Reverse Cumulative Distribution of Neutralizing Antibody against A/Michigan/45/2015 X-275(H1N1) by Study Day and Treatment Group, Per Protocol Population\*
- Figure 10: Reverse Cumulative Distribution of Hemagglutination Inhibition Antibody against A/Hong Kong/4801/2014 X263B (H3N2) by Study Day and Treatment Group, Modified Intent to Treat Population\*
- Figure 11: Reverse Cumulative Distribution of Hemagglutination Inhibition Antibody against A/Hong Kong/4801/2014 X263B (H3N2) by Study Day and Treatment Group, Per Protocol Population\*
- Figure 12: Reverse Cumulative Distribution of Neutralizing Antibody Against A/ Hong Kong/4801/2014 X263B (H3N2) by Study Day and Treatment Group, Modified Intent to Treat Population\*
- Figure 13: Reverse Cumulative Distribution of Neutralizing Antibody against A/ Hong Kong/4801/2014 X263B (H3N2) by Study Day and Treatment Group, Per Protocol Population\*
- Figure 14: Reverse Cumulative Distribution of Hemagglutination Inhibition Antibody against B/Phuket/3073/2013 (B Yamagata lineage) by Study Day and Treatment Group, Modified Intent to Treat Population\*
- Figure 15: Reverse Cumulative Distribution of Hemagglutination Inhibition Antibody against B/Phuket/3073/2013 (B Yamagata lineage) by Study Day and Treatment Group, Per Protocol Population\*
- Figure 16: Reverse Cumulative Distribution of Neutralizing Antibody Against B/Phuket/3073/2013 (B Yamagata lineage)by Study Day and Treatment Group, Modified Intent to Treat Population\*
- Figure 17: Reverse Cumulative Distribution of Neutralizing Antibody against B/Phuket/3073/2013 (B Yamagata lineage) by Study Day and Treatment Group, Per Protocol Population\*
- Figure 18: Reverse Cumulative Distribution of Hemagglutination Inhibition Antibody against B/Brisbane/60/2008 (B Victoria lineage) by Study Day and Treatment Group, Modified Intent to Treat Population\*
- Figure 19: Reverse Cumulative Distribution of Hemagglutination Inhibition Antibody against B/Brisbane/60/2008 (B Victoria lineage) by Study Day and Treatment Group, Per Protocol Population\*
- Figure 20: Reverse Cumulative Distribution of Neutralizing Antibody Against B/Brisbane/60/2008 (B Victoria lineage) by Study Day and Treatment Group, Modified Intent to Treat Population\*
- Figure 21: Reverse Cumulative Distribution of Neutralizing Antibody against B/Brisbane/60/2008 (B Victoria lineage) by Study Day and Treatment Group, Per Protocol Population\*

Figure 22: Geometric Mean Titers of Hemagglutination Inhibition Antibody Against 2017
A/H7N9 by Study Day and Treatment Group, Modified Intent to Treat Population\*

[Implementation Note: A generic sample figure is shown below. Planned Study Day is plotted along the x-axis, with visit labels as tick labels. Titer is plotted on the y-axis on the log-10 scale. GMT should be plotted at each visit with upper and lower error bars for the 95% CI for each treatment group with different marker shapes/colors for each treatment group. Each treatment group should have a separate color and marker shape]

Note: this figure will be generated for the preliminary report including data through Day 43, then regenerated for the final CSR to include all data through Day 202.



Figures with similar format:

- Figure 23: Geometric Mean Titers of Hemagglutination Inhibition Antibody against 2017 A/H7N9 by Study Day and Treatment Group, Per Protocol Population\*
- Figure 24: Geometric Mean Titers of Neutralizing Antibody against 2017 A/H7N9 by Study Day and Treatment Group, Modified Intent to Treat Population\*
- Figure 25: Geometric Mean Titers of Neutralizing Antibody against 2017 A/H7N9 by Study Day and Treatment Group, Per Protocol Population\*
- Figure 26: Geometric Mean Titers of Hemagglutination Inhibition Antibody Against A/Michigan/45/2015 X-275(H1N1) by Study Day and Treatment Group, Modified Intent to Treat Population\*
- Figure 27: Geometric Mean Titers of Hemagglutination Inhibition Antibody against A/Michigan/45/2015 X-275(H1N1) by Study Day and Treatment Group, Per Protocol Population\*
- Figure 28: Geometric Mean Titers of Neutralizing Antibody against A/Michigan/45/2015 X-275(H1N1) by Study Day and Treatment Group, Modified Intent to Treat Population\*
- Figure 29: Geometric Mean Titers of Neutralizing Antibody against A/Michigan/45/2015 X-275(H1N1) by Study Day and Treatment Group, Per Protocol Population\*
- Figure 30: Geometric Mean Titers of Hemagglutination Inhibition Antibody Against A/Hong Kong/4801/2014 X263B (H3N2) by Study Day and Treatment Group, Modified Intent to Treat Population\*
- Figure 31: Geometric Mean Titers of Hemagglutination Inhibition Antibody against A/Hong Kong/4801/2014 X263B (H3N2) by Study Day and Treatment Group, Per Protocol Population\*

- Figure 32: Geometric Mean Titers of Neutralizing Antibody against A/Hong Kong/4801/2014 X263B (H3N2) by Study Day and Treatment Group, Modified Intent to Treat Population\*
- Figure 33: Geometric Mean Titers of Neutralizing Antibody against A/Hong Kong/4801/2014 X263B (H3N2) by Study Day and Treatment Group, Per Protocol Population\*
- Figure 34: Geometric Mean Titers of Hemagglutination Inhibition Antibody Against B/Phuket/3073/2013 (B Yamagata lineage) by Study Day and Treatment Group, Modified Intent to Treat Population\*
- Figure 35: Geometric Mean Titers of Hemagglutination Inhibition Antibody against B/Phuket/3073/2013 (B Yamagata lineage) by Study Day and Treatment Group, Per Protocol Population\*
- Figure 36: Geometric Mean Titers of Neutralizing Antibody against B/Phuket/3073/2013 (B Yamagata lineage) by Study Day and Treatment Group, Modified Intent to Treat Population\*
- Figure 37: Geometric Mean Titers of Neutralizing Antibody against B/Phuket/3073/2013 (B Yamagata lineage) by Study Day and Treatment Group, Per Protocol Population\*
- Figure 38: Geometric Mean Titers of Hemagglutination Inhibition Antibody Against B/Brisbane/60/2008 (B Victoria lineage) by Study Day and Treatment Group, Modified Intent to Treat Population\*
- Figure 39: Geometric Mean Titers of Hemagglutination Inhibition Antibody against B/Brisbane/60/2008 (B Victoria lineage) by Study Day and Treatment Group, Per Protocol Population\*
- Figure 40: Geometric Mean Titers of Neutralizing Antibody against B/Brisbane/60/2008 (B Victoria lineage) by Study Day and Treatment Group, Modified Intent to Treat Population\*
- Figure 41: Geometric Mean Titers of Neutralizing Antibody against B/Brisbane/60/2008 (B Victoria lineage) by Study Day and Treatment Group, Per Protocol Population\*

Figure 42: Correlation of Hemagglutination Inhibition Antibody and Neutralizing Antibody Against 2017 A/H7N9 by Study Day and Treatment Group, Modified Intent-to-Treat Population\*

[Implementation Note: A generic sample figure is shown below. The scatter plots should be presented in a single figure with separate panels for each visit (baseline and 21, 42, 63, and 180 days post dose 1 and 180 days post final dose). Visit labels should be included in the panel header. Within each panel distinct marker types and colors should be used to indicate the treatment groups, with treatment group labels included in a legend. Each treatment group should have a unique color and marker shape. The spearman correlation should be calculated over all subjects and annotated within each panel as "Spearman Correlation (r=0.xx, p=0.xx)"]



Figure with Similar format:

Figure 43: Correlation of Hemagglutination Inhibition Antibody and Neutralizing Antibody Against 2017 A/H7N9 by Study Day and Treatment Group, Per Protocol Population\*

Figure 44: Correlation of Hemagglutination Inhibition Antibody and Neutralizing Antibody Against A/Michigan/45/2015 X-275(H1N1) by Study Day and Treatment Group, Modified Intent-to-Treat Population\*

- Figure 45: Correlation of Hemagglutination Inhibition Antibody and Neutralizing Antibody Against A/Michigan/45/2015 X-275(H1N1) by Study Day and Treatment Group, Per Protocol Population\*
- Figure 46: Correlation of Hemagglutination Inhibition Antibody and Neutralizing Antibody Against A/Hong Kong/4801/2014 X263B (H3N2) by Study Day and Treatment Group, Modified Intent-to-Treat Population\*
- Figure 47: Correlation of Hemagglutination Inhibition Antibody and Neutralizing Antibody Against A/Hong Kong/4801/2014 X263B (H3N2) by Study Day and Treatment Group, Per Protocol Population\*
- Figure 48: Correlation of Hemagglutination Inhibition Antibody and Neutralizing Antibody Against B/Phuket/3073/2013 (B Yamagata lineage) by Study Day and Treatment Group, Modified Intent-to-Treat Population\*
- Figure 49: Correlation of Hemagglutination Inhibition Antibody and Neutralizing Antibody Against B/Phuket/3073/2013 (B Yamagata lineage) by Study Day and Treatment Group, Per Protocol Population\*
- Figure 50: Correlation of Hemagglutination Inhibition Antibody and Neutralizing Antibody Against B/Brisbane/60/2008 (B Victoria lineage) by Study Day and Treatment Group, Modified Intent-to-Treat Population\*
- Figure 51: Correlation of Hemagglutination Inhibition Antibody and Neutralizing Antibody Against B/Brisbane/60/2008 (B Victoria lineage) by Study Day and Treatment Group, Per Protocol Population\*

#### 14.3.1 Safety Figures

#### 14.3.1.1 Solicited Adverse Events

#### Figure 52: Maximum Severity of Solicited Systemic Symptoms per Subject by Day Post Dose

[Implementation Note: A Generic figure is shown below. A <u>vertical</u> bar chart should be presented in 1 image file with separate panels for each treatment group and dose (3 rows (treatment groups) x 3 columns (dose #)). Axes should be labeled as follows: x-axis label: Study Day, y-axis label: Percentage of Subjects (%). The treatment groups should be indicated in the panel headers including "(N=X)", where N = the number of subjects in the in the Safety Population who received the relevant dose. Subjects are counted at most once at the maximum severity across all systemic events reported for the specified time point]



Figure with similar format:

Figure 53: Maximum Severity of Solicited Local Symptoms per Subject by Day Post Dose

#### 14.3.1.2 Unsolicited Adverse Events

# Figure 54: Frequency of Unsolicited Adverse Events by MedDRA® System Organ Class and Severity

[Implementation Note: A Generic figure is shown below. This figure includes all unsolicited events across all doses. A *horizontal* bar chart should be presented in 1 image file separate panels for each treatment group (3 columns (treatment groups)). Axes should be labeled as follows: y-axis label: System Organ Class, y-axis label: Number of Events. The treatment groups should be indicated in the panel headers including "(N=X)", where N = the number of subjects in the in the Safety Population. The y-axis should present all SOCs reported by at least 1 subject and an "All Events" category. Y-axis should be sorted with "All Events first, then in decreasing order of total incidence]



Figure 55: Incidence of Unsolicited Adverse Events by MedDRA® System Organ Class and Severity

[Implementation Note: A Generic figure is shown below. This figure includes all unsolicited events across all doses. A *horizontal* bar chart should be presented in 1 image file with separate panels for each treatment group (3 columns). Axes should be labeled as follows: y-axis label: System Organ Class, x-axis label: Percentage of Subjects (%). The treatment groups should be indicated in the panel headers including "(N=X)", where N = the number of subjects in the in the Safety Population. Subjects are counted at most once at the maximum severity across for any events in the applicable SOC. The y-axis should present all SOCs reported by at least 1 subject and an "All Events" category. Y-axis should be sorted with "All Events" first then in decreasing order of total incidence]



Figure 56: Frequency of Adverse Events by MedDRA® System Organ Class and Relationship to Treatment

[Implementation Note: A generic sample figure is shown below. This figure includes all unsolicited events across all doses. A *horizontal* bar chart should be presented in 1 image file with separate panels for each treatment group and study dose (3 columns (treatment groups). Axes should be labeled as follows: y-axis label: System Organ Class, y-axis label: Number of Events. The treatment groups should be indicated in the panel headers including "(N=X)", where N = the number of subjects in the in the Safety Population. The y-axis should present all SOCs reported by at least 1 subject and an "All Events" category. Y-axis should be sorted with "All Events first then in decreasing order of total frequency]



Figure 57: Incidence of Adverse Events by MedDRA® System Organ Class and Relationship to Treatment

[Implementation Note: A Generic figure is shown below. This figure includes all unsolicited events across all doses. A *horizontal* bar chart should be presented in a 1 image file with separate panels for each treatment group (3 columns (treatment groups)). Axes should be labeled as follows: y-axis label: System Organ Class, x-axis label: Percentage of Subjects (%). The treatment groups should be indicated in the panel headers including "(N=X)", where N = the number of subjects in the in the Safety Population. Subjects are counted at most once at the maximum relationship (related >not-related) across for any events in the applicable SOC. The y-axis should present all SOCs reported by at least 1 subject and an "All Events" category. Y-axis should be sorted with "All Events first, then in decreasing order of total incidence across groups]



#### 14.3.5 Displays of Laboratory Results

Figure 58: Laboratory Results by Scheduled Visits: Mean Changes from Baseline by Laboratory Parameter and Treatment Group – White Blood Cells

[Implementation note: A generic figure is shown below. Plot should be generated with all treatment groups in a single image file with panels for each treatment group (3 columns (treatment groups)) with a box plot shown for each post-baseline study day that labs are drawn (D8, D22, D29, D43, D50). Yaxis should be labeled "[Parameter] Change from baseline ([units]). Repeat for all clinical laboratory parameters: WBC, Hgb, PLT, ALT, T. Bili, Cr]



Figures with similar format:

- Figure 59: Laboratory Summary Statistics of Change from Baseline by Parameter, Maximum Severity, Study Day, and Treatment Group Hemoglobin
- Figure 60: Laboratory Summary Statistics of Change from Baseline Results by Parameter, Maximum Severity, Study Day, and Treatment Group Platelets
- Figure 61: Laboratory Summary Statistics of Change from Baseline by Parameter, Maximum Severity, Study Day, and Treatment Group Alanine Aminotransferase (ALT)

- Figure 62: Laboratory Summary Statistics of Change from Baseline Results by Parameter, Maximum Severity, Study Day, and Treatment Group Total Bilirubin
- Figure 63: Laboratory Summary Statistics of Change from Baseline Results by Parameter, Maximum Severity, Study Day, and Treatment Group Creatinine

## Appendix 3. LISTINGS MOCK-UPS

## **LIST OF LISTINGS**

| Listing 1: | 16.1.6 - Listing of Subjects Receiving Investigational Product | 164 |
|---|---|---|
| Listing 2: | 16.2.1 - Early Terminations or Discontinued Subjects | |
| Listing 3: | 16.2.2.1 - Subject-Specific Protocol Deviations | |
| Listing 4: | 16.2.2.2 - Non-Subject-Specific Protocol Deviations | 167 |
| Listing 5: | 16.2.3 - Subjects Excluded from Analysis Populations | |
| Listing 6: | 16.2.4.1 - Demographics Data | |
| Listing 7: | 16.2.4.2 – Pre-Existing and Concurrent Medical Conditions | |
| Listing 8: | 16.2.4.3 – Influenza Vaccination History | 171 |
| Listing 9: | 16.2.6 - Individual Immunogenicity Response Data | |
| Listing 10: | 16.2.7.1 - Solicited Events – Systemic Symptoms | 174 |
| Listing 11: | 16.2.7.2 - Solicited Events – Local Symptoms | 175 |
| Listing 12: | 16.2.7.3 - Unsolicited Adverse Events | |
| Listing 13: | 16.2.8.1 - Clinical Laboratory Results – Hematology | 177 |
| Listing 14: | 16.2.8.2 - Clinical Laboratory Results – Chemistry | |
| Listing 15: | 16.2.9.1 - Vital Signs | 179 |
| Listing 16: | 16.2.9.2 - Physical Exam Findings | |
| Listing 17: | 16.2.10 - Concomitant Medications | |
| Listing 18: | 16.2.11.1 - Pregnancy Reports – Maternal Information | 182 |
| Listing 19: | 16.2.11.2 - Pregnancy Reports – Gravida and Para | |
| Listing 20: | 16.2.11.3 - Pregnancy Reports – Live Birth Outcomes | 183 |
| Listing 21: | 16.2.11.4 - Pregnancy Reports – Still Birth Outcomes | |
| Listing 22: | 16.2.11.5 - Pregnancy Reports – Spontaneous, Elective, or Therapeutic Abortion | |
| - | Outcomes | 183 |

## 16.1.6 Listing of Subjects Receiving Investigational Product

**Listing 1: 16.1.6 - Listing of Subjects Receiving Investigational Product** 

| Subject ID | Randomized<br>Treatment Group | Product Received Study<br>Dose 1 | Product Received Study<br>Dose 2 | Product Received Study<br>Dose 3 |
|---|---|---|---|---|
| XXXXXXXXX | Group 1 | IIV4 / A/H7N9 | A/H7N9 | N/A |
| XXXXXXXXX | Group 2 | IIV4 | A/H7N9 | A/H7N9 |
| XXXXXXXXX | Group 3 | IIV4 | N/A | N/A |

- 16.2 Database Listings by Subject
- 16.2.1 Discontinued Subjects

#### **Listing 2: 16.2.1 - Early Terminations or Discontinued Subjects**

[Implementation Note: Category will be either "Early Termination" or "Treatment Discontinuation." In the "Reason" column, concatenate any "specify" fields, including AE number and DV number.]

| Subject ID | Treatment Group | Category | Reason for Early Termination or Treatment Discontinuation | Study Day |
|---|---|---|---|---|

#### 16.2.2 Protocol Deviations

#### **Listing 3: 16.2.2.1 - Subject-Specific Protocol Deviations**

[Implementation Note: In the "Deviation" column, concatenate any and all "specify" fields (including visit number, etc.). If "Reason for Deviation" is "Other," concatenate "specify" field, separate by a colon, e.g., "Other: Subject refusal."]

| Subject<br>ID | Treatment<br>Group | DV<br>Number | Deviation | Deviation<br>Category | Study<br>Day | Reason for<br>Deviation | Deviation<br>Resulted<br>in AE? | Deviation<br>Resulted in<br>Subject<br>Termination? | Deviation<br>Affected<br>Product<br>Stability? | Deviation<br>Resolution | Comments |
|---|---|---|---|---|---|---|---|---|---|---|---|

#### **Listing 4: 16.2.2.2 - Non-Subject-Specific Protocol Deviations**

[Implementation Note: In the "Deviation" column, concatenate any and all "specify" fields (including visit number, etc.). If "Reason for Deviation" is "Other," concatenate "specify" field, separate by a colon, e.g., "Other: Subject refusal."]

| Site | Deviation | Start<br>Date | End Date | Reason for<br>Deviation | Deviation<br>Resulted in<br>Subject<br>Termination<br>? | Deviation<br>Affected<br>Product<br>Stability? | Deviation<br>Category | Deviation<br>Resolution | Comments |
|---|---|---|---|---|---|---|---|---|---|

.

#### 16.2.3 Subjects Excluded from the Analysis

#### Listing 5: 16.2.3 - Subjects Excluded from Analysis Populations

[Implementation Note: This data in this listing should be congruent with the "Analysis Populations by Treatment Group" table. The reasons included here should match the SAP text that describes who will be excluded from analyses.]

| Treatment Group | Subject ID | Analyses in which<br>Subject is Included | Analyses from which<br>Subject is Excluded | Results Available? | Reason Subject Excluded |
|---|---|---|---|---|---|
| | | [e.g., Safety, ITT, PP] | [e.g., Safety, ITT, PP, Day x] | | |

Note: "Yes" in the "Results available" column indicates that available data were removed from the analysis. "No" indicates that no data were available for inclusion in the analysis.

## 16.2.4 Demographic Data

## **Listing 6: 16.2.4.1 - Demographics Data**

[Implementation Note: If a subject is multi-racial, in "Race" column, note "Multiple: (list races, separated by a comma)."]

| Subject ID | Treatment Group | Sex | Age at Enrollment<br>(years) | Ethnicity | Race | BMI |
|---|---|---|---|---|---|---|

#### Listing 7: 16.2.4.2 – Pre-Existing and Concurrent Medical Conditions

[Implementation Note: "Condition Start Day" and "Condition End Day" are relative to enrollment (which is Day 1, day before enrollment is Day 1). If ongoing, display "Ongoing" in the "Condition End Day" column]

| Subject ID | Treatment<br>Group | MH<br>Number | Medical History<br>Term | Condition Start<br>Day | Condition End<br>Day | MedDRA® System Organ<br>Class | MedDRA® Preferred Term |
|---|---|---|---|---|---|---|---|

## **Listing 8:** 16.2.4.3 – Influenza Vaccination History

| Subject ID | Treatment Group | Vaccine Type | Month/Year Received | Vaccination Type / Subtype |
|---|---|---|---|---|
| | | [Inactivated/ LAIV/<br>Unknown] | September 2017 | Seasonal Influenza Vaccination (2016-2017) |
| | | [Inactivated/ LAIV/<br>Unknown] | June 2017 | Non-Seasonal Influenza A Vaccine Subtype H5N8 |
| | | [Inactivated/ LAIV/<br>Unknown] | June 2017 | Non-Seasonal Influenza Vaccinae Subtype M-001 |

## 16.2.5 Compliance and/or Drug Concentration Data (if available)

Not applicable for this study.

## 16.2.6 Individual Immunogenicity Response Data

**Listing 9: 16.2.6 - Individual Immunogenicity Response Data** 

| Subject ID | Treatment Group | Planned Time Point | Actual Study<br>Day | Assay | Strain | Titer Replicate 1 | Titer Replicate 2 |
|---|---|---|---|---|---|---|---|

#### 16.2.7 Adverse Events

**Listing 10: 16.2.7.1 - Solicited Events – Systemic Symptoms** 

| Subject ID | Treatment Group | Dose Number | Post Dose Day | Assessment <sup>1</sup> | Symptom | Severity | Attributed to<br>Alternate<br>Etiology? <sup>2</sup> | Alternate<br>Etiology |
|---|---|---|---|---|---|---|---|---|
| | | | | MA | | | | |
| | | | | Clinic | | | | |

<sup>&</sup>lt;sup>1</sup> MA = Data reported by subject on the Memory Aid and reviewed by clinic staff and reported in Solicited Events eCRF.

Clinic = Data collected by clinic staff during physical exam or symptom assessment (treatment administration record, in-clinic assessment, etc.)

<sup>&</sup>lt;sup>2</sup> Grade 3 events only.

#### **Listing 11: 16.2.7.2 - Solicited Events – Local Symptoms**

[Implementation Note: For group 1, dose 1 match the product received to symptoms reported based on the arm the product (IIV4, A/H7N) was received in]

| Subject ID | Treatment Group | Dose Number | Product<br>Received <sup>1</sup> | Post Dose Day | Assessment <sup>2</sup> | Symptom | Severity |
|---|---|---|---|---|---|---|---|
| | | | | | MA | | |
| | | | | | Clinic | | |

<sup>&</sup>lt;sup>1</sup> For Group 1, IIV4 and A/H7N9 vaccines are both received at Dose 1 in separate arms.

<sup>&</sup>lt;sup>2</sup> MA = Data reported by subject on the Memory Aid and reviewed by clinic staff and reported in Solicited Events eCRF.

Clinic = Data collected by clinic staff during physical exam or symptom assessment (treatment administration record, in-clinic assessment, etc.)

**Listing 12: 16.2.7.3 - Unsolicited Adverse Events** 

| Adverse<br>Event | Associated with Dose # | # of Days Post Associated Dose (Duration) | Severity | SAE?<br>MAAE?<br>PIMMC? | Relationship<br>to Study<br>Treatment | In Not<br>Related,<br>Alternative<br>Etiology | Action<br>Taken<br>with<br>Study<br>Treatment | Subject<br>Discontinued<br>Due to AE | Outcome | MedDRA®<br>System<br>Organ<br>Class | MedDRA®<br>Preferred<br>Term |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject ID | : , Treatment | Group: , AE | Number: | | | | • | | • | | |
| | | | | SAE: No<br>MAAE: Yes<br>PIMMC: No | | | | | | | |
| Comments: | | | | | | | | | | | |
| Subject ID | :, Treatment | Group: , AE I | Number: | | | | | | | | |
| | | | | | | | | | | 1 | |
| Comments: | Comments: | | | | | | | | | | |
| Note: For a | Note: For additional details about SAEs, see Section 14.3.3 | | | | | | | | | | |

#### 16.2.8 Individual Laboratory Measurements

#### **Listing 13: 16.2.8.1 - Clinical Laboratory Results – Hematology**

[Implementation Note: These listings (for hematology and chemistry) include all laboratory results, scheduled and unscheduled. These listings are not color-coded, but the severity should be included in parentheses after the result for abnormal results, e.g., 16.2 (Mild). The "extra" fields that are completed for abnormal results are not included in this listing; they are included in the listing of abnormal laboratory results that is included in the table shells.]

| Subject ID | Treatment Group | Sex | Age<br>(years) | Planned<br>Time<br>Point | Actual<br>Study<br>Day | Alanine aminotransferase (IU/L) | Total Bilirubin<br>(mg/dL) | Creatinine<br>(mg/dL) |
|---|---|---|---|---|---|---|---|---|

**Listing 14: 16.2.8.2 - Clinical Laboratory Results - Chemistry** 

| Subject ID | Treatment Group | Sex | Age<br>(years) | Planned<br>Time<br>Point | Actual<br>Study<br>Day | White Blood Cell<br>(10³/μL) | Hemoglobin<br>(g/dL) | Platelets<br>(10³/μL) |
|---|---|---|---|---|---|---|---|---|

## 16.2.9 Vital Signs and Physical Exam Findings

#### **Listing 15: 16.2.9.1 - Vital Signs**

[Implementation Note: This listing includes all vital sign assessments, scheduled and unscheduled. These listings are not color-coded, but the severity should be included in parentheses after the result for abnormal assessments, e.g., 100.7 (Mild).]

| Subject ID | Treatment Group | Planned Time<br>Point | Actual Study<br>Day | Temperature<br>(°C) | Systolic Blood<br>Pressure<br>(mmHg) | Diastolic Blood<br>Pressure<br>(mmHg) | Pulse<br>(beats/min) |
|---|---|---|---|---|---|---|---|

#### Listing 16: 16.2.9.2 - Physical Exam Findings

[Implementation Note: This listing includes all physical exam findings, scheduled and unscheduled. If a subject does not have any findings upon examination, they will not be included in this listing. If reported as an AE, display "Yes" with the AE Number in parentheses, e.g., "Yes (7)".]

| Subject ID | Treatment Group | Planned<br>Time Point | Actual<br>Study Day | Body System | Abnormal Finding | Reported as an AE?<br>(AE Number) |
|---|---|---|---|---|---|---|

#### 16.2.10 Concomitant Medications

#### **Listing 17: 16.2.10 - Concomitant Medications**

[Implementation Note: "Medication Start Day" and "Medication End Day" are relative to enrollment (which is Day 1, day before enrollment is Day -1). For medication start dates that are > 30 days prior to enrollment, rather than use exact study days, categorize as follows:

- > 5 years prior to enrollment
- 1-5 years prior to enrollment
- 1-12 months prior to enrollment

If ongoing, display "Ongoing" in the "Medication End Day" column. If taken for an AE or MH, display "Yes" with the AE or MH Number in parentheses, e.g., "Yes (7)".]

| Subject<br>ID | Treatment<br>Group | CM<br>Number | Medication | Medication Start<br>Day | Medication End<br>Day | Indication | Taken for an<br>AE?<br>(AE Number) | Taken for a condition<br>on Medical History?<br>(MH Number) |
|---|---|---|---|---|---|---|---|---|

#### 16.2.11 Pregnancy Reports

[Implementation Note: Only include the "Pregnancy Number" column if a subject has more than 1 pregnancy. Date of Conception will be calculated based on estimated delivery date. BMI will be calculated based on pre-pregnancy height and weight. Mother's weight gain will be calculated based on pre-pregnancy weight and end of pregnancy weight. If a major congenital anomaly with previous pregnancy, display "Yes" and the text from the "specify" field, separated by a colon. If any substance use is reported, include a listing of substance use. If autopsy revealed an alternate etiology, display "Yes" and the text from the "specify" field, separated by a colon.]

**Listing 18: 16.2.11.1 - Pregnancy Reports – Maternal Information** 

| Subject ID | Treatment<br>Group | Pregnancy<br>Number | Study Day<br>Corresponding<br>to Estimated<br>Date of<br>Conception | Source of<br>Maternal<br>Information | Pregnancy<br>Status | Mother's<br>Pre-<br>Pregnancy<br>BMI | Mother's<br>Weight<br>Gain<br>During<br>Pregnancy | Tobacco, Alcohol, or Drug Use During Pregnancy? | Medications<br>During<br>Pregnancy? | Maternal<br>Complications<br>During<br>Pregnancy? | Maternal<br>Complications<br>During Labor,<br>Delivery, or<br>Post-Partum? |
|---|---|---|---|---|---|---|---|---|---|---|---|

Note: Maternal Complications are included in the Adverse Event listing. Medications taken during pregnancy are included in the Concomitant Medications Listing.

Listing 19: 16.2.11.2 - Pregnancy Reports - Gravida and Para

| | | | | Live Births | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject<br>ID | Pregnancy<br>Number | Gravida | Extremely PB <sup>1</sup> | Very<br>Early<br>PB <sup>1</sup> | Early<br>PB <sup>1</sup> | Late<br>PB <sup>1</sup> | Early<br>TB <sup>2</sup> | Full<br>TB <sup>2</sup> | Late<br>TB <sup>2</sup> | Post<br>TB <sup>2</sup> | Still<br>Births | Spontaneous<br>Abortion/<br>Miscarriage | Elective<br>Abortions | Therapeutic<br>Abortions | Major<br>Congenital<br>Anomaly with<br>Previous<br>Pregnancy? |

<sup>&</sup>lt;sup>1</sup> Preterm Birth

Note: Gravida includes the current pregnancy, para events do not.

<sup>&</sup>lt;sup>2</sup> Term Birth

#### Listing 20: 16.2.11.3 - Pregnancy Reports – Live Birth Outcomes

| Subject<br>ID | Pregnancy<br>Number | Fetus<br>Number | Pregnancy<br>Outcome<br>(for this<br>Fetus) | Fetal Distress During Labor and Delivery? | Delivery<br>Method | Gestational<br>Age at Live<br>Birth | Size for<br>Gestational<br>Age | Apgar<br>Score,<br>1<br>minute | Apgar<br>Score, 5<br>minutes | Cord<br>pH | Congenital<br>Anomalies? | Illnesses/<br>Hospitalizations<br>within 1 Month<br>of Birth? |
|---|---|---|---|---|---|---|---|---|---|---|---|---|

Note: Congenital Anomalies are included in the Adverse Event listing.

#### **Listing 21: 16.2.11.4 - Pregnancy Reports – Still Birth Outcomes**

| Subject<br>ID | Date of<br>Initial<br>Report | Fetus<br>Number | Pregnancy<br>Outcome<br>(for this<br>Fetus) | Fetal Distress During Labor and Delivery? | Delivery<br>Method | Gestational<br>Age at Still<br>Birth | Size for<br>Gestational<br>Age | Cord pH | Congenital Anomalies? | Autopsy<br>Performed? | If Autopsy,<br>Etiology for Still<br>Birth Identified? |
|---|---|---|---|---|---|---|---|---|---|---|---|

#### Listing 22: 16.2.11.5 - Pregnancy Reports – Spontaneous, Elective, or Therapeutic Abortion Outcomes

| Subject<br>ID | Date of Initial<br>Report | Fetus Number | Pregnancy<br>Outcome (for this<br>Fetus) | Gestational Age at<br>Termination | Abnormality in Product of Conception? | Reason for Therapeutic<br>Abortion |
|---|---|---|---|---|---|---|